#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : Reporting and Analysis Plan for BEL115467: A Randomized, Double-Blind, Placebo-Controlled 52-Week Study to Assess Adverse Events of Special Interest in Adults with Active, Autoantibody-Positive Systemic Lupus Erythematosus Receiving Belimumab. Years 2 to 5 post-treatment follow-up period. Amendment Version 1, Prior to Y3 reporting |
|---|---|
| Compound Number | GSK1550188 |
| Clinical Study<br>Identifier | BEL115467 |
| Effective Date | 22-SEP-2020 |

#### **Description:**

- The purpose of this RAP is to describe the planned summaries to be included in the Clinical Study Report for Protocol BEL115467 Years 2 to 5 post-treatment follow-up period and the annual summaries for reporting to regulatory authorities.
- This RAP is intended to describe the safety summaries required for the Years 2 to 5 post-treatment follow-up period part of the study, to assess mortality and malignancy (including non-melanoma skin cancers [NMSC]).
- A separate RAP to describe the safety and efficacy analyses that were performed through the Week 52 double-blind treatment period of Protocol BEL115467 was finalized on 18-OCT-2018. Data from the Week 52 double-blind treatment period was unblinded and Statistical Analysis Complete (SAC) was achieved on 7-FEB-2019.
- The Years 2 to 5 post-treatment follow-up period RAP was finalized on 23-SEP-2019, after unblinding and SAC for the Week 52 double-blind treatment period part of the study but prior to the Year 2 follow-up reporting. The Year 2 SAC was achieved on 20-DEC-2019.
- This amendment to the Years 2 to 5 post-treatment follow-up period RAP was created after the Year 2 follow-up reporting and finalized before the Year 3 follow-up reporting.
- This RAP will be provided to the study team to convey the content of the SAC deliverables for the Years 2 to 5 post-treatment follow-up period.

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# RAP Author(s)

| Author | Date |
|------------------------------------------------|-------------|
| Lead | |
| Statistics Leader (Development Biostatistics) | 21-SEP-2020 |
| Co-Authors<br>PPD | 21-SEP-2020 |
| Manager Statistics (Development Biostatistics) | |

## RAP Team Reviews:

## RAP Team Review Confirmations

(Method: E-mail)

| Reviewer | Date |
|--------------------------------------------------------------|-------------|
| Programming Leader (Development Biostatistics [Programming]) | 21-SEP-2020 |
| Clinical Development Director (II and Fibrosis) 21-SE | |

# Clinical Statistics and Clinical Programming Line Approvals:

# Clinical Statistics & Clinical Programming Line Approvals

(Method: eTMF eSignature)

| Approver | | Date |
|---|---|---|
| Senior Statistics D | rector (Development Biostatistics) | 22-SEP-2020 |
| Director (Development Biostatistics [Programming]) | | 22-SEP-2020 |

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | INTR | ODUCTIO | N | | 5 |
| 2. | SLIMI | MARY OF | KEY PRO | TOCOL INFORMATION | 7 |
| ۷. | 2.1. | | | otocol Defined Statistical Analysis Plan | |
| | 2.1. | | | and Endpoint(s) | |
| | 2.3. | | | and Endpoint(s). | |
| | 2.3.<br>2.4. | | | ses | |
| | 2.4. | Statistic | ат пуроше: | 565 | |
| 3. | PLAN | INED ANA | ALYSES | | 8 |
| | 3.1. | Interim | Analyses | | 8 |
| | 3.2. | Final Ar | nalysis | | 8 |
| 4. | ANAL | YSIS PO | PULATION | S | 9 |
| • | 4.1. | | | 5 | |
| 5. | CONS | SIDEDAT | IONS EOD | DATA ANALYSES AND DATA HANDLING | |
| J. | | | | | 11 |
| | 5.1. | | | Subgroup Display Descriptors | |
| | 5.2. | | | S | |
| | 5.3. | Multicer | nter Studies | | 12 |
| | 5.4. | | | variates, Other Strata and Subgroups | |
| | | 5.4.1. | Covariate | es and Other Strata | 12 |
| | | 5.4.2. | | ion of Subgroups | |
| | 5.5. | Multiple | | ons and Multiplicity | |
| | 5.6. | | | ns for Data Analyses and Data Handling | |
| | | Conven | tions | | 13 |
| | | 5.6.1. | | of Missing Data | |
| | | | 5.6.1.1. | | |
| | | 5.6.2. | Derived a | ind Transformed Data | |
| | | | 5.6.2.1. | Race Hierarchy Rule | 15 |
| | | | 5.6.2.2. | | |
| | | | 5.6.2.3. | Year Intervals | |
| | | | 5.6.2.4. | Deaths | 17 |
| | | | 5.6.2.5. | New Malignancy | |
| | | | 5.6.2.6. | Subjects Years Follow-Up: Mortality | |
| | | | 5.6.2.7. | Follow-Up Adjusted Subject Incidence Rate per | |
| | | | | 100 Subject Years: Mortality | 20 |
| | | | 5.6.2.8. | Subject Years Follow-Up: Malignancy Subject | |
| | | | 0.0.2.0. | Incidence Rate | 21 |
| | | | 5.6.2.9. | Subject Years Follow-Up: Malignancy Event | 00 |
| | | | E C O 40 | Rate | 22 |
| | | | 5.6.2.10. | Follow-Up Adjusted Subject Incidence Rate per | 0.4 |
| | | | 50044 | 100 Subject Years: Malignancy | 24 |
| | | | 5.6.2.11. | Follow-Up Adjusted Event Rate per 100 | 0.4 |
| | | | E 0 0 40 | Subject Years: Malignancy | 24 |
| | | | 5.6.2.12. | | 0.1 |
| | | | | than Study Treatment during Year 1) | 24 |

## CONFIDENTIAL

# BEL115467

| STUE | Y POPULATION ANALYSES | 25 |
|---|---|---|
| 6.2. | | |
| | | 26 |
| SAFE | TY ANALYSES | 26 |
| REFE | RENCES | 30 |
| IXLIL | INCINOLO | 50 |
| APPE | NDICES | 31 |
| 9.1. | Appendix 1: Countries by Region | 31 |
| 9.2. | Appendix 2: Reporting Process | 32 |
| 9.3. | Appendix 3: Abbreviations & Trade Marks | 33 |
| | 9.3.1. Abbreviations | 33 |
| 9.4. | Appendix 4: List of Data Displays | 34 |
| | 9.4.1. Data Display Numbering | 34 |
| | 9.4.3. Study Population Tables | 35 |
| | 9.4.4. Safety Tables | 36 |
| | 9.4.5. ICH Listings | 37 |
| 9.5. | Appendix 5: Example Mock Shells for Data Displays | 39 |
| | 6.1.<br>6.2.<br>SAFE<br>7.1.<br>7.2.<br>REFE<br>9.1.<br>9.2.<br>9.3. | other than study treatment in Year 1). SAFETY ANALYSES. 7.1. All-Cause Mortality. 7.2. Malignancy. REFERENCES. APPENDICES. 9.1. Appendix 1: Countries by Region. 9.2. Appendix 2: Reporting Process. 9.3. Appendix 3: Abbreviations & Trade Marks. 9.3.1. Abbreviations. 9.3.2. Trade Marks. 9.4. Appendix 4: List of Data Displays. 9.4.1. Data Display Numbering. 9.4.2. Deliverables. 9.4.3. Study Population Tables. 9.4.4. Safety Tables. 9.4.5. ICH Listings. |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the summaries to be included in the Clinical Study Report for the Years 2 to 5 post-treatment follow-up period for the HGS1006-C1113 study and the annual summaries for reporting to regulatory authorities. The study will be reported under its GSK study number BEL115467.

A separate RAP describes the safety and efficacy analyses that were performed through the Week 52 double-blind treatment period. A RAP Addendum prospectively describes additional safety analyses to supplement the planned analyses through the Week 52 double-blind treatment period specified in the main RAP. Summaries and analyses for the Week 52 double-blind treatment period have been produced and reported. The RAP for the Week 52 double-blind treatment period was finalized on 18-OCT-2018. The RAP Addendum was finalized on 13-DEC-2018. Data from the Week 52 double-blind treatment period was unblinded on 2-JAN-2019 and Statistical Analysis Complete (SAC) was achieved on 7-FEB-2019.

The Years 2 to 5 post-treatment follow-up period RAP was finalized on 23-SEP-2019, after unblinding and SAC for the Week 52 double-blind treatment period part of the study but prior to the Year 2 follow-up reporting. The Year 2 SAC, following this RAP, was achieved on 20-DEC-2019.

This amendment to the Years 2 to 5 post-treatment follow-up period RAP was created after the Year 2 follow-up reporting and finalised before the Year 3 follow-up reporting. It addresses: 1) adding commercial Benlysta use to listings for subjects who died or had malignancies, 2) removing the GSK (manually assigned) PSAP category death and malignancy outputs (for the reasons given in Section 5.6) and 3) adding 2 additional COVID-19 death summaries.

This is a global, multi-center, randomized, double-blind, placebo-controlled, 52-week study to assess mortality and adverse events of special interest (AESI) in adults with active, autoantibody-positive systemic lupus erythematosus (SLE) treated with belimumab plus standard therapy vs placebo plus standard therapy. Following the 52-week study, all subjects were to be contacted annually through Year 5 (Week 260) to assess mortality and malignancy (including non-melanoma skin cancers [NMSC]).

This RAP is based upon the following study documents:

- Study Protocol Amendment 03 (May 22, 2017)
- Final Case Report Form (CRF) Version 6.2 (June 19, 2017)
- Reporting and Analysis Plan (RAP) for BEL115467 Week 52 double-blind treatment period (October 18, 2018)
- BEL115467 Week 52 double-blind treatment period RAP Addendum (Dec 13, 2018)
- RAP for BEL115467 Years 2 to 5 post-treatment follow-up period (September 23, 2019)
- Program Safety Analysis Plan (PSAP) Version 6 (October 2, 2018). Note: for reporting purposes, the most current version of the PSAP at the time of annual reporting/Year 5 database freeze (DBF) will be used. For reference,

#### **CONFIDENTIAL**

BEL115467

sections of the PSAP that are relevant to reporting are given in the separate Week 52 double-blind treatment period RAP, Appendix 6: PSAP Sections for AESI Reporting.

This Amendment to the Years 2 to 5 post-treatment follow-up period RAP was finalized after unblinding and SAC for the Week 52 double-blind treatment period part of the study, after the Year 2 follow-up reporting but before the Year 3 follow-up reporting.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned summaries for the Years 2 to 5 post-treatment follow-up period as specified in protocol amendment 3 [(Dated: 22-MAY-2017)]. Information in the protocol regarding the summary of data from the Years 2 to 5 post-treatment follow-up period was minimal.

Information relating to changes to the protocol defined statistical analysis plan for the Week 52 double-blind treatment period can be found in the separate Week 52 double-blind treatment period RAP.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Years 2 to 5 Post-Treatment Follow-Up Period | |
| To assess mortality and malignancy | All-cause mortality |
| (including NMSC) during Years 2 to 5. | Malignancies (including NMSC) |

Objectives and endpoints for the Week 52 double-blind treatment period are described in the separate Week 52 double-blind treatment period RAP.

# 2.3. Study Design

This is a global, multi-center, randomized, double-blind, placebo-controlled, 52-week study to assess mortality and AESI in adults with active, autoantibody-positive SLE treated with belimumab plus standard therapy vs placebo plus standard therapy. It was planned that approximately 4,000 subjects would be randomized (1:1) to belimumab plus standard therapy or placebo plus standard therapy. Randomization was stratified for region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia; see Appendix 1: Countries by Region: Countries by Region for details of countries and regions), Safety of Estrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) score (≤9 vs ≥10), and steroid dose (≤7.5 mg/day vs >7.5 mg/day prednisone or equivalent). There was no minimum score required for the SELENA SLEDAI to be eligible for this study.

Subjects were to receive investigational product (IP) on Days 0, 14, 28, and every 28 days thereafter through Week 48 with a final visit conducted at Week 52. Following the 52-week study, all subjects were to be contacted annually through Year 5 to assess mortality and malignancy (including NMSC). Subjects who discontinued treatment at any time during the study but did not withdraw consent were to be followed at 28-day intervals through Week 52. If the subject withdrew consent prior to Week 52, an attempt was to be made to assess mortality and occurrence of malignancy (including NMSC) at Week 52 and annually for Years 2 to 5. See protocol Section 3.1 for further details. Protocol time windows are  $\pm$  30 days for annual follow-up contacts from Year 2 to Year 5.

In the Years 2 to 5 post-treatment follow-up period, subjects no longer receive study treatment, but instead receive physician directed standard of care.

Data collection in the Years 2 to 5 post-treatment follow-up period was limited and included information on survival status, information on new primary malignancies (including NMSC) and start date of first exposure to commercial Benlysta (other than investigational product during Year 1). For Years 2 to 5, annual follow-up was planned to be conducted via telephone.

Due to the COVID-19 pandemic (which started after all subjects completed Week 52 and Year 2), there may be more missed or out of window follow-up contacts and more study withdrawals (withdrew consent and lost to follow up). Site personnel may not be available to make calls or have access to the database. However, some of this data may be populated later once more normal activities resume. There may also be potentially more deaths. Therefore 2 additional death summaries have been added to enable the team to assess the impact of the COVID-19 pandemic on the mortality summaries.

# 2.4. Statistical Hypotheses

There are no formal statistical hypotheses for this study. The main purpose of the Years 2 to 5 post-treatment follow-up period is to provide an evaluation of the rates of all-cause mortality and malignancies (including NMSC) during Years 2 to 5 grouped by treatment received during the Week 52 double-blind treatment period (belimumab or placebo).

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

Following the final analysis of the double-blind treatment period through Week 52, interim summaries will be generated to report post-treatment follow-up mortality and malignancy rates at the end of Year 2, Year 3, and Year 4 for ongoing reporting purposes, including to health authorities.

Data will be cleaned in an ongoing way, so the data are as clean as possible for each annual reporting effort. In-stream database cuts (with no database lock) will be taken for the end of Year 2, Year 3 and Year 4 interim reporting efforts. However, as the database will not be formally locked until the end of Year 5 reporting, the data may change up until the time of the final analysis.

All outputs specified in the RAP will be produced as appropriate for the RAP version relevant for the end of Year 2, Year 3, and Year 4 interim reporting efforts. The final reporting effort will be the end of Year 5 reporting.

# 3.2. Final Analysis

Summaries and analyses for the Week 52 double-blind treatment period have been produced and reported. Data from the Week 52 double-blind treatment period was unblinded on 2-JAN-2019 and SAC was achieved on 7-FEB-2019.

The database release (DBR) for the Years 2 to 5 post-treatment follow-up period will occur after data through the Year 5 survival status and occurrence of malignancy follow-up have been collected, verified and validated.

The final planned analysis for the Years 2 to 5 post-treatment follow-up period will be performed when all required database cleaning activities for this part of the study have been completed and final database release (DBR) and database freeze (DBF) have been declared by Data Management.

All outputs required for the Post-Treatment Follow-Up Period (Years 2 to 5) will be listed in a Mock Tables, Listings and Figures (TLFs) Shells document.

#### 4. ANALYSIS POPULATIONS

The purpose of the post-treatment follow-up period is to assess mortality and malignancy, therefore the As-Treated population will be used. The As-Treated population will be defined as described in the Week 52 double-blind treatment period RAP. In addition, four subsets of this overall population will be defined — one for each year of the follow-up period.

#### **As-Treated**

The As-Treated population is defined using data from the Week 52 double-blind treatment period. It includes all subjects who were randomized and received at least one dose of study agent. The As-Treated population will group subjects according to the actual treatment administered to the subject based on the treatment that the subject received most of the time (>50% of the time). Therefore, if a subject received an incorrect treatment at more than half the visits, the As-Treated treatment group assignment will differ from the randomized treatment group assignment.

Summary tables which present the number of subjects at Week 52, for use as a denominator for Week 52, will include all subjects in the As-Treated population.

#### **As-Treated Follow-Up Population Subsets**

Separate populations will be created to identify which subjects are included in each post-treatment follow-up year (Year 2, Year 3, Year 4 and Year 5). Subjects will be included in the post-treatment follow-up subsets of the As-Treated population and summarized according to the actual treatment administered during the Week 52 double-blind treatment period (as defined for the As-Treated population). It should be noted that subjects in the post-treatment follow-up period will no longer be receiving study treatment.

Subjects will be included in the subset populations based on the completion of the survival status question at the follow-up visits and using nominal visit from the eCRF. The last post-treatment follow-up visit a subject completes will be identified from visits where the survival status question was completed. Completion of the survival status question would include responses of Alive, Dead, Lost to Follow-up or Withdrew Consent. If the response to the survival status question is missing (or the visit is not completed) then this visit will not be included when identifying the last post-treatment follow-up assessment completed.

Subjects will be included in the population subsets based on the last post-treatment follow-up assessment completed and included in the follow-up subsets for all years up to and including the last post-treatment follow-up visit completed.

Any subject who completes the follow-up assessments as described above will be included in the follow-up subsets, regardless of their status at Week 52.

| Population | Definition / Criteria |
|---|---|
| Year 2 Follow-Up | All subjects in the As-Treated population whose last completed post-<br>treatment follow-up visit was Year 2, Year 3, Year 4 or Year 5. |
| Year 3 Follow-Up | All subjects in the As-Treated population whose last completed post-<br>treatment follow-up visit was Year 3, Year 4 or Year 5. |
| Year 4 Follow-Up | All subjects in the As-Treated population whose last completed post-<br>treatment follow-up visit was Year 4 or Year 5. |
| Year 5 Follow-Up | All subjects in the As-Treated population whose last completed post-<br>treatment follow-up visit was Year 5. |
| Any Year 2 to 5 Follow-Up | <ul> <li>All subjects in the As-Treated population who completed at least one post-treatment follow-up visit for Year 2 to 5.</li> <li>Note: This will be the same as the Year 2 Follow-Up population. Its main use will be to describe subjects included in data listings.</li> </ul> |

#### 4.1. Protocol Deviations

Important protocol deviations relating to the Years 2 to 5 post-treatment follow-up period will be listed. Any protocol deviations due to COVID-19 will be prefixed with 'COVID-19'. Deviations already reported for the Week 52 double-blind treatment period (including deviations related to study inclusion/exclusion criteria) will not be considered, as these are reported separately as part of the Week 52 double-blind treatment period SAC.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP) for the annual follow-up phase [13 August 2019, Version 1.2]. If the PDMP is updated, the most current version of the PDMP will be used.

- Data will be reviewed on an ongoing basis and prior to freezing the database to
  ensure all important deviations are captured and categorized on the protocol
  deviations dataset.
- This dataset will be the basis for the listing of protocol deviations.
- Year 1 PDs which were identified and reported after completion of the Week 52 CSR but before 25 Sep 2019 were described in the Year 2 post-treatment follow-up report. Year 1 PDs which were identified and reported between 26 Sep 2019 and 23 Sep 2020 will be described in the Year 3 post-treatment follow-up report, and similarly for the Year 4 post-treatment follow-up report. All Year 1 PDs which were identified and reported after completion of the Week 52 CSR will be included in the final follow-up report.
- For the Year 3 post-treatment follow-up report, non-important protocol deviations due to COVID-19 will be provided in a PDF file directly from CTMS, for inclusion in an appendix in the Year 3 post-treatment follow-up report. For Year 4 and Year 5 reporting, non-important protocol deviations will be added to the SDTM DV data and a listing of non-important protocol deviations due to COVID-19 will be produced for inclusion in an appendix in the Year 4 and Year 5 post-treatment follow-up reports.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Subgroup Display Descriptors

In the Years 2 to 5 post-treatment follow-up period, subjects no longer receive study treatment, but instead receive physician directed standard of care. The following treatment descriptors from the Week 52 double-blind treatment period will be used on all data tabulations:

- Placebo
- Belimumab 10 mg/kg

In all summary tables, the data will also be presented for all subjects using a Total column.

A footnote will be added to all displays to indicate that subjects in the post-treatment follow-up period are no longer receiving study treatment, and the treatment group assignment is based on treatment received during the Week 52 double-blind treatment period part of the study.

## 5.2. Baseline Definitions

Demographic and baseline characteristics will be derived as described in the Week 52 double-blind treatment period RAP. Any summaries of demographic and baseline characteristics data presented as part of the Years 2 to 5 post-treatment follow-up period will summarize the demographic or baseline data as at the start of the Week 52 double-blind treatment period.

Analysis age is derived in years relative to the treatment start date for randomized subjects, and is calculated in SAS as follows:

INTCK ('YEAR', Date of birth, Date of treatment start date, 'C').

Region will be presented as US/Canada, Central America/South America/Mexico, Europe/Australia/Israel, and Asia.

Race will be presented in the demography table as Black vs. Other. The Black category is defined as subjects who are in the race category "Black or African American". The race hierarchy rule (Section 5.6.2.1) will not apply and a subject will be categorized as Black if they have selected multiple race categories and any of them is "Black or African American".

SLE Disease Duration is defined as

If either date is missing, then SLE Disease Duration will be missing. Partial dates for SLE diagnosis date will be imputed as described in Section 5.6.1.1.

Screening SELENA SLEDAI category will be presented as  $\leq 9$  and  $\geq 10$ . Note: if any individual item is missing the total score cannot be calculated, however if the subject can be definitively categorized as  $\leq 9$  or  $\geq 10$  regardless of the response to the missing item(s) then the appropriate category will be assigned.

Screening Complement Levels and Anti-dsDNA categories (Low Complement and High Anti-dsDNA binding, Not (Low Complement and High Anti-dsDNA binding)) will be derived from the screening SELENA SLEDAI assessment. This is intended to be an indicator of high versus low disease activity. Note: If the evaluations to the SELENA SLEDAI assessment questions "Low Complement" and "Increased DNA Binding" are both missing, the subject will not be classified into one of the categories. If either item is marked "No", the subject will be classified into the Not (Low Complement and High Anti-dsDNA binding) group regardless of whether the other item is missing or "Yes".

Complement Levels (Low, Not Low) and Anti-dsDNA Binding (High, Not High) will also be derived from the screening SELENA SLEDAI assessment.

Baseline Systemic Lupus International Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index will be derived as specified in Section 9.5.19 and Appendix 5 of the Week 52 double-blind treatment period RAP. Baseline SLICC category will be also be categorized as 0, 1 or >1.

#### 5.3. Multicenter Studies

This is a multi-center trial and subjects were randomized by region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia) –see Appendix 1 for details of countries and regions. There will be no summaries performed at the center level.

Enrollment by site will not be presented for the Years 2 to 5 post-treatment follow-up period, as this data has been summarized as part of the Week 52 double-blind treatment period part of the study.

# 5.4. Examination of Covariates, Other Strata and Subgroups

# 5.4.1. Covariates and Other Strata

Details of randomization strata are included in the separate Week 52 double-blind treatment period RAP (Section 8.2). Covariates are not relevant for these safety analyses.

## 5.4.2. Examination of Subgroups

Data from the Years 2 to 5 post-treatment follow-up period will not be summarized by subgroups.

## 5.5. Multiple Comparisons and Multiplicity

There is no statistical hypothesis to be tested (no formal statistical testing) for the safety analyses, and therefore no need to control for multiple comparisons.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

- All data summaries and analyses will be performed using the latest available version of SAS software (as available at GSK).
- Data displays will follow the shells outlined in the Mock TLFs document which will follow the Benlysta program standards and, as far as possible, follow the agreements proposed by the GSK Integrated Data Standards Library (IDSL).
- The most current version of Medical Dictionary for Regulatory Activities (MedDRA) at the time of DBF will be used for reporting.
- The most current version of the Benlysta PSAP at the time of DBF will be used for reporting.
- Where SDTM terminology differs from the eCRF and/or mock shells, the SDTM terminology will be presented in displays unless otherwise specified.

Unless otherwise stated, the following will apply:

- Continuous variables will be summarized with the statistics mean, median, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum.
- Categorical variables will be summarized with frequency counts and percentages, or proportions where specified. A 'Missing' category will be added to frequency counts if there is at least one missing record.
- Percentages will be calculated using the number of subjects in the relevant population/treatment group (denoted by N) as the denominator, unless otherwise stated.
- The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database.
- The mean, median, 25<sup>th</sup> percentile and 75<sup>th</sup> percentile will be reported to one more decimal place than the raw data recorded in the database.
- The SD will be reported to two more decimal places than the raw data recorded in the database.
- A maximum of four decimal places will be used.
- Percentages will be presented to one decimal place unless otherwise specified (i.e. deaths and malignancies will be presented to 2 decimal places). Incidence rates will be presented to two decimal places.
- A count of zero will have no corresponding percentage.
- Listings will be based on the As-Treated population (unless otherwise specified) and generally be limited to those required by ICH guidelines and will be sorted by treatment group, investigator number, subject number and visit (where appropriate).

#### MedDRA Coding of Death and Malignancy:

Deaths reported during the Week 52 double-blind study period were collected as adverse event data. In the year 2-5 follow up period for BEL115467 the primary reason of death is collected on the annual FU survival form and will be coded using

the latest version of MedDRA (with SOC and PT); detailed SAE information is NOT collected. There are coding limitations for death data from the post-treatment follow-up period, as the information available to code was limited to the verbatim 'primary reason for death'.

Malignancies reported during the 52-week double-blind treatment period of the study were collected as adverse event data. New primary malignancies reported in the post-treatment follow-up period are collected on the annual FU survival form and will be coded using the latest version of MedDRA (with SOC and PT). There are coding limitations for malignancy data from the post-treatment follow-up period, as the information available to code was limited to the verbatim 'diagnosis'.

For the interim reporting efforts (Years 2, 3 and 4) every effort will be made to code all reported terms, however this may not be possible and there may be un-coded terms for interim reporting efforts.

Data for deaths and malignancies from the Week 52 double-blind treatment period adverse event data will not be re-coded as part of Years 2-5 reporting. Summary tables presenting deaths and malignancies by MedDRA SOC/PT will not include data from the Week 52 double-blind treatment period. Summaries of these data can be found in the Week 52 double blind treatment period CSR and will not be duplicated in the post-treatment follow-up summaries.

A decision was made by the Benlysta Safety Review Team (SRT) in April 2020 to stop manual categorization (using the PSAP adjudication categories described in Appendix 6 of the Week 52 double-blind treatment period RAP) of Year 2-5 deaths and malignancies for Year 3 reporting onwards for the following reasons:

- Many events cannot be definitively categorised using the limited information
  available from verbatim primary cause of death/malignancy diagnosis.
  Clinical corroboration of the reported terms is generally not possible.
  Ambiguities often cannot easily be resolved because it is not possible to query
  the site staff to follow up with the subject and/or review medical records (as
  was done during the treatment period of the study).
- As a result, it is particularly difficult to overcome the inherent difficulties introduced by manual categorisation, such as inconsistencies between reviewers/review sessions and the need to protect against the potential for hidden biases/subjective interpretation of extremely minimal information.
- Therefore manual categorisation adds little value above programmatic coding.

Therefore summaries of deaths and malignancies by manual categorisation to GSK PSAP category have been omitted from this RAP Amendment Version 1 and the mock shells.

## 5.6.1. Handling of Missing Data

All safety summaries will use the observed data, which are the data collected or observed for the subject with no imputation for missing data, unless otherwise stated.

# **5.6.1.1.** Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | • Partial dates will be displayed as captured in subject listings. |
| Date of Birth | <ul> <li>Only year of birth is collected on the CRF.</li> <li>Day will be set to 30 and month will be set to JUNE for all subjects.</li> </ul> |
| Date of SLE diagnosis | • For records where month and day are missing for diagnosis date, impute with 01 for day and January for month to assume that the duration was the longest possible duration. |
| | • For records where the day only is missing for start date, impute with 01 for day to assume that the duration was the longest possible duration. |
| Date of Death | • For records where month and day are missing for date of death, impute 01 for day and January for month. |
| | • For records where the day only is missing, impute 01 for day. |
| | • Unless there is other information available which indicates a subject was alive at a later date, in which case the last known alive date will be imputed as the date of death i.e. maximum (imputed date of death, latest last known alive date). This will only be done where a partial date of death is recorded. |
| Last known to be alive | • For records where month and day are missing for last known to be alive date, impute 01 for day and January for month. |
| date | • For records where the day only is missing, impute 01 for day. |
| | • For subjects with a survival status of withdrew consent reported on the eCRF at a follow-up visit, there is no date of last known alive collected. In these cases, the date of follow-up contact will be used as the date the subject was last known alive. |
| Date of diagnosis (new | <ul> <li>For records where month and day are missing for date of<br/>diagnosis, impute 01 for day and January for month.</li> </ul> |
| malignancies) | • For records where the day only is missing, impute 01 for day. |

# 5.6.2. Derived and Transformed Data

# 5.6.2.1. Race Hierarchy Rule

If multiple race categories are checked on the eCRF, the subject will be assigned to a unique race group based on which of the races checked appears first in the list below:

- Native Hawaiian or Other Pacific Islander
- American Indian or Alaska Native

- Asian
- Black or African American
- White

For example, if Black or African American and Asian are both checked, then the subject will be assigned as Asian since it appears highest in the list. In the race and racial combination details table, subjects with multiple race categories checked will be reported in the race per the hierarchical rule as well as in the multiracial category. Subjects who select more than one Asian category and no other non-Asian categories will be represented in the Mixed Asian Race category as well as the Asian category. Similarly, subjects who select both white categories and no non-white categories will be represented in the Mixed White Race category as well as the White/Caucasian category. The Mixed Asian Race and Mixed White Race categories will only appear in the table if a subject selects multiple Asian or multiple white categories, respectively.

For the race categorization of Black vs Other, if a subject selects multiple races they will be assigned "Black" if any of the races is "Black or African American", i.e., the hierarchical rule will not apply in this instance (see Section 5.2).

#### 5.6.2.2. Study Day

Study Day is the number of days from the treatment start date to a study date of interest (e.g. event start date) and is calculated as follows:

| If condition is | Then Study Day is |
|---|---|
| study date <treatment date<="" start="" td=""><td>study date – treatment start date</td></treatment> | study date – treatment start date |
| study date is ≥treatment start date | study date – treatment start date +1 |

Note: Study Day cannot be zero. If either date is missing, then Study Day is missing.

Note: Study day is calculated from treatment start date in the Week 52 double-blind treatment period part of the study.

#### 5.6.2.3. Year Intervals

All-cause mortality and malignancies (including NMSC) will be summarized by follow-up year. The nominal visit will be used for yearly summaries. There will be no slotting of visits into years using dates.

The planned study day of each year is as follows (using a 365-day calendar year):

| Study Year | Planned Study Day of Visit |
|------------------|----------------------------|
| Week 52 | Day 365 ± 7 |
| Year 2 Follow-Up | Day 730 ± 30 |
| Year 3 Follow-Up | Day 1095 ± 30 |
| Year 4 Follow-Up | Day 1460 ± 30 |
| Year 5 Follow-Up | Day 1825 ± 30 |

Note: Treatment start date is Day 1.

Note: The protocol study calendar refers to Week 52 as Day 364 (and uses Day 0 terminology). This equates to study Day 365, as calculation of study day does not allow a Day 0 but starts at Day 1.

#### 5.6.2.4. Deaths

Deaths will be identified using data reported on the survival status form of the eCRF (i.e. survival status = DEAD).

In addition, sites have been instructed to collect additional data on deaths due to the COVID-19 pandemic. If COVID-19 was the primary reason for death, then the "Primary cause of death" field on the survival status form in the eCRF was to be recorded using specific COVID-19 terms. In the reporting, COVID-19 deaths will be identified per custom MedDRA query (CMQ), using GSK TOI LISTID 318947.

For deaths where COVID-19 may have been a contributory factor but was not the primary cause of death, sites have been instructed to add a comment in the eCRF. These comments are not included in the database, but will be extracted directly from the EDC (INFORM) system, for inclusion in the Year 3, 4 and 5 follow-up reports.

Deaths will be assigned to Week 52, Year 2 follow-up, Year 3 follow-up, Year 4 follow-up or Year 5 follow-up based on the nominal visit of the survival status form where death is reported. For deaths reported during the Week 52 double-blind treatment period, this is equivalent to deaths which occurred during the on-study period (see Section 9.1.1 of the separate Week 52 double-blind treatment period RAP) i.e. deaths reported up to study Day 372.

Date of death is not collected on the Week 52 survival status form. In these cases the date of death will be derived as the end date of the SAE with fatal outcome. For deaths reported after Week 52, date of death is collected on the survival status form.

#### 5.6.2.5. New Malignancy

Malignancies will be identified using data reported on the malignancy question of the eCRF (i.e. any new malignancies to report (including NMSC)). New malignancies will be assigned to Week 52, Year 2 follow-up, Year 3 follow-up, Year 4 follow-up or Year 5 follow-up based on the nominal visit of the malignancy form where a new malignancy is reported. For malignancies reported during the Week 52 double-blind treatment period, this is equivalent to PSAP defined malignancies reported in the adverse event data which occurred during the on-study period (see Section 9.1.1 of the separate Week 52 double-blind treatment period RAP).

New malignancies reported at Week 52 with a diagnosis of 'UNKNOWN,NO FOLLOW-UP' (SDTM.CE.CETERM) will not be considered to be malignancies.

For all malignancies, date of diagnosis will be the date of diagnosis collected on the malignancy form.

#### 5.6.2.6. Subjects Years Follow-Up: Mortality

Subject years follow-up for mortality is calculated as described below, regardless of the primary cause of death (COVID-19 or other).

In order to calculate the follow-up adjusted incidence rate of mortality per 100 subject years by follow-up year (cumulative), the subject years follow up will need to be defined for each subject at each follow-up time point.

For each subject a single date of death or last known alive date will be derived as follows.

For subjects who entered the follow-up period (i.e. are in any of the Year 2 to 5 population subsets):

- For subjects who have died, the date of death will be used in the subject follow-up years calculations.
- For subjects who have not died, the latest last known alive date across all follow-up visits will be found.

For subjects who did not enter the follow-up period (i.e. are not in any of the Year 2 to 5 population subsets):

- For subjects who have died, the date of death will be used in the subject follow-up years calculations.
- For subjects who were alive or lost to follow-up at the Week 52 survival status assessment, the last known alive date from the Week 52 survival status form will be used. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed 365 days for these subjects.
- For subjects where the Week 52 survival status was missing, the study withdrawal or completion date (DSSTDT) will be used as the last known alive date. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed 365 days for these subjects. Note: there were four subjects with missing Week 52 survival status where the study withdrawal or completion date was missing; for these subjects the study agent discontinuation date (IPDISCDT) was used as the last known alive date.

Using this date of death or last known alive date, the total subject follow-up will be derived for each subject as:

• Subject follow-up (days) = (Date of death/Last Known Alive Date – Study Treatment Start Date +1)

The amount of subject follow-up days contributing to each of the cumulative timepoints (by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up, by Year 5 follow-up) is described below. In order to account for date of death or last known alive date which is out of the correct range of study days for a particular year, the following derivation will be used:

| Study Year | Subject Follow-Up (days) |
|---|---|
| By Week 52 | Minimum (Date of death/Last Known Alive Date – Treatment<br>Start Date + 1, 365) |
| By Year 2 Follow-Up | Minimum (Date of death/Last Known Alive Date – Treatment<br>Start Date + 1, 730) |
| By Year 3 Follow-Up | Minimum (Date of death/Last Known Alive Date – Treatment Start Date + 1, 1095) |
| By Year 4 Follow-Up | Minimum (Date of death/Last Known Alive Date – Treatment<br>Start Date + 1, 1460) |

| Study Year | Subject Follow-Up (days) |
|---|---|
| By Year 5 Follow-Up | Minimum (Date of death/Last Known Alive Date – Treatment<br>Start Date + 1, 1825) |

Note: individual subjects will only be allowed to contribute a maximum of 365 days for each individual follow-up year, regardless of when the follow-up visit was performed.

Note: For each subject, subject follow-up for each time period is cumulative since study treatment start date. For example, 'by Year 2 follow-up' includes follow-up time during Year 1 and follow-up time during Year 2 (to a maximum of 730 days).

The subject follow-up days will be converted to years as follows:

• Subject follow-up (years) = subject follow-up (days) / 365.25

The total follow-up years will be calculated for each of the timepoints as the sum of the subject follow-up years for that timepoint for all subjects in the As-Treated population.

An example of the amount of subject follow-up days included in each year period, for subjects where the date of death or the last known alive date falls within the correct study day range for each year, is:

| Subjects Enter | | Subjects Years Follow-Up (days) |
|---|---|---|
| Follow-Up Period [1] | Subject Years | Subjects rears rollow-op (days) |
| Tollow-op reliou [1] | Follow-Up Included | |
| | By Year | |
| Subject death during | Week 52 | 365 |
| Year 2 Follow-Up | Year 2 Follow-Up | Date of death – Treatment Start Date +1 |
| . от 2 голон ор | Year 3 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 4 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 5 Follow-Up | Date of death – Treatment Start Date +1 |
| Subject death during | Week 52 | 365 |
| Year 3 Follow-Up | Year 2 Follow-Up | 730 |
| | Year 3 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 4 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 5 Follow-Up | Date of death – Treatment Start Date +1 |
| Subject death during | Week 52 | 365 |
| Year 4 Follow-Up | Year 2 Follow-Up | 730 |
| | Year 3 Follow-Up | 1095 |
| | Year 4 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 5 Follow-Up | Date of death – Treatment Start Date +1 |
| Subject death during | Week 52 | 365 |
| Year 5 Follow-Up | Year 2 Follow-Up | 730 |
| | Year 3 Follow-Up | 1095 |
| | Year 4 Follow-Up | 1460 |
| | Year 5 Follow-Up | Date of death – Treatment Start Date +1 |
| Subject Last Known | Week 52 | 365 |
| to be Alive during | Year 2 Follow-Up | Last known alive date – Treatment Start Date +1 |
| Year 2 Follow-Up | Year 3 Follow-Up | Last known alive date – Treatment Start Date +1 |
| | Year 4 Follow-Up | Last known alive date – Treatment Start Date +1 |
| | Year 5 Follow-Up | Last known alive date – Treatment Start Date +1 |
| Subject Last Known | Week 52 | 365 |
| to be Alive during | Year 2 Follow-Up | 730 |

| Subjects Enter<br>Follow-Up Period [1] | Subject Years<br>Follow-Up Included<br>By Year | Subjects Years Follow-Up (days) |
|---|---|---|
| Year 3 Follow-Up | Year 3 Follow-Up | Last known alive date – Treatment Start Date +1 |
| | Year 4 Follow-Up | Last known alive date – Treatment Start Date +1 |
| | Year 5 Follow-Up | Last known alive date – Treatment Start Date +1 |
| Subject Last Known | Week 52 | 365 |
| to be Alive during | Year 2 Follow-Up | 730 |
| Year 4 Follow-Up | Year 3 Follow-Up | 1095 |
| | Year 4 Follow-Up | Last known alive date – Treatment Start Date +1 |
| | Year 5 Follow-Up | Last known alive date – Treatment Start Date +1 |
| Subject Last Known | Week 52 | 365 |
| to be Alive during | Year 2 Follow-Up | 730 |
| Year 5 Follow-Up | Year 3 Follow-Up | 1095 |
| | Year 4 Follow-Up | 1460 |
| | Year 5 Follow-Up | Last known alive date – Treatment Start Date +1 |

<sup>[1]</sup> Based on As-Treated Population Subsets for Years 2 to 5 Follow-Up.

| Subjects Do Not Enter | | Subjects Years Follow-Up (days) |
|---|---|---|
| Follow-Up Period [1] | Subject Years | , , |
| | Follow-Up Included | |
| | By Year | |
| Subject death during | Week 52 | Date of death – Treatment Start Date +1 |
| Week 52 | Year 2 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 3 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 4 Follow-Up | Date of death – Treatment Start Date +1 |
| | Year 5 Follow-Up | Date of death – Treatment Start Date +1 |
| Subject Last Known | Week 52 | Minimum (Last known alive date – Treatment Start |
| to be Alive during | | Date +1, 365) |
| Week 52 | Year 2 Follow-Up | Minimum (Last known alive date – Treatment Start Date +1, 365) |
| | Year 3 Follow-Up | Minimum (Last known alive date – Treatment Start Date +1, 365) |
| | Year 4 Follow-Up | Minimum (Last known alive date – Treatment Start Date +1, 365) |
| | Year 5 Follow-Up | Minimum (Last known alive date – Treatment Start Date +1, 365) |

<sup>[1]</sup> Based on As-Treated Population Subsets for Years 2 to 5 Follow-Up.

# 5.6.2.7. Follow-Up Adjusted Subject Incidence Rate per 100 Subject Years: Mortality

Deaths will be assigned to a timepoint (i.e. Week 52, Year 2, Year 3, Year 4 or Year 5) using the survival status nominal visit where the death was reported. Cumulative deaths to each timepoint will be summarized and follow-up adjusted subject incidence rates calculated.

The follow-up adjusted subject incidence rate presented for each timepoint will be a cumulative follow-up adjusted subject incidence rate from study treatment start date to the appropriate follow-up period. The subject years will be the sum of subject years for all subjects to that timepoint (as described in Section 5.6.2.6).

 $Incidence \ Rate = 100 \ \times \frac{Number \ of \ subjects \ with \ an \ event}{Subject \ Years}$ 

#### 5.6.2.8. Subject Years Follow-Up: Malignancy Subject Incidence Rate

In order to calculate the follow-up adjusted subject incidence rate of new malignancies per 100 subject years by follow-up year (cumulative), the subject years follow up will need to be defined for each subject at each follow-up time point.

This will be done in a similar way to subject years follow-up for mortality (Section 5.6.2.6) but will use date of follow-up contact, rather than date last known alive, as the censoring date. And will use date of diagnosis, rather than date of death as the event date (note: date of diagnosis using SDTM.CE.CESTDTC).

Note: New malignancies reported at Week 52 with a diagnosis of 'UNKNOWN,NO FOLLOW-UP' (SDTM.CE.CETERM) will not be considered to be malignancies (see Section 5.6.2.5).

For each subject a single date of first new malignancy or last follow-up contact date will be derived as follows.

For subjects who entered the follow-up period (i.e. are in any of the Year 2 to 5 population subsets):

- For subjects who have a new malignancy reported, the date of diagnosis of the first new malignancy will be used in the subject follow-up years calculations. Note: this includes malignancies reported by Week 52.
- For subjects who have not reported a new malignancy at any follow-up visit, the date of last follow-up contact across all follow-up visits will be found (using all visits where the new malignancy question was answered as NO) and used as the censoring date. If this follow-up contact date is later than the last known alive date (or date of death) used in the mortality subject years follow-up then the date of last known alive (or date of death) will be used as the censoring date instead.
- For subjects where the date of last follow-up contact across all follow-up visits is missing (i.e. subjects who have not reported a new malignancy and have no Year 2-5 follow-up visits where the new malignancy question was answered as NO), then the study completion or withdrawal date from the Week 52 double-blind treatment period will be used as the censoring date. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed 365 days for these subjects.

For subjects who did not enter the follow-up period (i.e. are not in any of the Year 2 to 5 population subsets):

- For subjects who have a new malignancy reported, the date of diagnosis of the first new malignancy will be used in the subject follow-up years calculations.
- If a subject did not have a new malignancy reported by Week 52, the study completion or withdrawal date from the Week 52 double-blind treatment period will be used as the censoring date. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed

365 days for these subjects. Note: there were four subjects where the study withdrawal or completion date was missing; for these subjects the study agent discontinuation date (IPDISCDT) was used as the last known alive date.

Using this date of malignancy diagnosis or censoring date, the total subject follow-up will be derived for each subject as:

• Subject follow-up (days) = (Date of malignancy diagnosis/Censoring Date – Study Treatment Start Date +1)

The amount of subject follow-up contributing to each of the cumulative timepoints (by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up, by Year 5 follow-up) is described below. In order to account for date of diagnosis or censoring date which is out of the correct range of study days for a particular year, the following derivation will be used:

| Study Year | Subject Follow-Up (days) |
|---|---|
| By Week 52 | Minimum (Date of diagnosis/Censoring Date – Treatment Start Date + 1, 365) |
| By Year 2 Follow-Up | Minimum (Date of diagnosis/Censoring Date – Treatment Start Date + 1, 730) |
| By Year 3 Follow-Up | Minimum (Date of diagnosis/Censoring Date – Treatment Start Date + 1, 1095) |
| By Year 4 Follow-Up | Minimum (Date of diagnosis/Censoring Date – Treatment Start Date + 1, 1460) |
| By Year 5 Follow-Up | Minimum (Date of diagnosis/Censoring Date – Treatment Start Date + 1, 1825) |

Note: individual subjects will only be allowed to contribute a maximum of 365 days for each individual follow-up year, regardless of when the follow-up visit was performed.

Note: For each subject, subject follow-up for each time period is cumulative since study treatment start date. For example, 'by Year 2 follow-up' includes follow-up time during Year 1 and follow-up time during Year 2 (to a maximum of 730 days).

The subject follow-up days will be converted to years as follows:

• Subject follow-up (years) = subject follow-up (days) / 365.25

The total follow-up years will be calculated for each of the timepoints as the sum of the subject follow-up years for that timepoint for all subjects in the As-Treated population.

#### 5.6.2.9. Subject Years Follow-Up: Malignancy Event Rate

In order to calculate the follow-up adjusted event rate of new malignancies per 100 subject years by follow-up year (cumulative), the subject years follow up will need to be defined for each subject at each follow-up time point.

As subjects can report more than one new malignancy, and this is an event level calculation, subject follow-up years will not be truncated at the date of first diagnosis for subjects reporting a new malignancy.

For each subject a single date of last follow-up contact date will be derived as follows.

For subjects who entered the follow-up period (i.e. are in any of the Year 2 to 5 population subsets):

- The date of last follow-up contact across all follow-up visits will be found (using all visits where the new malignancy question was answered as NO or YES) and used as the censoring date. If this follow-up contact date is later than the last known alive date (or date of death) used in the mortality subject years follow-up then the date of last known alive (or date of death) will be used as the censoring date instead.
- For subjects where the date of last follow-up contact across all follow-up visits is missing (i.e. subjects who have not reported a new malignancy and have no Year 2-5 follow-up visits where the new malignancy question was answered as NO), then the study completion or withdrawal date from the Week 52 double-blind treatment period will be used as the censoring date. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed 365 days for these subjects.

For subjects who did not enter the follow-up period (i.e. are not in any of the Year 2 to 5 population subsets):

• The study completion or withdrawal date from the Week 52 double-blind treatment period will be used as the censoring date. In calculations, the data for these subjects will be truncated so that subject follow-up years does not exceed 365 days for these subjects. Note: there were four subjects where the study withdrawal or completion date was missing; for these subjects the study agent discontinuation date (IPDISCDT) was used as the last known alive date.

Using this censoring date, the total subject follow-up will be derived for each subject as:

• Subject follow-up (days) = (Censoring Date – Study Treatment Start Date +1)

The amount of subject follow-up contributing to each of the cumulative timepoints (by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up, by Year 5 follow-up) is described below. In order to account for a censoring date which is out of the correct range of study days for a particular year, the following derivation will be used:

| Study Year | Subject Follow-Up (days) |
|---|---|
| By Week 52 | Minimum (Censoring Date – Treatment Start Date + 1, 365) |
| By Year 2 Follow-Up | Minimum (Censoring Date – Treatment Start Date + 1, 730) |
| By Year 3 Follow-Up | Minimum (Censoring Date – Treatment Start Date + 1, 1095) |
| By Year 4 Follow-Up | Minimum (Censoring Date – Treatment Start Date + 1, 1460) |
| By Year 5 Follow-Up | Minimum (Censoring Date – Treatment Start Date + 1, 1825) |

Note: individual subjects will only be allowed to contribute a maximum of 365 days for each individual follow-up year, regardless of when the follow-up visit was performed.

Note: For each subject, subject follow-up for each time period is cumulative since study treatment start date. For example, 'by Year 2 follow-up' includes follow-up time during Year 1 and follow-up time during Year 2 (to a maximum of 730 days).

The subject follow-up days will be converted to years as follows:

• Subject follow-up (years) = subject follow-up (days) / 365.25

The total follow-up years will be calculated for each of the timepoints as the sum of the subject follow-up years for that timepoint for all subjects in the As-Treated population.

# 5.6.2.10. Follow-Up Adjusted Subject Incidence Rate per 100 Subject Years: Malignancy

New malignancies will be assigned to a timepoint (i.e. Week 52, Year 2, Year 3, Year 4 or Year 5) using the nominal visit where the malignancy was reported. The first timepoint a subject reports a new malignancy will be used in the calculations of follow-up adjusted subject incidence rate per 100 subject years. The cumulative number of subjects with new malignancies to each timepoint will be summarized and follow-up adjusted subject incidence rates calculated.

The follow-up adjusted subject incidence rate presented for each timepoint will be a cumulative follow-up adjusted subject incidence rate from study treatment start date to the appropriate follow-up period. The subject years will be the sum of subject years for all subjects to that timepoint (as described in Section 5.6.2.8).

$$\label{eq:ncidence_rate} \textit{Incidence Rate} = 100 \ \times \frac{\textit{Number of subjects with an event}}{\textit{Subject Years}}$$

# 5.6.2.11. Follow-Up Adjusted Event Rate per 100 Subject Years: Malignancy

Subjects may report more than one new malignancy.

New malignancies will be assigned to a timepoint (i.e. Week 52, Year 2, Year 3, Year 4 or Year 5) using the nominal visit where the malignancy was reported. All new malignancy events will be included in the calculation of follow-up adjusted event rate per 100 subject years. The cumulative number of new malignancy events to each timepoint will be summarized and follow-up adjusted event rates calculated.

The follow-up adjusted event rate presented for each timepoint will be a cumulative follow-up adjusted event rate from study treatment start date to the appropriate follow-up period. The subject years will be the sum of subject years for all subjects to that timepoint (as described in Section 5.6.2.9).

Event Rate = 
$$100 \times \frac{Number\ of\ Events}{Subject\ Years}$$

# 5.6.2.12. First Exposure to Commercial Benlysta (other than Study Treatment during Year 1)

The first exposure to commercial Benlysta (other than study treatment during Year 1) will be summarized. Date of first exposure to commercial Benlysta is recorded in the concomitant medications dataset. For each subject the earliest recorded date of first exposure to commercial Benlysta (other than study treatment during Year 1) will be derived. The study day of earliest date of first exposure to commercial Benlysta will be calculated:

Study Day of First Exposure to Commercial Benlysta = Date of Exposure – Treatment Start Date +1

First commercial Benlysta exposure will be assigned to a year using a 365-day calendar year as follows:

| Study Year | Study Day of First Exposure to Commercial Benlysta |
|------------------|----------------------------------------------------|
| Week 52 | Day 1 to Day 365 (inclusive) |
| Year 2 Follow-Up | Day 366 to Day 730 (inclusive) |
| Year 3 Follow-Up | Day 731 to Day 1095 (inclusive) |
| Year 4 Follow-Up | Day 1096 to Day 1460 (inclusive) |
| Year 5 Follow-Up | ≥ Day 1461 |

Note, this assignment of first exposure to commercial Benlysta means it is possible that a subject is first exposed to commercial Benlysta during a year for which they are not in the population subset (i.e. if the last follow-up visit was performed later than the planned study day, even if it was within the visit window +30 days).

## 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population summaries will be based on the As-Treated population, unless otherwise stated. Summaries will be presented by treatment group and overall.

The number and percentage of subjects at each follow-up visit will be summarized by treatment group and overall. Week 52 will summarize all subjects in the As-Treated population. Summaries of any Year 2 to 5 follow-up, Year 2 follow-up, Year 3 follow-up, Year 4 follow-up and Year 5 follow-up will include subjects in each of the As-Treated population subsets as appropriate.

Important protocol deviations relating to the Years 2 to 5 post-treatment follow-up period will be listed for subjects in the any Year 2 to 5 follow-up subset of the As-Treated population. Protocol deviations will not be assigned to a particular follow-up year, but instead data will be combined across the Years 2 to 5 follow-up period.

For the final Year 5 reporting, demographic and baseline characteristics (including baseline disease activity) will be summarized for subjects in the Year 5 follow-up subset of the As-Treated population. For the interim Year X reporting, demographic and baseline characteristics (including baseline disease activity) will be summarized for subjects in the Year X follow-up subset of the As-Treated population i.e. for Year 2 interim reporting then Year 2 follow-up population subset will be used, for Year 3 interim reporting the Year 3 follow-up population subset will be used, etc.

Descriptive statistics will be used to summarize the continuous demographic and baseline characteristics of age (years) and weight (kg). Counts and percentages of the following categorical demographic and baseline characteristics will be presented: country region/country, gender, Hispanic or Latino origin, age group ( $\leq$ 45 years, >45 – <65 years and  $\geq$ 65 years and then within this last group:  $\geq$ 65 – <75 years and  $\geq$ 75 years) and race (Black or Other; see Section 5.2).

The number and percentage of subjects reporting each race and racial combination will be summarized. For subjects who check more than one race category, the race hierarchy rule defined in Section 5.6.2.1 will apply for this summary. Note that this differs to the handling of the race categorization of Black vs Other which ignores the hierarchy rule.

A summary of baseline disease activity will be provided, including counts and percentages for screening SELENA SLEDAI category (≤9, ≥10), complement levels (Low, Not Low), anti-dsDNA (High, Not High), complement and anti-dsDNA (Low Complement and High Anti-dsDNA, Not (Low Complement and High Anti-dsDNA)), and univariate statistics for SLE disease duration (years), screening SELENA SLEDAI total score, and SLICC/ACR Damage Index.

Demographic and baseline characteristics (age, gender, ethnicity, weight, race [Black vs. Other]) will be listed by subject. Race as assigned using the hierarchy rule (Section 5.6.2.1) will be listed by subject. These listings will be produced for subjects in the any Year 2 to 5 follow-up population subset (for all reporting efforts).

# 6.2. Concomitant Medications (First exposure to commercial Benlysta, other than study treatment in Year 1)

The number of subjects who are exposed to commercial Benlysta (other than study treatment in Year 1) will be summarized by treatment group and overall. The earliest timepoint of exposure to commercial Benlysta (other than study treatment in Year 1) will be summarized and a data listing produced.

The number of subjects first exposed to commercial Benlysta will be summarized by year for subjects in the As-Treated population for: Week 52, Year 2 Follow-up, Year 3 Follow-up, Year 4 Follow-up, and Year 5 Follow-up. The denominator for each year will be subjects included in the relevant As-Treated population subset (i.e. Year 2 follow-up, Year 3 follow-up, Year 4 follow-up, Year 5 follow-up).

In addition, the cumulative number of subjects first exposed to commercial Benlysta will also be summarized by year. The denominator will be the number of subjects in the As-Treated population.

Summaries will be presented by treatment group and overall.

Note, these summaries only provide information on the number of subjects who received commercial Benlysta, there is no information available on duration of exposure.

Note, due to the assignment of Benlysta exposure to year periods using a 365-day calendar year, it is possible that a subject might be exposed to commercial Benlysta for a year in which they did not perform a follow-up visit i.e. a subject might be in the numerator but not in the denominator.

#### 7. SAFETY ANALYSES

The safety summaries will be based on the As-Treated population, unless otherwise specified. Summaries will be presented by treatment group and overall.

Only serious adverse events (SAEs) and adverse events of special interest (AESI) were collected during the Week 52 double-blind treatment period of the study. Serious adverse events and AESIs were not collected as part of the clinical database for the Years 2 to 5 post-treatment follow-up period, therefore no summaries of adverse event data will be produced.

Any serious adverse events reported via paper CRFs during the Years 2 to 5 post-treatment follow-up period will be reported from the GSK safety database as part of the Clinical Study Report (CSR), but no summaries or listings will be produced by the programming group (as this data does not form part of the clinical database).

# 7.1. All-Cause Mortality

Survival status and mortality will be summarized by nominal follow-up visit.

#### **Survival Status**

Survival status by follow-up year will be summarized by treatment group and overall. The number and percentage of subjects will be summarized at each follow-up year for the following categories: alive, deaths (including a breakdown of deaths where COVID-19 was the primary cause of death, per CMQ and Other Deaths for Years 3, 4 and 5 – see Section 5.6.2.4), lost-to-follow-up and withdrew consent. NOTE that the COVID-19 pandemic started after all subjects completed Week 52 and Year 2. Percentages for each follow-up year will be calculated from the number of subjects at the follow-up visit, defined as subjects included in the relevant As-Treated population subset (i.e. Year 2 follow-up, Year 3 follow-up, Year 4 follow-up, Year 5 follow-up).

An additional category 'Not completed' will be summarized for follow-up years, this includes subjects who had a subsequent follow-up visit with a non-missing survival status, but did not complete the survival status form at this visit.

For completeness, survival status at the Week 52 visit will also be presented in the same table, with categories of alive, dead, lost to follow-up and unattainable, using subjects in the As-Treated population as the denominator for percentages.

A listing of survival status by follow-up year will be presented, including first commercial Benlysta use.

# **Deaths by System Organ Class and Preferred Term**

A summary of deaths will be produced for each follow-up year separately (Years 2, 3, 4 and 5). For each follow-up year, the summary will include the number and percentage of subjects who died for each SOC, each PT, and overall; based on subjects in the associated year follow-up subset of the As-Treated population and deaths reported during that follow-up year.

By default, the deaths will be sorted by MedDRA SOCs, in descending order from the SOC with the highest total incidence (i.e., summed across all treatment groups) for any deaths within the class, to the SOC with the lowest total incidence. If the total incidence for any two or more SOCs is equal, the events will be presented in alphabetical order. Only SOCs with observed AE PTs will be presented. Repeat sort order for MedDRA PTs within each SOC.

# Cumulative Mortality and Follow-up Adjusted Incidence Rate

The cumulative number of subjects who have died by follow-up year will be summarized by treatment group and overall for i) all deaths, ii) Deaths where COVID-19 was the primary cause of death, per CMQ iii) Deaths excluding those where COVID-19 was the primary cause of death. The number of subjects who have died by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up and by Year 5 follow-up will be presented. The total subject follow-up years will be presented for each follow-up year by treatment group and overall. The follow-up adjusted subject incidence rate of deaths per 100 subject years will be presented for each follow-up year by treatment group and overall.

# 7.2. Malignancy

Malignancies will be summarized by nominal follow-up visit for each treatment group and overall.

#### **New Malignancy Percentages**

The number and percentage of subjects reporting new malignancies will be summarized at each follow-up year for the categories of: new malignancy, no new malignancy and not completed. Percentages for each follow-up visit will be calculated from the number of subjects at the follow-up visit, defined as subjects included in the relevant As-Treated population subset (i.e. Year 2 follow-up, Year 3 follow-up, Year 4 follow-up, Year 5 follow-up).

The additional category 'Not completed' will be summarized for follow-up years, this includes subjects who had a non-missing survival status at this visit or a subsequent follow-up year, but did not complete the new malignancy form at this visit.

For completeness, new malignancies at the Week 52 visit will also be presented in the same table, using subjects in the As-Treated population as the denominator for percentages.

A listing of new malignancies by follow-up year will be presented, including first commercial Benlysta use.

#### Malignancies by System Organ Class and Preferred Term

A summary of new malignancies will be produced for each follow-up year separately (Years 2, 3, 4 and 5). For each follow-up year, the summary will include the number and percentage of subjects with new malignancies for each SOC, each PT, and overall; based on subjects in the associated year follow-up subset of the As-Treated population and malignancies reported during that follow-up year.

By default, the malignancies will be sorted by MedDRA SOCs, in descending order from the SOC with the highest total incidence (i.e., summed across all treatment groups) for any malignancies within the class, to the SOC with the lowest total incidence. If the total incidence for any two or more SOCs is equal, the events will be presented in alphabetical order. Only SOCs with observed AE PTs will be presented. Repeat sort order for MedDRA PTs within each SOC.

# Cumulative Malignancies and Follow-up Adjusted Subject Incidence Rate

The cumulative number of subjects who have new malignancies by follow-up year will be summarized by treatment group and overall. A subject will be included using the first nominal visit a new malignancy is reported at. The number of subjects who have a new malignancy by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up and by Year 5 follow-up will be presented. The total subject follow-up years will be presented for each follow-up year by treatment group and overall. Subject follow-up years will be truncated at the date of first diagnosis for subjects who report as new malignancy (Section 5.6.2.8). The follow-up adjusted subject incidence rate of malignancy per 100 subject years will be presented for each follow-up year by treatment group and overall.

#### Follow-Up Adjusted Event Rate

In addition, as a subject may report more than one new malignancy the cumulative number of malignancy events will be summarized by treatment group and overall. A subject will be included using malignancies reported at all nominal visits. The cumulative number of events will be summarized by Week 52, by Year 2 follow-up, by Year 3 follow-up, by Year 4 follow-up and by Year 5 follow-up. The total subject follow-up years will be presented for each follow-up year by treatment group and overall. As this is an event rate, subject follow-up years will not be truncated at the date of diagnosis for subjects who report a new malignancy (Section 5.6.2.9). The follow-up adjusted event rate of malignancy per 100 subject years will be presented for each follow-up year by treatment group and overall.

## 8. REFERENCES

Buyon JP, Petri MA, Kim MY, et al. The Effect of Combined Estrogen and Progesterone Hormone Replacement Therapy on Disease Activity in Systemic Lupus Erythematosus: A Randomised Trial. Ann Internal Med. 2005;142(12 Pt 1):953-62.

Petri M, Kim MY, Kalunian KC, Grossman J, Hahn BH, Sammaritano LR, et al. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med. 2005;353:2550-8.

# 9. APPENDICES

# 9.1. Appendix 1: Countries by Region

| Country Canada USA US/Canada Argentina Brazil Chile Colombia Central America/South America/Mexico Mexico Peru Puerto Rico Australia Bulgaria |
|---|
| Argentina Brazil Chile Colombia Central America/South America/Mexico Mexico Peru Puerto Rico Australia Bulgaria |
| Brazil Chile Colombia Central America/South America/Mexico Mexico Peru Puerto Rico Australia Bulgaria |
| Chile Colombia Central America/South America/Mexico Mexico Peru Puerto Rico Australia Bulgaria |
| Colombia Central America/South America/Mexico Mexico Peru Puerto Rico Australia Bulgaria |
| Mexico Peru Puerto Rico Australia Bulgaria |
| Peru Puerto Rico Australia Bulgaria |
| Puerto Rico Australia Bulgaria |
| Australia<br>Bulgaria |
| Bulgaria |
| Croatia |
| Czech Republic |
| Estonia |
| Hungary |
| Israel |
| Italy |
| Lithuania |
| New Zealand |
| Norway Europe/Australia/Israel |
| Poland |
| Portugal |
| Romania |
| Russia |
| Serbia |
| Slovakia |
| Spain |
| Switzerland |
| Turkey |
| Ukraine |
| China |
| Hong Kong |
| India |
| Indonesia<br>Korea Asia |
| Malaysia Philippings |
| Philippines<br>Taiwan |
| Thailand |

# 9.2. Appendix 2: Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : us1salx00259 |
| HARP Compound | : gsk1550188/bel115467/ |
| | Note: each reporting effort will use a different reporting area. Year 2 interim will use safety_12, Year 3 interim will use safety_13. Other reporting efforts will be allocated when necessary. |
| Analysis Datasets | |
| Analysis datasets IG Version 1.1 | s will be created according to CDISC standards SDTM IG Version 3.1.2 & ADaM |
| • The version of the CDISC standards at the time of annual reporting/Year 5 database freeze (DBF) will be decided by the study team. | |
| Generation of RTF Files | |
| RTF files will be g | generated for the interim and final reporting efforts. |

# 9.3. Appendix 3: Abbreviations & Trade Marks

# 9.3.1. Abbreviations

| Abbreviation | Description |
|--------------|-----------------------------------------------------|
| ACR | American College of Rheumatology |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| Anti-dsDNA | Anti-double-stranded DNA |
| CDISC | Clinical Data Interchange Standards Consortium |
| CMQ | Custom MedDRA Query |
| COVID-19 | Coronavirus Disease 2019 |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DBF | Database freeze |
| DBR | Database release |
| eCRF | Electronic Case Report Form |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| II | Immuno-Inflammation |
| IM | Intramuscular(ly) |
| IP | Investigational Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NMSC | Non-melanoma skin cancer |
| PDMP | Protocol Deviation Management Plan |
| PSAP | Program Safety Analysis Plan |
| RAP | Reporting and Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SD | Standard deviation |
| SDAC | Statistical Data Analysis Center |
| SDTM | Study Data Tabulation Models |
| SELENA | Safety of Estrogen in Lupus National Assessment |
| SLE | Systemic Lupus Erythematosus |
| SLEDAI | Systemic Lupus Erythematosus Disease Activity Index |
| SLICC | Systemic Lupus International Collaborating Clinics |
| SRT | Safety Review Team |
| TLFs | Tables, Listings and Figures |

# 9.3.2. Trade Marks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| BENLYSTA |

| Trademarks not owned by the GlaxoSmithKline Group of Companies | <b>;</b> |
|----------------------------------------------------------------|----------|
| SAS | |

# 9.4. Appendix 4: List of Data Displays

# 9.4.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables |
|------------------|--------------|
| Study Population | 1.01 to 1.nn |
| Safety | 3.01 to 3.nn |
| Section | Listings |
| ICH Listings | 1 to x |
| Other Listings | y to z |

# 9.4.2. Deliverables

| Delivery | Description |
|---|---|
| IA SAC Interim Analysis Statistical Analysis Complete for Year 2, Year 3 & Yea | |
| SAC Final Statistical Analysis Complete for Year 5 | |

# 9.4.3. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition/Popu | ulations | | | |
| 1.1. | As-Treated | Table 1.01 | Number (%) of Subjects in Years 2-5 Post-treatment Follow-up | | IA SAC, SAC |
| Demog | raphic and Baseli | ne Characteris | tics | | |
| 1.2. | As-Treated<br>Year X Follow-<br>up | Table 1.02 | Summary of Demographic and Baseline Characteristics for Subjects with Year X Follow-up | Population dependent on the reporting effort year (e.g. at Year 2 reporting, use Year 2 follow-up population subset) | IA SAC, SAC |
| 1.3. | As-Treated<br>Year X Follow-<br>up | Table 1.03 | Summary of Race and Racial Combination Details for Subjects with Year X Follow-up | Population dependent on the reporting effort year (e.g. at Year 2 reporting, use Year 2 follow-up population subset) | IA SAC, SAC |
| 1.4. | As-Treated<br>Year X Follow-<br>up | Table 1.04 | Summary of Baseline Disease Activity for Subjects with Year X Follow-up | Population dependent on the reporting effort year (e.g. at Year 2 reporting, use Year 2 follow-up population subset) | IA SAC, SAC |
| Conco | Concomitant Medication (First exposure to commercial Benlysta, other than study treatment in Year 1) | | | | |
| 1.5. | As-Treated | Table 1.05 | Summary of Number of Subjects Exposed to Commercial Benlysta (Other than Study Treatment during Year 1) | | IA SAC, SAC |

# 9.4.4. Safety Tables

| Safety: | Safety: Tables | | | | | |
|---|---|---|---|---|---|--|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable | |
| Mortality | | | | | | |
| 3.1. | As-Treated | Table 3.01 | Survival Status for Years 2-5 Post-treatment Follow-up Period | | IA SAC, SAC | |
| 3.2. | As-Treated<br>Year 2<br>Follow-up | Table 3.02 | Summary of Deaths by SOC and PT -Year 2 Post-treatment Follow-up | | IA SAC, SAC | |
| 3.3. | As-Treated<br>Year 3<br>Follow-up | Table 3.03 | Summary of Deaths by SOC and PT -Year 3 Post-treatment Follow-up | | IA SAC, SAC | |
| 3.4. | As-Treated<br>Year 4<br>Follow-up | Table 3.04 | Summary of Deaths by SOC and PT -Year 4 Post-treatment Follow-up | | IA SAC, SAC | |
| 3.5. | As-Treated<br>Year 5<br>Follow-up | Table 3.05 | Summary of Deaths by SOC and PT -Year 5 Post-treatment Follow-up | | IA SAC, SAC | |
| 3.6. | As-Treated | Table 3.06 | Summary of Cumulative Mortality Rate by Follow-up Year | | IA SAC, SAC | |
| 3.7. | As-Treated | Table 3.07 | Summary of Cumulative Mortality Rate by Follow-up Year (<br>Deaths where COVID-19 was the Primary Cause of Death) | | IA Y3, 4, 5<br>SAC, SAC | |
| 3.8. | As-Treated | Table 3.08 | Summary of Cumulative Mortality Rate by Follow-up Year (Excluding Deaths where COVID-19 was the Primary Cause of Death) | | IA Y3, 4, 5<br>SAC, SAC | |
| Malignancy | | | | | | |
| 3.9. | As-Treated | Table 3.09 | Summary of Subjects with New Malignancies for Years 2-5 Post-treatment Follow-up Period | | IA SAC, SAC | |
| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.10. | As-Treated<br>Year 2<br>Follow-up | Table 3.10 | Summary of New Malignancies by SOC and PT -Year 2 Post-treatment Follow-up | | IA SAC, SAC |
| 3.11. | As-Treated<br>Year 3<br>Follow-up | Table 3.11 | Summary of New Malignancies by SOC and PT -Year 3 Post-treatment Follow-up | | IA SAC, SAC |
| 3.12. | As-Treated<br>Year 4<br>Follow-up | Table 3.12 | Summary of New Malignancies by SOC and PT -Year 4 Post-treatment Follow-up | | IA SAC, SAC |
| 3.13. | As-Treated<br>Year 5<br>Follow-up | Table 3.13 | Summary of New Malignancies by SOC and PT -Year 5 Post-treatment Follow-up | | IA SAC, SAC |
| 3.14. | As-Treated | Table 3.14 | Summary of Cumulative New Malignancy Rate by Follow-up Year | | IA SAC, SAC |

# 9.4.5. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell | | Title | Programming Notes | Deliverable |
| Subject | Subject Disposition | | | | |
| 1. | As-Treated | Listing 1 | Subject Disposition for Years 2-5 Post-treatment Follow-up Period | | IA SAC, SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Baselir | ne/Demographic | Characteristics | | | |
| 2. | As-Treated<br>Any Year 2<br>to 5 Follow-<br>Up | Listing 2 | Demographic and Baseline Characteristics | | IA SAC, SAC |
| 3. | As-Treated<br>Any Year 2<br>to 5 Follow-<br>Up | Listing 3 | Listing of Race | | IA SAC, SAC |
| Concor | mitant Medicati | on (First exposure | e to commercial Benlysta, other than study treatment in Year 1) | | |
| 4. | As-Treated | Listing 4 | Listing of Subjects Receiving First Commercial Benlysta including Week 52 and Years 2-5 Post-treatment Follow-up | | IA SAC, SAC |
| Safety | | | | | |
| 5. | As-Treated | Listing 5 | Listing of Survival Status for Years 2-5 Post-treatment Follow-up | | IA SAC, SAC |
| 6. | As-Treated | Listing 6 | Listing of Deaths for Years 2-5 Post-treatment Follow-up | | IA SAC, SAC |
| 7. | As-Treated | Listing 7 | Listing of Subjects with New Malignancies for Years 2-5 Post-treatment Follow-up | | IA SAC, SAC |
| Protoc | Protocol Deviations | | | | |
| 8. | As-Treated<br>Any Year 2<br>to 5 Follow-<br>Up | Listing 8 | Listing of Important Protocol Deviations for Years 2-5 Post-treatment Follow-up Period | ICH E3 | IA SAC, SAC |

# 9.5. Appendix 5: Example Mock Shells for Data Displays

See separate Mock Shell TFL document.

### The GlaxoSmithKline group of companies

**Division:** World Wide Development

**Retention Category:** GRS019

Information Type: Reporting and Analysis Plan

**Title:** Reporting and Analysis Plan (RAP) for BEL115467, A

Randomized, Double-Blind, Placebo-Controlled 52-Week Study to Assess Adverse Events of Special Interest in Adults with Active, Autoantibody-Positive Systemic Lupus Erythematosus

Receiving Belimumab

Compound Number: GSK1550188

**Effective Date:** 18-OCT-2018

**Description**: This is a global, multi-center, randomized, double-blind, placebo-controlled, 52-week study to assess mortality and adverse events of special interest in adults with active, autoantibody-positive systemic lupus erythematosus (SLE) receiving belimumab. Subjects will receive belimumab or placebo through Week 48 with a final visit conducted at Week 52 and standard therapy will be received throughout the study. Subjects will be assessed for malignancies including non-melanoma skin cancers (NMSC), serious infections, opportunistic infections and other infections of interest, selected serious psychiatric events, suicidality, and serious infusion and hypersensitivity reactions. All-cause mortality will be reported. All other serious adverse events regardless of causality will also be recorded. Efficacy endpoints are secondary in nature. Following the 52-week study, all subjects will be contacted annually through Year 5 to assess mortality and malignancy (including NMSC). This Reporting and Analysis Plan (RAP) prospectively describes the safety and efficacy analyses that will be performed through the Week 52 treatment period. Details of the planned summaries for the post-treatment follow-up for Years 2 to 5 will be described in a separate RAP.

**Subject:** Systemic Lupus Erythematosus, SLE, belimumab, GSK1550188, Benlysta, efficacy, safety, placebo, mortality, adverse events of special interest.

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## Author's Name, Title and Functional Area:

| Statistics Leader<br>Clinical Statistics | Date: 18-OCT-2018 |
|-------------------------------------------------------|-------------------|
| Approved by: | |
| PPD | Date: 17-OCT-2018 |
| Senior Statistics Director | |
| Clinical Statistics | |
| PPD | Date: 18-OCT-2018 |
| Programming Manager | |
| Clinical Programming | |
| PPD | Date: 17-OCT-2018 |
| Director, Clinical Programming | |
| Clinical Programming | |
| PPD | D 17.00T 2010 |
| | Date: 17-OCT-2018 |
| Clinical Development Director<br>Clinical Development | |
| Clinical Development | |
| PPD MD | Date: 18-OCT-2018 |
| Clinical Development Director | 2010 |
| Clinical Development | |

## The GlaxoSmithKline group of companies

Safety and Medical Governance

| Global Clinical Development Manager Global Clinical Sciences and Operations | <b>Date:</b> 18-OCT-2018 |
|---|---|
| PPD | D |
| Manager, Clinical Data Management Clinical Data Management | <b>Date:</b> 18-OCT-2018 |
| PPD | <b>Date:</b> 18-OCT-2018 |
| Medical Writing & Clinical Submission Planning Manager Medical Writing | |
| PPD | <b>Date:</b> 18-OCT-2018 |
| Senior Director, Global Regulatory Affairs<br>Global Regulatory Affairs | |
| PPD | <b>Date:</b> 18-OCT-2018 |
| SERM Senior Director | |

## **TABLE OF CONTENTS**

| | | F | AGE |
|---|---|---|---|
| ABI | BREVIA | ATIONS | 7 |
| 1. | INTRO | DDUCTION | 9 |
| 2. | CTLID | Y OBJECTIVES AND ENDPOINTS | 0 |
| ۷. | 2.1. | Study Objectives | |
| | 2.1. | Study Endpoints | |
| | ۷.۷. | 2.2.1. Safety Endpoints | |
| | | 2.2.2. Efficacy Endpoints | |
| | | 2.2.3. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.3. | Statistical Hypotheses | |
| 3. | STUD | Y DESIGN | 12 |
| 4. | | NED ANALYSES | 10 |
| 4. | 4.1. | Interim Analyses | |
| | 4.1. | Final Analysis | |
| | 1.2. | Tindi / tidiyolo | |
| 5. | SAMP | LE SIZE CONSIDERATIONS | 14 |
| | 5.1. | Sample Size Assumptions | 14 |
| 6. | ΔΝΔΙΝ | YSIS POPULATIONS | 14 |
| Ο. | 6.1. | Analysis Datasets | |
| | | , | |
| 7. | TREAT | TMENT COMPARISONS | |
| | 7.1. | Data Display Treatment and Other Subgroup Descriptors | 15 |
| 8. | GENE | RAL CONSIDERATIONS FOR DATA ANALYSES | 16 |
| | 8.1. | Multicenter Studies | |
| | 8.2. | Other Strata and Covariates | 17 |
| | 8.3. | Examination of Subgroups | 17 |
| | 8.4. | Multiple Comparisons and Multiplicity | 18 |
| 9. | DATA | HANDLING CONVENTIONS | 18 |
| | 9.1. | Study Periods | |
| | | 9.1.1. Treatment Period (to Week 52) | |
| | | 9.1.2. Post-Treatment Follow-Up | |
| | 9.2. | GSK Adjudication of Death Categories and AESI | 20 |
| | 9.3. | Hospitalizations Review | |
| | 9.4. | Premature Withdrawal and Missing Data | |
| | | 9.4.1. Premature Withdrawal from 'IP only' Prior to Week 52 | |
| | | 9.4.2. Withdrawal from Study Prior to Week 52 | |
| | 0.5 | 9.4.3. Missing Data | |
| | 9.5. | Derived and Transformed Data | |
| | | 9.5.1. Baseline | |
| | | 9.5.2. Study Day | |
| | | 9.5.4. Subject Years of Follow-Up to Week 52 | |
| | | 9.5.5. Change from Baseline | |


BEL115467

| | | 9.5.6. | Percent Change from Baseline | 27 |
|---|---|---|---|---|
| | | 9.5.7. | Treatment Completer | 2 <mark>7</mark> |
| | | 9.5.8. | Study Completer | 27 |
| | | 9.5.9. | Analysis Age | 27 |
| | | 9.5.10. | Race Hierarchical Rule | 28 |
| | | 9.5.11. | SLE Disease Duration | 28 |
| | | 9.5.12. | Mortality and Protocol-Defined AESI | 28 |
| | | 9.5.13. | Treatment-Emergent AEs and AE Duration | 29 |
| | | 9.5.14. | Incidence Rate | 30 |
| | | 9.5.15. | Treatment-Emergent C-SSRS | 31 |
| | | 9.5.16. | Prednisone | 32 |
| | | | 9.5.16.1. Average Daily Prednisone Equivalent | |
| | | | 9.5.16.2. Average Daily Prednisone Dose during Weeks | |
| | | | 40 to 52 | 33 |
| | | | 9.5.16.3. Cumulative Prednisone Dose | 33 |
| | | 9.5.17. | Immunomodulatory Medications | 34 |
| | | 9.5.18. | Baseline Allowable SLE Medications | |
| | | 9.5.19. | SLICC/ACR Scoring | |
| | | | <b>C</b> | |
| 10. | STUD | Y POPUL | ATION | 35 |
| | 10.1. | Dispositi | ion of Subjects | 35 |
| | 10.2. | | Deviations | |
| | 10.3. | Demogra | aphic and Baseline Characteristics | 37 |
| | 10.4. | Concom | itant Medications | 40 |
| | 10.5. | Extent of | f Exposure | 40 |
| 11. | PRIMA | | OTHER SAFETY ANALYSES | |
| | 11.1. | Primary | Analysis: All-Cause Mortality, AESI and SAEs | |
| | | 11.1.1. | <b>,</b> | |
| | | 11.1.2. | | |
| | | 11.1.3. | SAEs | 44 |
| | 11.2. | Other Sa | afety Summaries | 44 |
| | | 11.2.1. | AESI and SAEs | 44 |
| | | 11.2.2. | Deaths and Serious Adverse Events | 47 |
| | | 11.2.3. | AESIs and SAEs Leading to Discontinuation of | |
| | | | Investigational Product or Withdrawal from Study | 48 |
| | | 11.2.4. | PSAP-Defined Adverse Events of Special Interest | |
| | | | 11.2.4.1. Post-infusion Systemic Reactions | 50 |
| | | 11.2.5. | Columbia-Suicide Severity Rating Scale (C-SSRS) | |
| | | | 11.2.5.1. C-SSRS Suicidal Ideation or Behavior | 51 |
| | | | 11.2.5.2. C-SSRS Suicidal Ideation or Behavior Relative | |
| | | | to Pre-Treatment | 51 |
| | | | 11.2.5.3. C-SSRS Shift Changes in Categories from Pre- | |
| | | | Treatment to On-Treatment | 5 <mark>2</mark> |
| 12. | EFFIC | | ALYSES | |
| | 12.1. | Major Ef | ficacy Analyses | 52 |
| | | 12.1.1. | Percent of Subjects with Prednisone Reduction by ≥25% | |
| | | | from baseline to ≤7.5 mg/day during Week 40 through | |
| | | | Week 52 | |
| | 12.2. | | ficacy Analyses | |
| | | 12.2.1. | Immunomodulatory Agents to Treat SLE | <mark>5</mark> 3 |


| | 445405 |
|-----|---------|
| BEL | .115467 |

| | 12.2.2 | . Hospitaliz | ations | 54 |
|---|---|---|---|---|
| | 12.2.3 | | CR Damage Index | |
| | | | SLICC/ACR Damage Index Change from | |
| | | | Baseline at Week 52 | 54 |
| | | 12.2.3.2. | SLICC/ACR Damage Index Worsening at | |
| | | | Week 52 | 54 |
| 13. | PHARMACO | SENETIC DA | TA ANALYSES | 55 |
| 14. | REFERENCE | S | | 56 |
| 15. | <b>APPENDICES</b> | 3 | | <mark>57</mark> |
| | 15.1. Appen | dix 1: Countr | ies by Region | <mark>57</mark> |
| | 15.2. Appen | dix 2: SELEN | NA SLEDAI Organ System Domains | 58 |
| | 15.3. Appen | dix 3: SLE Al | llowable Medication Categories | 59 |
| | 15.4. Appen | dix 4: Predni | sone Equivalent Conversion | 60 |
| | 15.5. Appen | dix 5: SLICC | ACR Damage Index | 63 |
| | 15.6. Appen | dix 6: PSAP | Sections for AESI Reporting | 65 |
| | 15.7. Appen | dix 7: Mortali | ty Missing Data Exploratory Sensitivity Analyses | 77 |
| | 15.7.1 | . Estimand | Framework | 77 |
| | | 15.7.1.1. | Main Estimand: While On Treatment | 77 |
| | | 15.7.1.2. | Supplemental Estimand: While On Study | 78 |
| | | 15.7.1.3. | Supplemental Estimand Sensitivity: Treatment | |
| | | | Policy | 79 |
| 16. | | | | |
| | | | or Data Display Specifications | |
| | 16.2. Data I | Display Speci | fications | 81 |
| | 16.3. Headli | ne Results | | 81 |
| | 16.4. Disclo | sure Outputs | | 82 |

### **ABBREVIATIONS**

ACR American College of Rheumatology

ADaM Analysis Data Model

AE Adverse Event

AESI AEs of special interest Anti-dsDNA Anti-double-stranded DNA

ATC Anatomical Therapeutic Chemical

AUC Area under the curve

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval
CIL Clinical investigative lead
CMQ Customized MedDRA Query

CRF Case Report Form

C-SSRS Columbia Suicide Severity Rating Scale

DBF Database freeze
DBR Database release

eCRF Electronic Case Report Form
EMA European Medicines Agency
GCP Good Clinical Practice

IDMC Independent Data Monitoring Committee

IDSL Integrated Data Standards Library

IM Intramuscular(ly)
IP Investigational Product
ITT Intention-to-treat
IV Intravenous(ly)

IXRS Interactive response system

MedDRA Medical Dictionary for Regulatory Activities

MM Medical monitor

NMSC Non-melanoma skin cancer NTM Non-tuberculous mycobacterium PSAP Program Safety Analysis Plan

PSRO Possible Suicidality Related Ouestionnaire

PT Preferred Term

RAP Reporting and Analysis Plan
SAC Statistical Analysis Complete

SAE Serious Adverse Event
SC Subcutaneous(ly)
SD Standard deviation

SDAC Statistical Data Analysis Center SDTM Study Data Tabulation Models

SELENA Safety of Estrogen in Lupus National Assessment

SLE Systemic Lupus Erythematosus

SLEDAI Systemic Lupus Erythematosus Disease Activity Index SLICC Systemic Lupus International Collaborating Clinics

SOC System Organ Class SRT Safety Review Team

TB Tuberculosis


BEL115467

Tables, Listings and Figures Worst Observation Carried Forward TLFs

WOCF

## **Trademark Information**

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| group of companies |

BENLYSTA

Trademarks not owned by the GlaxoSmithKline group of companies

SAS

### 1. INTRODUCTION

This reporting and analysis plan (RAP) documents the planned summaries through the Week 52 treatment period for the HGS1006-C1113 study. The study will be reported under its GSK study number BEL115467. A separate RAP will be produced to document the planned summaries of the post-treatment follow-up for Years 2 to 5.

This is a global, multi-center, randomized, double-blind, placebo-controlled, 52-week study to assess mortality and adverse events of special interest (AESI) in adults with active, autoantibody-positive systemic lupus erythematosus (SLE) treated with belimumab plus standard therapy vs placebo plus standard therapy. Following the 52-week study, all subjects will be contacted annually through Year 5 (Week 260) to assess mortality and malignancy (including non-melanoma skin cancers [NMSC]).

This RAP is based upon the following study documents:

- Study Protocol Amendment 03 (May 22, 2017)
- Final Case Report Form (CRF) Version 6.4 (February 05, 2018)
- Program Safety Analysis Plan (PSAP) Version 6 (October 2, 2018).
   Note: for reporting purposes, the most current version of the PSAP at the time of database freeze (DBF) will be used. For reference, sections of the PSAP that are relevant to reporting are given in Appendix 6: PSAP Sections for AESI Reporting. The most current MedDRA version at the time of database freeze (DBF) will be used.

### 2. STUDY OBJECTIVES AND ENDPOINTS

## 2.1. Study Objectives

To evaluate the following in adult SLE subjects receiving belimumab plus standard therapy versus subjects receiving placebo plus standard therapy:

- Mortality and adverse events of special interest (AESI) over 1 year (through 52 weeks).
- Corticosteroid reduction during Weeks 40-52.

## 2.2. Study Endpoints

## 2.2.1. Safety Endpoints

- All-cause mortality
- Serious infections (including serious opportunistic infections and any event of TB or TB reactivation)
  - See clarification in Section 2.2.3 (this endpoint will be referred to in the RAP as Serious Infections)

- Non-serious opportunistic infections and other infections of interest (protocol Appendix 2)
  - See clarification in Section 2.2.3 (this endpoint will be referred to in the RAP as Opportunistic Infections and Other Infections of Interest)
- Non-melanoma skin cancers (NMSC)
- Malignancies (excluding NMSC)
- Psychiatric events suggesting serious mood disorders and anxiety
- Suicidality (using C-SSRS; see protocol Appendix 4 and Appendix 5)
- Serious infusion and hypersensitivity reactions
- All serious adverse events (SAEs)

Section 9.5.12 provides definitions for all the protocol-defined AESIs. Section 2.2.3 provides the rationale for cases in which these may differ from the protocol.

## 2.2.2. Efficacy Endpoints

The major efficacy endpoint is:

• Percent of subjects whose average prednisone (or equivalent) dose has been reduced by ≥25% from baseline to ≤7.5 mg/day during Weeks 40 through 52 in subjects receiving greater than 7.5 mg/day at baseline.

Other efficacy endpoints include:

- Use of immunomodulatory medications to treat SLE.
- Number of hospitalizations per patient.
- Percent of patients hospitalized.

Systemic Lupus International Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index will be recorded at baseline and at Week 52 to permit assessment of accrual of damage in subjects who may be followed in a subsequent study.

Section 2.2.3 provides the rationale for cases in which these may differ from the protocol.

## 2.2.3. Changes to the Protocol Defined Statistical Analysis Plan

Changes/clarifications from the original planned summaries specified in the protocol are as follows:

• Whilst the protocol description of the AESI for serious infections was stated to include "any event of TB or TB reactivation", this has been defined in the RAP as All Serious Infections from the MedDRA 'Infections and Infestations' System Organ Class (SOC) aligned with the focus on serious infections. Hence any non-serious events, including those of 'TB or TB reactivation', would not be included in the endpoint but will be summarized separately.

- Whilst the protocol description of the AESI "Non-serious opportunistic infections and other infections of interest" refers to only non-serious events, the main summary will be of overall incidence (i.e., serious and non-serious events) aligned with focusing on all events of opportunistic infections and other infections of interest. Supplemental summaries of study agent related non-serious events will be produced, which will include non-serious opportunistic infections and other infections of interest. The endpoint will be derived using the "All infections" definition from the PSAP, Section 16.3 (See Appendix 6: PSAP Sections for AESI Reporting). This definition encompasses all infections of interest as defined in protocol Appendix 2. See Section 9.5.12.
- For the mortality endpoint, the protocol specifies that a hazard ratio (and 95% confidence interval [CI]) for belimumab vs placebo will be estimated using a Cox Proportional Hazards model. However due to the small number of events and low incidence rate, estimation using a difference in rates (and 95% CI) is considered more informative and so this supplemental analysis will not be conducted. A Kaplan-Meier curve and cumulative mortality counts by visit will be generated to illustrate the time profile.
- For the major efficacy endpoint (steroid dose reduction), the protocol states that if a subject switches immunomodulatory medications for reasons other than toxicity or lack of availability they should be considered a non-responder. However, the eCRF has not been designed to collect data on reasons for switches and therefore all new immunomodulatory agents to treat SLE will render a subject a non-responder in the analysis. Hence, subjects who switch will be considered non-responders regardless of the reason for switching. Additionally prednisone analyses and summaries are based only on steroids used to treat SLE (see Section 9.5.16 and Section 12.1.1).
- "Immunomodulatory medications" will be identified as immunosuppressants (ATC code beginning "L04A") plus cyclophosphamide and mercaptopurine, per the definition used across the Benlysta program.
- The number of hospitalizations per patient and percent of patients hospitalized will be derived from the SAE data. See Section 9.3 for further detail.
- SLICC/ACR Damage Index is not explicitly stated as an endpoint in the protocol. However, this is an endpoint of interest and therefore analyses will be performed as described in Section 12.2.3.

## 2.3. Statistical Hypotheses

There are no formal statistical hypotheses for the primary safety endpoints in the study. The main purpose of this study is to provide an evaluation of the difference in the rates of all-cause mortality and all prespecified AESI between the belimumab and placebo groups with a 2-sided 95% CI. SAEs will be summarized descriptively only. See Section 11.1.2 for details of the protocol-defined AESIs.

### 3. STUDY DESIGN

This is a global, multi-center, randomized, double-blind, placebo-controlled, 52-week study to assess mortality and AESI in adults with active, autoantibody-positive SLE treated with belimumab plus standard therapy vs placebo plus standard therapy. Approximately 4,000 subjects will be randomized (1:1) to belimumab plus standard therapy or placebo plus standard therapy. Randomization will be stratified for region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia; see Appendix 1: Countries by Region for details of countries and regions), Safety of Estrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) score (≤9 vs ≥10), and steroid dose (≤7.5 mg/day vs >7.5 mg/day prednisone or equivalent). There is no minimum score required for the SELENA SLEDAI to be eligible for this study.

Subjects will receive investigational product (IP) on Days 0, 14, 28, and every 28 days thereafter through Week 48 with a final in clinic visit conducted at Week 52. Subjects who discontinue treatment at any time during the study but do not withdraw from study visits will be followed at 28-day intervals through Week 52. If the subject withdraws from study visits prior to Week 52, an attempt will be made to assess mortality and occurrence of malignancy (including NMSC) at Week 52 and annually for Years 2 through 5. See protocol Section 3.1 for further details. If a subject is not contactable (withdrew consent or lost to follow-up), where allowed by individual subject's legal consent status and individual country regulations, sites may utilize other available records to perform a mortality assessment at Week 52 - this may include search of public records aided by an independent party.

An Independent Data Monitoring Committee (IDMC) will review unblinded safety data until the data are locked and analyzed. The IDMC will monitor all SAEs (including all-cause mortality), serious infections, opportunistic infections and other infections of interest, malignancies (including NMSC), selected serious psychiatric events, suicidality and serious infusion and hypersensitivity reactions. Details of the summaries provided to the IDMC by an Independent Statistical Data Analysis Center (SDAC) are described in the IDMC Charter and IDMC Report Template.

## 4. PLANNED ANALYSES

### 4.1. Interim Analyses

The EMA requested that an interim analysis be carried out for monitoring patients' safety.

An interim analysis was planned to be conducted when at least 2,000 randomized subjects had completed through Week 52. The database was released when individual subject records for all subject visits that occurred within the timeframe of the Week 52 visit of the 2,000<sup>th</sup> subject had been locked. Therefore, the interim analysis also included data for subjects who were randomized but had not yet completed Week 52.

The interim analysis was solely for monitoring patients' safety and reporting event rates to health authorities. It was descriptive in nature and no comparative statistical inferences for claims were to be made.

To minimize bias and maintain data integrity the interim analysis was performed by Statistics Collaborative Inc (SCI), an independent SDAC. They prepared the interim summaries and generated the interim report for IDMC review, producing the same summaries as those created for bi-annual IDMC reviews.

This interim analysis was conducted as planned and submitted to EMA in December 2016.

Following the final analysis of the treatment period through Week 52 as described in Section 4.2, interim summaries will be generated to report post-treatment follow-up mortality and malignancy rates at the end of Year 2, Year 3, and Year 4 for reporting to health authorities.

## 4.2. Final Analysis

There will be two database releases corresponding to the end of the following study periods as described in Section 9.1.1 and Section 9.1.2:

- Treatment Period (through Week 52)
- Post-Treatment Follow-Up (Years 2 to 5)

The first database release will occur after data through the Week 52 visit (occurring approximately 4 weeks after the last dose of study agent) for all subjects have been collected, verified and validated. Data for subjects who withdraw from IP but stay in the study through Week 52 will be included in this database release. This database will include Year 1 survival status and occurrence of malignancy for subjects who withdraw from the study prior to the Week 52 visit and have follow-up mortality and malignancy data at Week 52. Data for the Years 2 to 5 post-treatment follow-up that has been obtained to this point will be included in the first database release but these data will not be fully validated or locked and will not be reported unless otherwise specified.

The second database release will occur after data through the Year 5 survival status and occurrence of malignancy follow-up have been collected, verified and validated.

This RAP details the planned summaries through the Week 52 treatment period. All outputs required for the Treatment Period (through Week 52) will be listed in the Mock Tables, Listings and Figures (TLFs) Shells document. A separate RAP will be produced to document the planned summaries of the post-treatment follow-up for Years 2-5.

### 5. SAMPLE SIZE CONSIDERATIONS

## 5.1. Sample Size Assumptions

It was originally planned that a target of 5,000 SLE subjects would be enrolled in this safety study. The sample size was based on the feasibility of enrolling a large number of SLE subjects in a global trial that would provide a reasonable estimate for mortality and other AESI rates. Assuming a common first year mortality rate of 0.68% for both treatment groups, the precision of the 95% CI for the difference between treatment groups is  $\pm 0.46\%$ .

Following the completion of 2 additional placebo-controlled trials (BEL112341/C1115, BEL113750), revised mortality estimates based on data from all 5 of the completed studies were as follows: 0.504% (6/1,190 for the placebo group) and 0.564% (14/2,484 for the belimumab group) with a delta of 0.060%.

Using a conservative revised mortality rate of 0.564%, the 95% CI for a 4,000-subject sample size with 1:1 randomization was also  $\pm 0.46\%$ . As a result, given the revised mortality estimate, a sample size of 4,000 subjects would not result in any loss of precision (i.e., the width of the 95% CI remains unchanged). Therefore, agreement was reached with regulatory authorities to reduce the sample size from 5,000 to 4,000 subjects.

All sample size calculations were performed using the Chi-Square Simple Asymptotic Pearson method in Power Analysis and Sample Size software (PASS 2012).

### 6. ANALYSIS POPULATIONS

### Randomized

The Randomized population is defined as all subjects who are randomized. Summaries using the Randomized population will group subjects according to the treatment that a subject was randomized to receive, regardless of the actual treatment received.

Any subject assigned a treatment randomization number by the Interactive Response System (IXRS) system is considered to have been randomized.

One subject was randomized in the IXRS system but was not entered as a randomized subject into the eCRF, since the site had not administered study agent to the subject. It was not possible to subsequently update the randomization number into the eCRF because the site was closed. Therefore the subject cannot be included in the data displays as part of the randomized population. A footnote will be included on relevant tables to indicate this.

#### **Intention-to-Treat (ITT)**

The ITT population is defined as all subjects who are randomized and received at least one dose of study agent. The ITT analysis will be performed per the treatment that a

subject was randomized to receive, regardless of the actual treatment received. All efficacy endpoints will be analyzed using the ITT population unless otherwise specified.

#### **As-Treated**

The As-Treated population is defined as all subjects who are randomized and received at least one dose of study agent. The As-Treated population will group subjects according to the actual treatment administered to the subject based on the treatment that the subject received most of the time (>50% of the time). Therefore, if a subject received an incorrect treatment at more than half the visits, the As-Treated treatment group assignment will differ from the randomized treatment group assignment. Safety analysis will be performed on the As-Treated population.

Note: Two investigative sites (PPD and PPD ) were investigated for potential GCP non-compliance. These sites were closed during the conduct of the study. The data from both these sites will be included in all analyses/summaries since the primary endpoint and several of the secondary endpoints relate to safety and there were no concerns noted with the AE data. Also, in view of the large total sample size, inclusion of data from these sites (N=14 and N=4 at PPD and PPD in the As Treated population, respectively) is not considered to impact the overall study conclusions.

## 6.1. Analysis Datasets

All safety summaries will use the observed data, which are the data collected or observed for the subject with no imputation for missing data. Summaries may also include data as adjudicated by the safety review team (SRT) and/or clinical team where specified (see Section 9.2 and Section 9.3 for detail). See Section 9.5.16 for imputation rules for steroid reduction.

### 7. TREATMENT COMPARISONS

The difference in the rates of all protocol-defined AESI and all-cause mortality, between the belimumab and the placebo groups will be evaluated with a 2-sided 95% CI.

## 7.1. Data Display Treatment and Other Subgroup Descriptors

The following treatment descriptors will be used on all data tabulations:

- Placebo
- Belimumab 10 mg/kg

For tables presenting baseline demographics and characteristics described in Section 10, the data will also be presented for all subjects using a Total column. Other subgroup descriptors will be described in more detail in Section 8.3.

### 8. GENERAL CONSIDERATIONS FOR DATA ANALYSES

- All data summaries and analyses will be performed using the latest available version of SAS software (as available at GSK).
- Data displays will follow the shells outlined in the Mock TLFs document which will follow the Benlysta program standards and, as far as possible, follow the agreements proposed by the GSK Integrated Data Standards Library (IDSL).
- The most current version of MedDRA at the time of DBF will be used for reporting.
- The most current version of the Benlysta PSAP at the time of DBF will be used for reporting.
- Where SDTM terminology differs from the eCRF and/or mock shells, the SDTM terminology will be presented in displays unless otherwise specified.

Unless otherwise stated, the following will apply:

- Continuous variables will be summarized with the statistics mean, median, standard deviation (SD), 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum.
- Categorical variables will be summarized with frequency counts and percentages, or proportions where specified. A 'Missing' category will be added to frequency counts if there is at least one missing record.
- Percentages will be calculated using the number of subjects in the relevant population/treatment group (denoted by N) as the denominator, unless otherwise stated.
- The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database.
- The mean, median, 25<sup>th</sup> percentile and 75<sup>th</sup> percentile will be reported to one more decimal place than the raw data recorded in the database.
- The SD will be reported to two more decimal places than the raw data recorded in the database.
- A maximum of four decimal places will be used.
- The same rules apply to scores calculated in the derived datasets.
- Percentages will be presented to one decimal place. Incidence rates and difference in incidence rates for the primary analyses will be presented to two decimal places.
- A count of zero will have no corresponding percentage.
- For statistical analyses, all tests will be two-sided and p-values will be presented to a maximum of 4 decimal places.
- Listings will be based on the Randomized population and generally be limited to those required by ICH guidelines and will be sorted by treatment group, investigator number, subject number and visit (where appropriate).

#### 8.1. Multicenter Studies

This is a multicenter trial and subjects will be centrally randomized by region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia – See Appendix 1). There will be no analyses performed at the center level.

Note that in this study, no subjects from Israel were randomized.

### 8.2. Other Strata and Covariates

In addition to randomization by region, randomization will include stratification by subjects' screening SELENA SLEDAI score ( $\leq 9$  vs.  $\geq 10$ ) and steroid dose ( $\leq 7.5$  mg/day vs  $\geq 7.5$  mg/day prednisone or equivalent). Any subgroup summaries (or analyses controlling for stratification factors as covariates, as applicable) will use data from the eCRF, not the strata variable from the randomization dataset.

Differences are anticipated between the randomization strata and the eCRF strata for baseline steroid dose. Sites were instructed to calculate the baseline dose for randomization using all steroids received for any indication (i.e. SLE and non-SLE). However, in the eCRF completion guidelines sites were instructed to record only steroids taken for SLE, pre-infusion (as prophylaxis against infusion reactions and hypersensitivity reaction), for AESI and SAEs in the eCRF. For subgroup summaries and for derivation as covariates (where used for analysis adjustment), only steroids received for SLE will be used to calculate baseline steroid dose. See Section 9.5.16 for details.

Other covariates of interest may include age, race, gender, complement levels and antidsDNA as defined in Section 8.3.

## 8.3. Examination of Subgroups

Since the reported incidence for primary safety endpoints is expected to be low, subgroup categories may be refined where necessary.

Mortality, AESIs and all AEs (i.e. AESI and SAEs) during the On-Treatment period will be summarized by the following subgroups:

- Age (<65 years vs.  $\ge 65$  years)
- Gender (Male vs. Female)
- Race Stratification (Black vs. Other). The Black category is defined as subjects who are in the race category "Black or African American". The race hierarchy rule (Section 9.5.10) will not apply and a subject will be categorized as Black if they have selected multiple race categories and any of them is "Black or African American".
- Randomization Stratification Factors (see Section 8.2, derived from eCRF data):
  - Region (US/Canada, Central America/South America/Mexico, Europe/Australia/Israel, Asia)
  - Screening SELENA SLEDAI ( $\leq 9, \geq 10$ ). Note: if any individual item is missing the total score cannot be calculated, however if the subject can be definitively

- categorized as  $\leq 9$  or  $\geq 10$  regardless of the response to the missing item(s) then the appropriate subgroup will be assigned.
- Steroid dose (≤7.5 mg/day, >7.5 mg/day prednisone or equivalent) (baseline average daily dose, see Section 9.5.16.1). Note: Only systemic steroids given for SLE are included in the derivation.
- Screening Complement Levels and Anti-dsDNA (Low Complement and High Anti-dsDNA binding, Not (Low Complement and High Anti-dsDNA binding)), derived from the screening SELENA SLEDAI assessment. This subgroup is intended to be an indicator of high versus low disease activity. Note: If the evaluations to the SELENA SLEDAI assessment questions "Low Complement" and "Increased DNA Binding" are both missing, the subject will not be classified into one of the subgroup categories. If either item is marked "No", the subject will be classified into the Not (Low Complement and High Anti-dsDNA binding) group regardless of whether the other item is missing or "Yes".

Demographic and baseline characteristics and baseline disease activity will also be summarized by all subgroups except Screening Complement Levels and Anti-dsDNA.

## 8.4. Multiple Comparisons and Multiplicity

There is no statistical hypothesis to be tested (no formal statistical testing) for the primary safety analyses, and therefore no need to control for multiple comparisons. Analyses of the secondary efficacy endpoints will also not be subject to any multiple comparison procedure. All statistical tests will be 2-sided and performed at an overall significance level of 0.05.

### 9. DATA HANDLING CONVENTIONS

This section describes data handling conventions including the study periods, handling of premature withdrawal and missing data and derived and transformed data.

## 9.1. Study Periods

The study has a Treatment Period (to Week 52) and a Post Treatment Follow-up (Years 2 through 5) as described below. Summaries of data collected during the latter will be defined in more detail in a separate RAP.

## 9.1.1. Treatment Period (to Week 52)

Subjects will receive IP through Week 48 with a final treatment period in clinic visit conducted at Week 52. Subjects who discontinue IP prior to Week 48 will have a follow-up in clinic visit performed approximately 4 weeks after the last dose of IP.

Per protocol, subjects may withdraw from IP during Year 1 and continue on study, or may withdraw from Year 1 study visits and reconsent to a Week 52 follow up. As a result, the time 'on treatment' versus the time 'on study' will differ for some subjects. Therefore, 2 analysis periods have been defined as the 'On-Treatment' and 'On-Study' periods. Further detail below.

The primary analysis summaries of Mortality, AESIs and SAEs will be performed using the 'On-Treatment' Period (defined in the table below).

Supportive summaries of the primary analysis will be performed using the 'On-Study' Period (includes on and off treatment data to Week 52).

For subjects who withdraw and reconsent for a Week 52 assessment only mortality and malignancy are assessed at Week 52, whereas all other endpoints will be assessed only up until the time of withdrawal. Therefore, in this case follow-up for mortality and malignancy will be longer than for other assessments.

| Study Period | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Study to<br>Week 52 | All data except Mortality and Malignancy events: Study Treatment Start Date ≤ Date ≤ minimum (Date of Death, maximum (Study Withdrawal or Completion Date (DSSTDT), Study Treatment Stop Date + 28 Days)) |
| | Mortality and all Malignancy events including NMSC (see Section 9.5.12 for definitions of mortality and malignancy events): |
| | Alive or Lost to Follow Up at Week 52 Follow-Up: Study Treatment Start Date ≤ Date ≤ minimum (Last Known to be Alive Date, Study Treatment Start date + 371) |
| | <ul> <li>Dead at Week 52 Follow-Up: Study Treatment Start Date ≤ Date of<br/>Death</li> </ul> |
| | <ul> <li>Week 52 follow-up missing: Study Treatment Start Date ≤ Date ≤ minimum<br/>(Date of Death, maximum (Study Withdrawal or Completion Date<br/>(DSSTDT), Study Treatment Stop Date + 28 Days))</li> </ul> |
| | Note: If the derived on-treatment period (i.e. study treatment stop date + 28 days) ends later than the derived on-study to Week 52 period, the derived on-study period will be updated such that it ends in line with the derived on-treatment period. |
| On-Treatment | All data: |
| | Study Treatment Start Date ≤ Date ≤ minimum (Date of Death, Study Treatment Stop Date + 28 days) |

Note: After study withdrawal or last exposure plus 28 days (whichever occurs later) if AESIs and SAEs are recorded, other than mortality and malignancy, these will not be included in the on-study period. See Section 11.2.1 for further detail on how these events will be handled.

Note: For mortality, date of death will be derived as the end date of the SAE with fatal outcome.

Note: Each study treatment infusion should have a start date and end date recorded, but in some cases only one variable is completed. The study treatment stop date is the date of the final study treatment infusion (taken as the first non-missing date of the final study treatment infusion start or end date).

Note: Only dates will be used to identify start and end of treatment (times will not be considered).

### 9.1.2. Post-Treatment Follow-Up

After the Treatment Period (to Week 52) all subjects will be contacted annually through Year 5 (Week 260) to assess mortality and malignancy (including NMSC). Annual follow-up also applies to subjects who discontinue IP before Week 48 and have remained in monthly follow-up and to subjects who withdraw consent from the study prior to Week 52 but re-consent for this annual follow-up.

## 9.2. GSK Adjudication of Death Categories and AESI

See Appendix 6: PSAP Sections for AESI Reporting for sections of the PSAP relating to death categories and AESI adjudication.

All fatalities (reported during the Week 52 study period) will be identified in the clinical database and subsequently adjudicated by the GSK SRT into a general category of death.

AESI are identified per the preferred terms and other criteria described in Appendix 6: PSAP Sections for AESI Reporting. Malignancies, serious post-infusion systemic reactions, potential opportunistic infections, suicidality and fatalities are adjudicated at the subject level by the GSK SRT. The adjudication occurs prior to database release and is performed for reporting purposes. Final confirmation of adjudications is required before database freeze (DBF).

## 9.3. Hospitalizations Review

A specific subject hospitalization form was not generated in the eCRF system for this study. Therefore, to measure all hospitalizations in this study, a manual clinical review process to identify the number of hospitalization events through review of all the SAEs has been implemented. The basis of this approach is that any event resulting in hospitalization mandates reporting as a SAE (refer to protocol Section 7.1).

#### Main review

The spreadsheet containing hospitalization data will be reviewed and updated in-stream and will be available for reporting. The summary of the process is presented below:

- 1. Clinical Programming will extract all SAEs from the eCRF into a spreadsheet listing for clinical review. Updates of SAE data will be extracted into the spreadsheet approximately every 4-6 weeks.
- 2. SAEs are reviewed by the study clinical investigation lead (CIL) and medical monitor (MM), or their equivalent designees. The reviewer determines the number of hospitalizations, and then assigns a hospitalization code for each hospitalization identified. The code consists of a combination of the Subject ID number and the hospitalization number for that subject (e.g., hospitalization code PPD = Subject ID and hospitalization PP).
- 3. In the absence of a 'reason for hospitalization' data field in the eCRF, to avoid the potential bias and/or influence of the Sponsor (GSK) in the determination of reason for hospitalization in any way, the SAE source verbatim term will be reported in the

- listing of hospitalizations and indicated as 'SAE(s) contributing to Hospitalization'. If more than one SAE is reported within the same hospitalization, all SAE source verbatim terms will be reported on the listing.
- 4. Once there are no outstanding issues after review of each SAE case (either after initial review, or after resolution of any queries), the review is then documented in the spreadsheet as completed with an initial and date by the reviewer. The spreadsheet is then reflected back into the ADaM datasets by Clinical Programming for reporting.

At any time, any SAEs from individual reviewers can be flagged for further team discussion / review to occur during ad hoc roundtable SAE review meetings, or by consult with the MM.

### Independent secondary review

In addition, a second independent review of the SAEs for the hospitalization events will be performed by an independent medical reviewer. The reviewer will be provided with the guidelines for review based on the protocol and following the same convention of the main review described above.

Once the review is completed, a comparison between the main review and the independent secondary review spreadsheets will be performed for the number of hospitalization and the assigned hospitalization code where applicable. Identified discrepancies will be discussed and reconciled at a round table meeting between the GSK clinical representatives (MM and study CIL or designee) and the independent medical reviewer. The reconciled records will be reflected on the main spreadsheet following the round table review meeting.

Full details of the hospitalizations review process will be documented as part of the Study Data Quality Plan and associated documents.

## 9.4. Premature Withdrawal and Missing Data

## 9.4.1. Premature Withdrawal from 'IP only' Prior to Week 52

Subjects who discontinue IP but do not withdraw from the study will continue the visit schedule through Week 52 and will be contacted annually for Years 2 through 5 to assess mortality and malignancy.

- All data collected through Week 52 post withdrawal from IP will be included in summaries unless otherwise specified.
- Annual assessment of mortality and malignancy will be included in the summaries of Year 2 to 5 (to be detailed in a separate RAP).

## 9.4.2. Withdrawal from Study Prior to Week 52

For subjects who withdraw from the study prior to Week 52, an attempt will be made to assess mortality and occurrence of malignancy (including NMSC) at Week 52 and annually for Years 2-5.

- For subjects who withdraw from the study, all data reported on the database will be used in the summaries through Week 52 unless otherwise specified.
- For subjects that withdraw early from Year 1 of the study, Week 52 mortality information will be collected if allowed by individual subject's legal consent status. This includes the potential use of a third party to aid sites in identifying information available from public sources.

## 9.4.3. Missing Data

## Adverse Events (AESIs, Serious Adverse Events) and Concomitant Medications

## **Missing Dates**

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listings. |
| Concomitant Medications | <ul> <li>Where medication start date (CMSTDT) is completely missing but medication end date (CMENDT) is on or after Day 1, the medication start date (CMSTDT) will be imputed as study treatment start date (TRTSDT).</li> <li>Where medication start date (CMSTDT) is completely missing and medication end date (CMENDT) is missing and the medication is ongoing (CMONGO = "Y"), the medication start date (CMSTDT) will be imputed as study treatment start date (TRTSDT) and the medication will be considered as ongoing.</li> <li>Medication End Date (CMENDT)</li> <li>Missing end dates for concomitant medications will not be imputed, and the medication will be considered ongoing.</li> <li>For corticosteroids, the medication end date will be imputed as study completion or withdrawal date during the ADPRED dataset creation in order for those medications to be included in prednisone summaries. However, if the start date of the medication is greater than the study completion or withdrawal date, the end date will not be imputed.</li> </ul> |
| Adverse<br>Events | The eCRF does not allow for the possibility of missing or partial AE dates (except for missing AE end dates which are allowed if the AE is ongoing). |

See Section 9.5.13 for further details on whether AE is considered as treatment-emergent.

Other than described above, missing data will not be imputed unless stated otherwise for an individual endpoint.

A missing category will be added to frequency counts if there is at least one missing record.

## **Partial Dates**

| Element | Reporting Detail |
|---|---|
| Date of | Only year of birth is collected on the eCRF. |
| Birth | • Day will be set to 30 and month will be set to JUNE for all subjects. |
| Concomitant<br>Medications | Medication Start Date (CMSTDT) Medication start date (CMSTDT) is imputed as study treatment start date (TRTSDT) unless: • CMENDT is < TRTSDT, whether CMENDT is complete (DD/MM/YY) or partial (some combination of CMENDT day, month or year imputed) OR |
| | The month or month and year of the partial CMSTDT are different from the month and/or year of TRTSDT OR |
| | • "Taken prior to study?" is checked. |
| | If any of the above conditions are met then medication start date (CMSTDT) is imputed with JAN for missing month and 01 for missing day, whatever is applicable. |
| | Medication End Date (CMENDT) |
| | If month and year are present, then: |
| | If the medication started on or after study withdrawal or completion then set to the last day of that month. |
| | If the medication started prior to study withdrawal or completion set to the last day of that month, unless the end month and year are the same as the month and year of the study withdrawal or completion date, in which case set to the study withdrawal or completion. date. |
| | <ul> <li>If only year present, then:</li> <li>if the medication started on or after study withdrawal or completion then set to 31DEC.</li> <li>if the medication started prior to study withdrawal or completion then set to 31DEC, unless the end year is the same as the year of</li> </ul> |
| | their set to 31DEC, timess the end year is the same as the year of the study withdrawal or completion date, in which case set to the study withdrawal or completion date. |
| Date of SLE diagnosis | • For records where month and day are missing for diagnosis date, impute with 01 for day and January for month to assume that the duration was the longest possible duration. |
| | • For records where the day only is missing for start date, impute with 01 for day to assume that the duration was the longest possible duration. |

| Element | Reporting Detail |
|---|---|
| Last known to be alive | • For records where month and day are missing for last known to be alive date, impute 01 for day and January for month. |
| date | For records where the day only is missing, impute 01 for day. |

#### 9.5. Derived and Transformed Data

#### 9.5.1. Baseline

The protocol specifies Day 0 as Baseline/Treatment Start date, but the CDISC standard is to refer to the Baseline/Treatment Start date as Day 1; therefore Baseline/Treatment Start date will be referenced as Day 1 in this document. A table indicating the target study day for each planned visit is in Section 9.5.3.

The baseline value of a variable is defined as the last available value measured prior to dosing on or before the date of first dose (Day 1), unless otherwise specified.

If the last available value occurs on Day 1 but the time of the assessment is not collected, then the assessment will be assumed to be prior to dosing. Noted exceptions to this rule are concomitant medications and AEs; these will be considered as being concomitant and treatment-emergent, respectively, if the start date occurs on the first day of dosing. However, if time is available for an AE or concomitant medication and the end time is earlier than the start time of first dose of IP, the AE or concomitant medication will not be considered as treatment-emergent or concomitant, respectively.

## 9.5.2. Study Day

Study Day is the number of days from the treatment start date to a study date of interest (e.g. event start date) and is calculated as follows:

| If condition is | Then Study Day is |
|---|---|
| study date <treatment date<="" start="" td=""><td>study date – treatment start date</td></treatment> | study date – treatment start date |
| study date is ≥treatment start date | study date – treatment start date +1 |

Note: Study Day cannot be zero. If either date is missing, then Study Day is missing.

### 9.5.3. Analysis Visit and Analysis Visit Number

Where applicable, the data are summarized per the planned visit assignment in the data. The visit windows below will be used to assign events to scheduled visits for tabular summaries of time to withdrawal from study, time to premature withdrawal from IP by clinical visit, cumulative time to mortality (On-Treatment Period) and cumulative time to mortality (On-Study Period).

| | Analysis | | Interval Start Day | Interval End Day |
|---|---|---|---|---|
| Analysis Visit | Visit Number | Target Study Day <sup>1</sup> | | • |
| Screening | 10 | -30 | Na | Na |
| Treatment Period visits: | | | | |
| Baseline | 25 | 1 | Na | Na |
| Week 2 | 30 | 15 | 1 | 15 |
| Week 4 | 40 | 29 | 16 | 29 |
| Week 8 | 50 | 57 | 30 | 57 |
| Week 12 | 60 | 85 | 58 | 85 |
| Week 16 | 70 | 113 | 86 | 113 |
| Week 20 | 80 | 141 | 114 | 141 |
| Week 24 | 90 | 169 | 142 | 169 |
| Week 28 | 100 | 197 | 170 | 197 |
| Week 32 | 110 | 225 | 198 | 225 |
| Week 36 | 120 | 253 | 226 | 253 |
| Week 40 | 130 | 281 | 254 | 281 |
| Week 44 | 140 | 309 | 282 | 309 |
| Week 48 | 150 | 337 | 310 | 337 |
| Week 52 | 160 | 365 | 338 | [2] |

<sup>&</sup>lt;sup>1</sup>Study Day with Baseline/Treatment Start Date as Day 1.

### 9.5.4. Subject Years of Follow-Up to Week 52

Start and end dates for study periods are defined in Section 9.1. For calculation of exposure adjusted incidence rates (during the on-treatment period) and study follow-up adjusted incidence rates (during the on-study period), the following will be derived (in years) for each subject. Additionally, for summaries of subject follow-up time, the off-treatment, missing and total possible follow-up will be derived in years.

Note: The On-Study (to Week 52) terminology reflects the intended duration of follow-up for mortality and AESIs during the main study (i.e. 52 weeks). Some subjects will have less than 52 weeks of follow-up (e.g. where the subject has died or withdrawn from the study). The terminology 'follow-up' has been used to describe the time periods during which subjects are followed up for event assessment during the main 1-year study and does not refer to the post-treatment follow-up period in Years 2-5 (described in Section 9.1.2).

#### On-Treatment Follow-Up: Mortality and Malignancy and Other Data

[(End Date for On-Treatment Period – Study Treatment Start Date) + 1]/365.25

### On-Study Follow-Up (to Week 52): Mortality and Malignancy

[(End Date of On-Study Period for Assessment of Mortality and Malignancy (to Week 52) – Study Treatment Start Date) + 1]/365.25

<sup>[2]</sup> Any events on or after Day 338 will be assigned to Week 52

#### On-Study Follow-Up (to Week 52): Other Data

[(End Date of Study Period for assessment of all data excluding mortality and malignancy (to Week 52) – Study Treatment Start Date) + 1]/365.25

#### Off-Treatment Follow-Up Time: Mortality and Malignancy

[(End Date for On-Study Period for Assessment of Mortality and Malignancy – [End Date for On-Treatment Period + 1]) + 1]/365.25

## Off-Treatment Follow-Up Time: Other Data

[(End Date for On-Study Period for assessment of all data excluding mortality and malignancy – [End Date for On-Treatment Period + 1]) + 1]/365.25

### Total Possible Follow-Up Time: Mortality and Malignancy

[(Possible Follow-Up Date – Study Treatment Start Date) + 1]/365.25

For subjects whose end of on-study period for mortality and malignancy is on or after Study Day 358 (lower allowable visit window for Week 52 assessment) the possible follow-up date will be assigned as the end date for the on-study period for assessment of mortality and malignancy.

For subjects whose end of on-study period for mortality and malignancy is before Study Day 358 (lower allowable visit window for Week 52 assessment) the possible follow-up date will be assigned as the minimum of Study Day 365 and date of death.

#### **Total Possible Follow-Up Time: Other Data**

[(Possible Follow-Up Date – Study Treatment Start Date) + 1]/365.25

For subjects whose end of on-study period for all data excluding mortality and malignancy is on or after Study Day 358 (lower allowable visit window for Week 52 assessment) the possible follow-up date will be assigned as the end date for the on-study period for assessment of all data excluding mortality and malignancy.

For subjects whose end of on-study period for all data excluding mortality and malignancy is before Study Day 358 (lower allowable visit window for Week 52 assessment) the possible follow-up date will be assigned as the minimum of Study Day 365 and date of death.

### Missing Follow-Up Time (Years): Mortality and Malignancy / Other Data

Total possible follow-up time – (on-treatment follow-up + off-treatment follow-up)

### 9.5.5. Change from Baseline

Change from baseline will be calculated as:

Visit value – baseline value.

If either value is missing the change from baseline will be missing.

### 9.5.6. Percent Change from Baseline

Percent change from baseline will be calculated as

If the baseline value is zero or missing, then the percent change should be set to missing.

### 9.5.7. Treatment Completer

A "treatment completer" is defined as a subject who does not discontinue study agent prematurely. Treatment completion date or treatment discontinuation date is defined using the date from SDTM.DS where DSSCAT='STUDY TREATMENT'. Treatment completion date is assigned for subjects who completed study treatment (DSDECOD='COMPLETED') and study treatment discontinuation date is assigned for subjects who did not complete study treatment (DSDECOD not missing and not equal 'COMPLETED').

## 9.5.8. Study Completer

A "study completer" is defined as a subject who does not withdraw from the study prior to Week 52. Data for 'study completers' can include off-treatment data for subjects who discontinue study agent but continue on the visit calendar for study assessments.

Note: Each subject should have a date of study withdrawal or completion. Study withdrawal or completion date is defined using the date from SDTM.DS where DSSCAT='STUDY CONCLUSION'. Study completion date is assigned for subjects who completed the study (DSDECOD='COMPLETED') and study discontinuation date is assigned for subjects who did not complete the study (DSDECOD not missing and not equal 'COMPLETED').

### 9.5.9. Analysis Age

Analysis age is derived in years relative to the treatment start date for randomized subjects, and is calculated in SAS as follows:

INTCK ('YEAR', Date of birth, Date of treatment start date, 'C').

For subjects who are randomized but do not receive study agent and therefore have no treatment start date, randomization date will be used instead.

#### 9.5.10. Race Hierarchical Rule

If multiple race categories are checked on the eCRF, the subject will be assigned to a unique race group based on which of the races checked appears first in the list below:

- Native Hawaiian or Other Pacific Islander
- American Indian or Alaska Native
- Asian
- Black or African American
- White

For example, if Black or African American and Asian are both checked, then the subject will be assigned as Asian since it appears highest in the list. In the race and racial combination details table, subjects with multiple race categories checked will be reported in the race per the hierarchical rule as well as in the multiracial category. Subjects who select more than one Asian category and no other non-Asian categories will be represented in the Mixed Asian Race category as well as the Asian category. Similarly, subjects who select both white categories and no non-white categories will be represented in the Mixed White Race category as well as the White/Caucasian category. The Mixed Asian Race and Mixed White Race categories will only appear in the table if a subject selects multiple Asian or multiple white categories, respectively.

For the Race subgroup, if a subject selects multiple races they will be assigned "Black" if any of the races is "Black or African American", i.e., the hierarchical rule will not apply in this instance (see Section 8.3).

#### 9.5.11. SLE Disease Duration

SLE Disease Duration is defined as

If either date is missing, then SLE Disease Duration will be missing. Partial dates for SLE diagnosis date will be imputed as described in Section 9.4.3.

## 9.5.12. Mortality and Protocol-Defined AESI

Mortality status will be derived from the SAE data, where outcome is fatal.

The derivation for the protocol-defined AESIs are provided in the table below. Treatment emergent AESIs (see Section 9.5.13 and Section 9.5.15) only will be summarized.

Where the protocol defined AESI utilize definitions from the PSAP, the detailed derivations from the PSAP are provided in Appendix 6: PSAP Sections for AESI Reporting. AESI are identified per the preferred terms and other criteria described in the PSAP.

| Protocol-Defined AESI<br>(see Section 2.2.1 and<br>Section 2.2.3 for<br>clarification) | Definition | Programming Derivation (Protocol Definition) |
|---|---|---|
| Serious infections | SAEs within Infections and Infestations SOC. | SOC=Infections and Infestations & AESER = 'Y' |
| Opportunistic infections and other infections of interest | "All Infections" per PSAP definition to cover all OI and infections of interest. | CQ06NAM ne " or<br>CQ07NAM ne " or<br>CQ08NAM ne " |
| Non-melanoma skin cancers (NMSC) | NMSC per PSAP definition. | CQ00MLFL = 'Y' and<br>CQ03NAM ne '' and<br>CQ03NMFL = 'Y' |
| Malignancies (excluding NMSC) | PSAP defined, "all malignancies excluding NMSC". | [CQ00MLFL = 'Y' and<br>(CQ01NAM ne " or<br>CQ02NAM ne " or<br>(CQ03NAM ne " and<br>CQ03NMFL ne 'Y'))]<br>Or<br>(CQ04NAM ne " and<br>CQ04NPFL = 'Y') |
| Psychiatric events suggesting serious mood disorders and anxiety | Serious events from the depression CMQ (PSAP defined – depression including mood disorders and anxiety). | CQ09NAM ne '' and<br>AESER = "Y" |
| Suicidality (C-SSRS) | Any treatment-emergent C-SSRS suicidal ideation (1-5) or suicidal behavior (6-10) (defined in Section 9.5.15) – i.e. maximum ideation score worsens relative to pretreatment or maximum behavior score worsens relative to pretreatment | C-SSRS Ideation categories 1-5 and Behavior categories 6-10; any subject with ideation or behavior that is treatment-emergent (defined in Section 9.5.15). |
| Serious infusion and hypersensitivity reactions | Serious infusion and hypersensitivity reactions per the PSAP definition. Includes all SAEs from the anaphylactic reactions CMQ broad search (see Section 11.2.4, includes events on the day of the infusion or within 3 days after the infusion). | CQ05NAM ne '' and<br>AESER='Y' and<br>AEINF3FL='Y' |

## 9.5.13. Treatment-Emergent AEs and AE Duration

Only treatment-emergent AESIs and SAEs, will be summarized, unless otherwise stated. A treatment-emergent AE is an AE that emerges on or after the first treatment dose, having been absent pre-treatment, or that worsens relative to the pre-treatment state.

The duration of the AE will be calculated as follows:

Duration of AE (days) = Date of AE resolution – AE start date + 1.

If the AE is ongoing the duration will be left blank and no imputation will be done.

#### 9.5.14. Incidence Rate

Event incidence rates and subject incidence rates will be calculated for Mortality and Malignancy and other AESIs during the on-treatment and on-study (to Week 52) periods as defined below. Note, for Mortality only subject incidence rates will be calculated. Subject incidence rates will also be calculated for SAEs during the on-treatment and on-study periods at the SOC level only.

Typically for subject incidence rates the subject years would be censored at the time of the event for subjects who experience the event i.e. the subject years contributed to the incidence rate calculation for a subject would be the total years from treatment start date to the event date. However, in consideration of the low number of events, this additional adjustment is not anticipated to have a significant impact. Therefore, the additional adjustment will not be used and the subject years contributed by a subject with an event will be the total years from treatment start date to the end of the treatment period of interest for all AESIs and mortality.

#### **On-treatment**

Subject Incidence Rate = 100 
$$X \frac{Number\ of\ Subjects\ with\ an\ Event}{Overall\ Subject\ Years\ On-Treatment}$$

Event Incidence Rate = 
$$100 X \frac{Number\ of\ Events}{Overall\ Subject\ Years\ On-Treatment}$$

Where overall subject years of on-treatment follow-up =

 $\sum$  all subjects in population [on-treatment follow-up in years]

See Section 9.5.4 for detail on the calculation of on-treatment follow-up.

On-study (to Week 52)

Subject Incidence Rate = 100 X 
$$\frac{Number\ of\ Subjects\ with\ an\ Event}{Overall\ Subject\ Years\ On-Study}$$

Event Incidence Rate = 
$$100 X \frac{Number of Events}{Overall Subject Years On - Study}$$

Where overall subject years on-study =

 $\sum$  all subjects in population [on-study follow-up in years]

See Section 9.5.4 for detail on the calculation of on-study follow-up.

As described in Section 9.1.1, the on-study follow-up (to Week 52) will be different for Mortality and Malignancy compared with other AESIs. This is expected because subjects who withdraw from the study may reconsent to be followed up at Week 52 where only mortality and malignancy data are collected.

## 9.5.15. Treatment-Emergent C-SSRS

For suicidal ideation, the pre-treatment reference period is the lifetime history, current history and baseline (for further detail refer to the IDSL documentation). For suicidal behavior, the pre-treatment reference period is the lifetime history and baseline (note: suicidal behavior is not re-assessed for the current history time period).

Suicidal ideation and suicidal behavior will be considered as distinct categories and assessed independently of each other. Treatment emergence will be assessed for the ontreatment period and the on-study period.

Suicidal ideation will be assessed using responses to C-SSRS ideation questions (categories 1 to 5) only. Suicidal behavior will be assessed using responses to C-SSRS behavior questions (categories 6 to 10) only.

- Treatment emergent suicidal ideation will be assessed using the maximum ideation score pre-treatment, compared to the maximum ideation score post-treatment (on-treatment or on-study as appropriate). If the maximum ideation score worsens relative to the pre-treatment reference period then this will be considered a treatment emergent suicidal ideation. This is derived from responses to suicidal ideation questions (categories 1 to 5).
- Treatment emergent suicidal behavior will be assessed using the maximum behavior score pre-treatment, compared to the maximum behavior score post-treatment (on-treatment or on-study as appropriate). If the maximum behavior score worsens relative to the pre-treatment reference period then this will be considered a treatment emergent suicidal behavior. This is derived from responses to suicidal behavior questions (categories 6 to 10).
- Treatment emergent suicidal ideation or behavior will be defined as a subject having a treatment emergent suicidal ideation (as defined above) and/or a treatment emergent suicidal behavior (as defined above). This definition is used to assess the protocol defined AESI endpoint of 'Suicidality (C-SSRS)' (see Section 9.5.15).

## **Suicidal Ideation (categories):**

- 1. Wish to be Dead
- 2. Non-Specific Active Suicidal Thoughts
- 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act
- 4. Active Suicidal Ideation with Some Intent to Act, Without Specific Plan
- 5. Active Suicidal Ideation with Specific Plan and Intent

#### **Suicidal Behavior (categories):**

- 6. Preparatory Acts or Behavior
- 7. Aborted Attempt
- 8. Interrupted Attempt
- 9. Non-Fatal Actual Suicide Attempt
- 10. Completed Suicide

A subject must have at least one pre-treatment C-SSRS assessment (screening and/or baseline) and at least one on-treatment C-SSRS assessment (post-baseline) to be included in any assessment of treatment emergent.

#### 9.5.16. Prednisone

All prednisone analyses and summaries will consider SLE-related steroids only but data will also be derived for all indications steroids (SLE and non-SLE) for reference where indicated below.

The following will apply to all derivations in this section unless otherwise stated:

- For steroid use analyses, all steroid dosages are converted to a prednisone equivalent in milligrams; therefore, analyses refer to average daily prednisone dose instead of average daily steroid dose. See Appendix 4: Prednisone Equivalent Conversion for instructions on converting steroids to prednisone equivalents.
- This appendix will be updated throughout the course of the study to include all corticosteroids taken by subjects and will be finalized prior to the first database release and unblinding.
- For all derivations of the average daily prednisone equivalent dose including baseline, days on which a subject does not have prednisone use recorded will be considered as 0 mg for the day.
- Steroids taken intravenously (IV), intramuscularly (IM), subcutaneously (SC), intradermally, and orally are considered in prednisone dose derivations only.
- All steroids taken on any given day, including overlaps, will be accounted for in calculations of average daily prednisone dose. To achieve this programmatically, each entry is converted to the prednisone equivalent daily dose (see Appendix 4: Prednisone Equivalent Conversion) and the sum of the prednisone equivalent doses on Day X gives the total prednisone equivalent daily dose on Day X. For example, if two steroids are given on the same day they will be converted to a prednisone equivalent daily dose and then added together to achieve a total for that day.

Steroids used to treat SLE are those with medication type corticosteroid for SLE (SDTM.CM.CMCAT = 'CORTICOSTEROID FOR SYSTEMIC LUPUS ERYTHEMATOSUS').

### 9.5.16.1. Average Daily Prednisone Equivalent

Prior to carrying out calculations, each steroid must be converted to its prednisone equivalent and then the daily dose calculated using the frequency factors provided in

Appendix 4: Prednisone Equivalent Conversion. Days on which the subject has no steroid use will be considered as 0mg.

#### <u>Baseline</u>

At baseline, the average daily prednisone equivalent dose is the sum of all prednisone doses over 7 consecutive days up to, but not including Day 1, divided by 7.

This will be derived for both steroids used to treat SLE and steroids used to treat all indications (SLE and non-SLE) separately. The baseline average daily prednisone dose for all indications will not be reported but will be used to carry out a cross-check against the randomization strata, which were determined by sites based on steroids received for any indication.

### <u>Treatment completion average dose</u>

The average daily prednisone dose is the sum of all prednisone doses over 7 consecutive days up to and including the date of treatment completion, divided by 7.

This will be derived for steroids received for SLE only.

## 9.5.16.2. Average Daily Prednisone Dose during Weeks 40 to 52

The average daily prednisone dose during Weeks 40 to 52 is the sum of all prednisone doses from the day following the Week 40 visit date up to but not including the Week 52 study completion date divided by the number of days between Week 40 visit date and study completion date (study completion date – Week 40 visit date).

For subjects who withdraw from the study prior to the Week 40 visit date, the average daily prednisone dose during Weeks 40 to 52 will be missing.

For subjects who withdraw from the study after the Week 40 visit date, the average daily dose will be calculated as the sum of all prednisone doses from the day after the Week 40 visit date up to and including the date of withdrawal or death, whichever is earlier divided by the number of days between Week 40 visit date and the date of withdrawal or death, whichever is earlier (date of withdrawal or death – Week 40 visit date + 1). If the Week 40 visit is missing for any subject who has not withdrawn or died prior to Week 40, the Week 40 visit date will be imputed as treatment start date + 40 \* 7 for this derivation.

This will be derived for steroids received for SLE only.

#### 9.5.16.3. Cumulative Prednisone Dose

Cumulative SLE-related prednisone dose (area under the curve [AUC]) is defined as the sum of daily prednisone dose from Day 1 to the Week 52 study completion date, considering only corticosteroids used to treat SLE. Missing values will be imputed for each day following the last visit day up to the scheduled Week 52 visit date (treatment start date + 52 \* 7) for subjects who die or withdraw. The daily prednisone dose up to Week 52 after the last visit day, if prior to Week 52 visit date (i.e. for subjects who withdraw from the study or die), will be imputed using the average of the last 28 daily
prednisone doses prior to the day of last visit. For subjects who withdraw from study or die before Day 27, the daily prednisone dose up to Week 52 after early withdrawal or death will be imputed using the average post-baseline daily doses available prior to withdrawal or death.

## 9.5.17. Immunomodulatory Medications

Immunomodulatory medications are identified as all immunosuppressants with ATC code beginning "L04A" plus cyclophosphamide and mercaptopurine. For further detail see Appendix 3: SLE Allowable Medication Categories.

Only immunomodulatory medication used to treat SLE will be included in summary tables of immunomodulatory medication usage (with the exception of the concomitant medication summaries which will include all medications). These are identified as those with a medication type of treatment for SLE (SDTM.CM.CMCAT = 'SYSTEMIC LUPUS ERYTHEMATOSUS').

It will be determined whether immunomodulatory agents are being received at any given reference date by using medication start and stop dates as follows:

- Start date and stop date are prior to reference date → subject is not on immunomodulatory agents
- Start date on or before date and stop date on or after reference date → subject is on immunomodulatory agents
- Start date on or before reference date, stop date is missing and medication is ongoing → subject is on immunomodulatory agents

Status of immunomodulatory medication is assessed at the following dates (i.e. these are the reference dates for the above derivation):

- Baseline
- Treatment completion date in treatment completers (Section 9.5.7)

It is also assessed for shift tables from baseline to:

- Treatment completion date (treatment completers)
- Study agent discontinuation date (subjects who prematurely discontinued study agent)

## 9.5.18. Baseline Allowable SLE Medications

It will be determined whether medications defined in Appendix 3: SLE Allowable Medication Categories, with the exception of steroids, are being received at baseline by using medication start and stop dates as follows:

- Start date and stop date are prior to Day  $1 \rightarrow$  medication not taken at baseline
- Start date on or before Day 1 and stop date on or after Day 1 → medication is taken at baseline

• Start date on or before Day 1, stop date is missing and medication is ongoing → medication is taken at baseline

For steroids, baseline medication will be identified as that taken in the 7 days up to but not including Day 1 as described in Section 9.5.16.1.

## 9.5.19. SLICC/ACR Scoring

- For a given SLICC assessment, if any item(s) is missing, the entire assessment is excluded from summaries and analyses. The only exception to this is if the missing item has previously been scored with damage, in which case damage will be carried forward as detailed below.
- The SLICC/ACR Damage Index (see Appendix 5: SLICC/ACR Damage Index) increases over time. Once a subject meets the criteria for positive scoring of an item, that item should always be marked as present, even if the subject subsequently recovered. This includes baseline assessment.
- In the event the SLICC/ACR Damage Index is scored inconsistently (a decrease at Week 52 relative to baseline has occurred) and the data are unable to be queried and/or corrected, the baseline will be carried forward at the item level for the SLICC/ACR Damage Index questions, i.e. worst observation carried forward (WOCF). These carried forward values will then be used to calculate the total score which will be the value summarized and displayed for reporting. Within the renal domain, damage scored on the first two items (estimated glomerular filtration rate <50%, proteinuria >3.5 gm/24hours) should only be carried forward to Week 52 if the third item (end stage renal disease) has not been scored at Week 52. The reason for this is that scores on the first two items can decrease but only if the third item is then scored.
- Worsening is defined as an increase from baseline in SLICC/ACR Damage Index score (post-baseline visit score baseline score) >0.
  Note: SLICC/ACR is collected only at baseline and Week 52 (in subjects who do not withdraw from the study). It is not collected at the time of IP and or study withdrawal (where applicable) for potential imputation (i.e. carry forward) at Week 52 (see Section 12.2.3 for details).

## 10. STUDY POPULATION

The ITT population will be used to summarize the study population data and data will be presented by treatment and for all subjects combined, unless otherwise specified.

## 10.1. Disposition of Subjects

The number and percentage of subjects randomized by site will be grouped by country and summarized overall and by treatment group using the Randomized population.

Using the Randomized population, the number of subjects in each population (Randomized, ITT, As-Treated) will be summarized overall and by treatment group.

The database did not include all subjects screened for study participation or the number excluded before randomization. Therefore, screening data (including reason for screen failure) will not be summarized or included in the CSR submission datasets since it is not part of the database.

Using the ITT population, an overall summary of subject disposition will be presented with the following included:

- The number and percentage of subjects who completed IP.
  - The number and percentage of subjects who completed the study.
  - The number and percentage of subjects who withdrew from the study
- The number and percentage of subjects who withdrew early from IP.
  - The number and percentage of subjects who completed the study.
  - The number and percentage of subjects who withdrew from the study.
    - The number and percentage of subjects who withdrew from the study on the same date as study agent discontinuation.
  - The number and percentage of subjects who withdrew from the study at a later date than study agent discontinuation.

Further summaries of the ITT population will be produced of subject years' follow-up on-treatment, off-treatment and missing. This will also be given as a percentage of the total possible subject years. Summary statistics will be presented for each category of follow-up: total possible, on-treatment, off-treatment and missing. The summary will be provided for the mortality and malignancy data and all other data separately as the follow-up time differs (except for on-treatment follow-up time which is the same for mortality and malignancy and other data).

Using the ITT population, the subject's study completion status will be assessed to evaluate percentages of withdrawals from study by treatment group as well as the reasons for withdrawal from study. The number and percentage of subjects who completed through Week 52 and who withdrew, including reasons for withdrawal, will be displayed by treatment group and overall. Additionally, the cumulative number and percentage of subjects who withdrew by study visit, derived using visit windows defined in Section 9.5.3, will be displayed by treatment group and overall. A Kaplan-Meier plot of time to study withdrawal will be generated to evaluate the pattern of dropouts over time. Subjects who complete through Week 52 will be censored at the study completion date. The Kaplan-Meier plot will be truncated at Week 52.

Using the ITT population, the subject's IP completion status will be assessed to evaluate percentages of IP withdrawals by treatment group as well as the reasons for IP withdrawal. The number and percentage of subjects who completed IP through Week 48 and who withdrew, including reasons for IP withdrawal, will be displayed by treatment group and overall. Additionally, the cumulative number and percentage of subjects who withdrew from IP by study visit, derived using visit windows defined in Section 9.5.3, will be displayed by treatment group and overall. A Kaplan-Meier plot of time to study treatment withdrawal will be generated to evaluate the pattern of dropouts over time. Subjects who complete IP through Week 48 will be censored at the study treatment

completion date and for subjects who discontinue IP prematurely, the study treatment discontinuation date will be used as the discontinuation date. The Kaplan-Meier plot will be truncated at Week 52.

The number and percentage of subjects who deviated from the inclusion or exclusion criteria will be displayed by treatment group and overall. A listing of subjects who had a deviation from the inclusion or exclusion criteria will be provided.

A listing of subject disposition will be provided showing their completion status and whether they are included in each population. Subjects who are randomized but do not receive any study agent will be identified in this listing. A listing of subjects who withdrew from the study, including reason for and time to withdrawal will also be provided. An additional listing will be provided of subjects who withdrew from IP, including reason and time to withdrawal. Subjects for whom the treatment blind was broken during the study will be listed. A listing of planned and actual treatment arms will be provided. Subjects excluded from any population will be listed.

## 10.2. Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan [Version 8; 19JUL2018].

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorized on the protocol deviations dataset.
- This INFORM dataset (DV) will be the basis for the summaries and listings of protocol deviations.

The percent of subjects who experience an important protocol deviation will be presented by treatment arm for the treatment period. The table will display the number and percentage of subjects with any important protocol deviation and each deviation type. A listing of subjects with an important protocol deviation will be provided by treatment group.

## 10.3. Demographic and Baseline Characteristics

Descriptive statistics will be used to summarize the continuous demographic and baseline characteristics of age (years) and weight (kg). Counts and percentages of the following categorical demographic and baseline characteristics will be presented: country region/country, gender, Hispanic or Latino origin, age group ( $\leq$ 45 years, >45 – <65 years and  $\geq$ 65 years and then within this last group:  $\geq$ 65 – <75 years and  $\geq$ 75 years) and race (Black or Other; see Section 8.3).

The above summary of demographic and baseline characteristics will be repeated for the following subgroups, where the subgroup categories are defined in Section 8.3:

- Age
- Gender

- Race
- Region
- SELENA SLEDAI
- Baseline steroid dose (based on systemic steroids used to treat SLE)

The number and percentage of subjects reporting each race and racial combination will be summarized. For subjects who check more than one race category, the race hierarchy rule defined in Section 9.5.10 will apply for this summary. Note that this differs to the handling of the race subgroup which ignores the hierarchy rule.

A standard summary of the number and percentage of subjects by age ranges Adolescents (12-17 Years), Adult (18–64 Years), from 65 - 84 Years and  $\geq 85$  Years will be provided for disclosure purposes.

A summary of the number and percentage of subjects reporting current medical conditions and a separate summary of number and percentage of subjects reporting past medical conditions will be provided. A summary of the history of tobacco usage will also be provided.

A summary of the randomization stratification factors [screening SELENA SLEDAI score (≤9 vs. ≥10), region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia), and steroid dose (≤7.5 mg/day vs >7.5 mg/day prednisone or equivalent)] will be presented per the randomization and eCRF data.

A cross-tabulation of stratification factors will also be produced summarizing the categories of the randomization strata from IXRS to the eCRF strata for SELENA SLEDAI score (≤9 vs. ≥10), region (US/Canada vs Central America/South America/Mexico vs Europe/Australia/Israel vs Asia), and steroid dose (≤7.5 mg/day vs >7.5 mg/day prednisone or equivalent).

Note that for stratification factors summaries, the steroid dose will be derived from the eCRF considering steroids received for SLE only, whereas the randomization strata were derived by sites considering all steroids.

Demographic and baseline characteristics (age, gender, ethnicity, weight, race [black vs. other]), as well as stratification factors per IXRS, will be listed by subject. Race as assigned using the hierarchy rule (Section 9.5.10) will be listed by subject. Current and past medical conditions and tobacco use history will be listed by subject.

A summary of baseline disease activity will be provided, including counts and percentages for screening SELENA SLEDAI category ( $\leq 9$ ,  $\geq 10$ ), complement levels (Low, Not Low), anti-dsDNA (High, Not High), complement and anti-dsDNA (Low Complement and High Anti-dsDNA, Not (Low Complement and High Anti-dsDNA)). and univariate statistics for SLE disease duration (years), screening SELENA SLEDAI total score, and SLICC/ACR Damage Index. This summary will be repeated for the following subgroups, where the subgroup categories are defined in Section 8.3:

- Age
- Gender
- Race
- Region
- SELENA SLEDAI
- Baseline steroid dose (based on systemic steroids used to treat SLE)

The following indicators of baseline disease activity will also be summarized:

- Screening SELENA SLEDAI category by organ domain and item (count and percentage with each item present)
- Baseline SLICC by organ domain and item (count and percentage with each item present)
- Allowable SLE medication usage (see Appendix 3: SLE Allowable Medication Categories) at baseline counts and percentages by class (Steroids, Anti-Malarials, and Other Immunosuppressive/Immunomodulatory Agents, Aspirin and NSAIDs) and drug as well as summary statistics for average daily prednisone dose (mg/day) (see Section 9.5.16.1 for derivation of average daily prednisone equivalent dose) at baseline and counts and percentages for average daily prednisone dose (mg/day) at baseline (0, >0 ≤7.5, >7.5). See Appendix 4: Prednisone Equivalent Conversion for instructions on converting steroids to prednisone equivalents. Only steroids with medication type corticosteroid for SLE will be included. Only immunomodulatory modulatory medications used to treat SLE will be included. For other medications, all medication types will be included.
- Steroid, Anti-malarial and Immunosuppressant use at Baseline counts and percentages by class (No Steroid, Immunosuppressant or Anti-malarial use, Steroid Only, Immunosuppressant Only, Anti-malarial Only, Steroid and Immunosuppressant Only, Steroid and Anti-Malarial Only, Immunosuppressant and Anti-Malarial Only, Steroid and Immunosuppressant and Anti-malarial). Only steroids with medication type corticosteroid for SLE will be included. Only immunomodulatory modulatory medications used to treat SLE will be included. For other medications, all medication types will be included.

Screening Columbia Suicide Severity Rating Scale (C-SSRS) scores by behavior and ideation components for lifetime and current (counts and percentages) will be presented.

Day 1 C-SSRS components since last visit will be summarized using counts and percentages.

In the screening (lifetime/current) and Day 1 C-SSRS summaries, the number (%) of subjects reporting each individual suicidal ideation (1-5) or behavior (6-10) will be presented (as opposed to the maximum ideation/behavior score).

A listing of screening SELENA SLEDAI results will be provided, including result for individual items and total score.

## 10.4. Concomitant Medications

Concomitant medications will be coded per drug name as defined in the GSK Drug Dictionary, and classified per the GSK-Drug ATC classification level 1 and ATC level 4. Concomitant medications are defined as medications that start on or before the first dose date of study treatment, and end on or after the first dose date of study treatment, or medications that start after the first dose date of study treatment. Note that medications with partial or missing start and/or stop dates will be assumed to be concomitant unless there is evidence through comparison of partial dates to suggest otherwise, for example, if the day is missing, then the month and year will be compared to the month and year of the first dose date of study treatment and if the month and year are the same or later, then the medication will be considered concomitant. See Section 9.4.3 for handling of missing and partial dates. Medications in the database that are determined to not be concomitant will be excluded from table summaries but included in the listing.

A summary of the number and percentage of subjects with concomitant medications by ATC level 1 term and ATC level 4 term will be displayed for the On-Study period. A further summary of concomitant medications by ATC level 4 term and preferred term will be provided for the on-study period (to Week 52). A listing of all concomitant medication data will be displayed by treatment and subject.

Commercial Benlysta is prohibited during the 52-week treatment period of the study, however, if subjects withdraw from IP and begin receiving it they can continue monthly visits as per the study calendar. As such, a listing of subjects who receive commercial Benlysta during the 52-week treatment period will be reported (from both the concomitant medication and the Years 2 to 5 CRF follow-up forms) with the caveat that the Years 2 to 5 data will not be locked at the time of reporting.

## 10.5. Extent of Exposure

The extent of exposure to study treatment through Week 52 will be assessed by examining the duration of exposure to belimumab/placebo in days and the total number of infusions a subject receives. Note that receipt of commercial Benlysta will not be included in exposure calculations.

Duration of exposure in days will be calculated as:

Duration of exposure (days) = Last infusion date – First infusion date +28.

Only complete dates will be used when calculating duration of exposure. First and last infusion dates will be used, regardless of any missed doses.

If a subject has more than one infusion on any given day (i.e. infusion is stopped and then restarted), this will be counted as a single infusion in summaries but both infusions will be listed.

Where a partial infusion is received, this will be counted as one infusion in the calculation of number of infusions.

The duration of exposure and the total number of infusions will be summarized using descriptive statistics for the ITT population. The total number of infusions will also be summarized using counts and percentages using the following categories: 1-5 doses, 6-10 doses and, 11-14 doses.

Subject level exposure data will be listed for all subjects by treatment group and subjects using the Randomized population, flagging subjects whose treatment group differs from the As-Treated population. A listing of study agent administration, including whether total dose was administered and if not the reason why, will be provided. A listing of subjects for whom the blind was broken will also be provided.

## 11. PRIMARY AND OTHER SAFETY ANALYSES

AESI are defined endpoints in the protocol (and clarified in Section 2.2.3). There are also AESI defined in the Benlysta PSAP (Section 15 and Section 16; see Appendix 6: PSAP Sections for AESI Reporting), which overlap with the protocol-defined AESIs.

Analyses and summaries described in Section 11.1.2 will use the protocol-defined AESIs. All safety data from the AE dataset will be displayed in summaries described in Section 11.2.1. This is expected to cover protocol-defined AESIs and SAEs and additionally, though not anticipated, any non-serious AEs which were not in scope for collection in the protocol but remained on the database at database release. The required PSAP summaries for AESI are described in Section 11.2.4.

The primary study summaries will be of overall subject incidence rates of all-cause mortality and AESIs during the on-treatment period, with supportive summaries during the on-study period. SAEs will be descriptively summarized during the on-treatment and on-study periods.

Safety will also be reported using more detailed summaries of deaths, AESIs (per PSAP), and standard summaries of SAEs. Since there is targeted collection of AEs in the study i.e. AESIs and SAEs, this will be clarified where applicable.

To allow comparison with other studies in the Benlysta program, the format and content of the more detailed AESI summaries will be per PSAP standards. Therefore, data on the primary safety endpoints may be contained both at a high level within Section 11.1 and in more detail in Section 11.2.

Safety analysis will be performed on the As-Treated population.

The extent of missing follow-up data (i.e. for subjects who have withdrawn from the study prior to the Week 52 visit) and off-treatment data will be summarized by treatment group. Exploratory analyses may be performed to characterize the potential impact of off-treatment and missing data on the primary mortality endpoint results (see Appendix 7, Mortality Missing Data Exploratory Sensitivity Analyses).

## 11.1. Primary Analysis: All-Cause Mortality, AESI and SAEs

The primary analyses will be performed for both the on-treatment and on-study periods, as defined in Section 9.1. The primary interest is in the on-treatment period, with the on-study considered an important supportive analysis.

The primary analyses for the on-treatment period will be repeated for subgroups as defined in Section 8.3. Follow-up adjusted summaries (i.e. subject incidence rate/event incidence rate) will not be included in subgroup tables.

An overall Double Dotplot for the percentage of subjects with an event will be provided for mortality and other AESIs for the on-treatment period. This is a panel display with two associated dot-plots; the left-hand panel will show the percentage of subjects with an event in each arm. The right-hand panel will show the difference in percentages, with bars for the 95% confidence interval around the difference. All AESIs and mortality will be displayed on the same plot. Further detail on methodology is given in Section 11.1.1 and Section 11.1.2.

An overall Double Dotplot for exposure-adjusted subject incidence rate will be provided for mortality and other AESIs for the on-treatment period. This is a panel display with two associated dot-plots; the left-hand panel will show the exposure-adjusted subject incidence rate in each arm. The right-hand panel will show the difference in the exposure-adjusted subject incidence rate, with bars for the 95% confidence interval around the difference. All AESIs and mortality will be displayed on the same plot. Further detail on methodology is given in Section 11.1.1 and Section 11.1.2.

## 11.1.1. All-Cause Mortality

See Section 11.2.1 and Section 11.2.2 for further summaries and listings of deaths.

## **Percentages**

A summary of the number and percentage of subjects who have died will be provided for belimumab and placebo as well as the difference in the percentage of subjects between the belimumab and placebo groups. The difference in percentages will be evaluated with a 2-sided 95% CI, using the simple asymptotic Chi-Square (Pearson) method [Newcombe, 1998]. This will be considered as the primary method of assessment of the treatment difference.

## **Subject Incidence Rate**

Whilst a difference between belimumab and placebo groups in IP exposure and overall study duration (to Week 52) is not anticipated, to account for this, supplemental summaries using subject incidence rates will be provided.

The subject incidence rate of mortality per 100 subject years will be provided for belimumab and placebo as well as the difference between belimumab and placebo with 95% CIs. For within-group rates per 100 subject years, the 95% CI will be obtained via

on an exact Poisson method [Stokes, 2012]. For differences in rates between groups, the 95% CI will be constructed using a Normal approximation (Wald's method, [Liu, 2006]).

See Section 9.5.14 for further details on the calculation of incidence rates for the ontreatment and on-study periods.

### Kaplan-Meier Figure

A plot of the Kaplan-Meier curve, including standard error bands, for all-cause mortality for belimumab and placebo will be provided to show the change in risk over time. The Kaplan-Meier estimates table will be outputted for quality control purposes but will not be used included in the tables or listings.

Time to Event is defined for the On-Treatment Period and On-Study Period as follows:

- For subjects who died during the evaluation period of interest (i.e. on-treatment or on-study): Time to event is the date of death first exposure date +1.
- For subjects who did not die or died after the end of the evaluation period of interest (i.e. on-treatment or on-study): Time to event (censored) is the censoring date first exposure date + 1.

Occurrence and date of death will be determined based on the AE dataset where outcome = fatal (date of death will be derived as the end date of the SAE with fatal outcome).

The censoring date will be assigned based on the evaluation period of interest as follows:

- **On-treatment**: end date for On-Treatment period (see Section 9.1.1)
- **On-study:** end date for On-Study period for mortality and malignancy events (see Section 9.1.1)

The time to event will be calculated in days, as described above. However, the x-axis of the KM plot will display time in weeks. The following conversion will be applied for time to event days to weeks, in order to display the correct week according to the scheduled visit plan (see Section 9.5.2). For example, Day 57 as Week 8, Day 113 as Week 16.

Time to event (weeks) = [Time to event (days) -1] /7

The number of subjects at risk at certain timepoints [i.e. Week 8 (Day 57), Week 16 (Day 113), etc.] will be presented for each treatment group. The number of subjects at risk is defined as the number of subjects alive and uncensored at a time just prior to time t (e.g. for Week 8, this would be the number of subjects at risk at the start of Day 57). The Kaplan-Meier plot will be truncated at Week 52.

#### **Cumulative Time to Mortality**

The cumulative number and percentage of subjects who died by study visit, derived using visit windows defined in Section 9.5.3, will be displayed by treatment group for the On-Treatment Period and the On-Study Period.

### 11.1.2. Protocol-Defined AESI

Protocol-defined AESIs are defined in Section 9.5.12.

Note, for Suicidality (C-SSRS) only, a subject must have at least one pre-treatment C-SSRS assessment (screening and/or baseline) and at least one on-treatment C-SSRS assessment (post-baseline) to be included in the summaries.

## **Percentages**

For each of the AESIs a summary of the number and percentage of subjects experiencing at least one event will be provided for belimumab and placebo as well as the difference in the percentage of subjects (and 95% CI) between the belimumab and placebo groups using the same methodology as for mortality.

## **Subject Incidence Rate**

The incidence rate for each AESI per 100 subject years will be provided for belimumab and placebo groups as well as the difference between placebo and belimumab (and 95% CI) using the same methodology as for mortality.

#### **Event Incidence Rate**

The number of events and event rate for each AESI, except Suicidality (C-SSRS), per 100 subject years will be provided for belimumab and placebo groups.

#### 11.1.3. SAEs

SAEs will be presented using descriptive statistics.

A summary of the number and percentage of subjects with SAEs reported during the ontreatment and on-study (to Week 52) periods will be provided along with the number of events. Subject incidence rates will also be provided at the SOC level only (see Section 9.5.14 for derivation) for on-treatment and on-study periods.

See Section 11.2.1 for further details of SAE summaries and Section 11.2.2 for a description of the SAE listings.

## 11.2. Other Safety Summaries

#### 11.2.1. AESI and SAEs

This section describes additional summaries to be generated for all safety data in the AE dataset. These data will be referred to as AESIs and SAEs throughout this section but could include out of scope AEs if entered by sites. For the AESI analysis/groupings as per the Belimumab PSAP definitions, see Section 11.2.4 (and Section 9.2 for AESI adjudication details).

For the following summaries, only treatment-emergent AESIs and SAEs will be summarized, unless otherwise stated (see Section 9.5.13 for definitions of Treatment Emergent and derivation of AE duration).

All treatment-emergent AESIs and SAEs will be summarized for the On-Treatment and On-Study (to Week 52) periods, unless otherwise specified in the list of displays.

All AESIs and SAEs will be classified using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary, and grouped by SOC and preferred term (PT), unless otherwise stated.

The investigator will evaluate all AESIs and SAEs with respect to seriousness, severity, and causality. The severity of an AESI or SAE is to be evaluated according to the Adverse Event and Laboratory Value Severity Grade Tables in Protocol Appendix 8, if a grade is defined for the AE of interest.

An overall summary of AESIs and SAEs will be presented showing the number and percent of subjects with at least one: AESI or SAE, Study Agent related AESI or SAE, serious AE (SAE), severe AESI or SAE, AESI or SAE resulting in premature study agent discontinuation, AESI or SAE resulting in study withdrawal, AESI or SAE resulting in premature study agent discontinuation and/or study withdrawal, deaths (timing based on fatal SAE start date) and deaths (timing based on fatal SAE end date i.e. date of death). This summary will be presented for the On-Treatment and On-Study periods.

The number and percentage of subjects experiencing an AESI or SAE and the total number of AESIs and SAEs will be summarized for AE categories and treatment periods as shown in Table 1.

A listing of subject numbers for each AESI or SAE will also be produced. AESIs and SAEs will be grouped and sorted by SOC and PT. A listing of all AESIs and SAEs and study agent related AESIs and SAEs will be presented, including duration and study day of onset/resolution.

Table 1 AESIs and SAEs Displays

| Category | On-Treatment Period | On-Study (to Week 52)<br>Period |
|---|---|---|
| All AESIs and SAEs | by SOC<br>by SOC and PT<br>by PT only | by SOC and PT |
| AESIs and SAEs by Severity | by SOC and PT | |
| Serious AEs | by SOC<br>by SOC and PT<br>by PT | by SOC and PT |
| Study Agent Related AESIs and SAEs | by SOC<br>by SOC and PT<br>by PT only | |
| Study Agent Related AESIs and SAEs by Severity | by SOC and PT | |

| Category | On-Treatment Period | On-Study (to Week 52)<br>Period |
|---|---|---|
| AESIs and SAEs Leading to<br>Premature Discontinuation of<br>Study Agent | by SOC and PT<br>by PT | by SOC and PT |
| AESIs and SAEs Leading to Withdrawal from Study | by SOC and PT | by SOC and PT |
| Common Non-Serious AESI<br>≥1% | by SOC and PT | |
| Non-serious Study Agent<br>Related AESI | by PT | |
| Study Agent Related SAEs | by SOC and PT<br>by PT | |
| Fatal SAEs (assigned to period based on SAE start date) | by SOC and PT<br>by PT | by SOC and PT |
| Study Agent Related Fatal<br>SAEs (assigned to period<br>based on SAE start date) | by SOC and PT | |
| AESIs and SAEs by Age group | by SOC and PT | |
| AESIs and SAEs by Gender | by SOC and PT | |
| AESIs and SAEs by Race | by SOC and PT | |
| AESIs and SAEs by Region | by SOC and PT | |
| AESIs and SAEs by<br>Complement Levels and Anti-<br>dsDNA | by SOC and PT | |

The tabular summary for each category of AESIs and SAEs listed above will include the number of events, number of subjects who reported at least one event, and percentage of subjects who reported at least one AESI or SAE (incidence) by treatment group for each SOC (where applicable), each PT, and overall. By default, adverse events will be sorted by MedDRA SOCs, in descending order from the SOC with the highest total incidence (i.e., summed across all treatment groups) for any adverse event within the class, to the SOC with the lowest total incidence. If the total incidence for any two or more adverse events is equal, the events will be presented in alphabetical order. Only SOCs with observed AE PTs will be presented. Repeat sort order for MedDRA PTs within each SOC.

Common AESIs and SAEs will be defined as  $\geq 1\%$  in either treatment group.

For disclosure, an additional summary of SAEs by SOC and PT will be produced in the format required for the on-treatment period. The table will include the number and percentage of subjects with an SAE along with the number of SAEs, drug-related SAEs, fatal SAEs and drug-related fatal SAEs.

A summary of AESIs and SAEs by SOC, PT and severity will be provided by treatment group. For this display, the number and percentage of subjects will be summarized as mild, moderate or severe based on the maximum severity observed across all PTs within the SOC for a given subject.

The hierarchical relationship between MedDRA SOCs, PTs, and verbatim text will be listed for all AESIs and SAEs.

A listing that displays which subjects reported each AESI or SAE will also be produced. AESIs and SAEs will be grouped and sorted by SOC and PT.

A listing of all AESIs and SAEs and study agent related AESIs and SAEs will be presented, including duration and study day of onset/resolution.

A listing of SAEs and AESIs that are recorded between withdrawal of consent and Week 52 Follow-Up, excluding mortality and malignancy, will be produced. The intent is to capture events that were not included in summaries for the on-study period as the protocol did not specify to collect them.

#### 11.2.2. Deaths and Serious Adverse Events

In addition to the tabular summaries of AESIs and SAEs described in Section 11.2.1, listings for all SAEs, all fatal SAEs (deaths) and all non-fatal SAEs will be produced. A listing of reasons for considering an AE as an SAE will be provided. The categorization of the cause of death will be adjudicated by GSK (see Section 9.2).

A summary of deaths (fatal SAEs) by category and preferred term will be produced based on the start date of the fatal SAE (to determine whether the event occurred during the relevant study period). A separate summary will be produced of deaths by category and preferred term based on end date of fatal SAE (i.e. using date of death to determine whether the event occurred during the relevant study period). Both summaries will be for the on-treatment period.

Survival status will also be summarized at Week 52, based on information collected on the Week 52 Survival form, for all subjects in the As-Treated population. The number and percentage of subjects will be summarized for each of the following categories:

- Alive
- All Deaths (based on date of death)
  - Deaths on Treatment (during the on-treatment period)
  - Deaths Post-Treatment (after the on-treatment period)
- Unknown
  - Lost to Follow-Up
  - Unattainable

A listing of survival status at Week 52 will also be presented.

# 11.2.3. AESIs and SAEs Leading to Discontinuation of Investigational Product or Withdrawal from Study

In addition to the tabular summaries described in Section 11.2.1, the following listings will also be produced:

- all AESIs and SAEs leading to premature discontinuation of study agent.
- all AESIs and SAEs leading to withdrawal from the study (i.e., withdrawal of consent).

Note that non-serious AEs leading to withdrawal that are not protocol-defined AESI are not collected in the database.

## 11.2.4. PSAP-Defined Adverse Events of Special Interest

The PSAP has been developed to include AESI summaries for consistent reporting across belimumab studies which will be included here in addition to the primary summary of overall AESI rates described in Section 11.1.2 of this RAP.

Categorizations for the AESIs from the PSAP are defined Appendix 6: PSAP Sections for AESI Reporting and reporting of AESIs for these analyses is defined below.

An overall summary of AESI will be presented. Selected categories of AESI will be presented separately by PT. Infection AESIs will also be presented by PT for infections leading to discontinuation of study agent. The number and percentage of subjects with at least one occurrence and the number of events of the following AESI will be provided.

- Malignant Neoplasms
  - Malignancies Excluding non-melanoma skin cancer (NMSC) [see Section 9.5.12, protocol defined AESI]
  - Malignancies Including NMSC
  - Solid Tumour
  - Hematologic
  - Skin (All)
    - NMSC [see Section 9.5.12, protocol defined AESI]
    - Excluding NMSC
  - Tumours of unspecified malignancy adjudicated as malignant per GSK adjudication
- Post-Infusion Systemic Reactions
  - Post-Infusion Systemic Reactions per Anaphylactic Reaction
     Customized MedDRA Query (CMQ) narrow search (on the day of the infusion or within 3 days after the infusion)
    - Serious Post-Infusion Systemic Reactions per Anaphylactic Reaction Customized MedDRA Query (CMQ) narrow search (on the day of the infusion or within 3 days after the infusion)

- Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion)
  - Serious Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion) [see Section 9.5.12, protocol defined AESI]
- Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ algorithmic search (on the day of the infusion or within 3 days after the infusion)
  - Serious Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ algorithmic search (on the day of the infusion or within 3 days after the infusion)
- Serious Anaphylaxis per Sampson Criteria
- Serious Acute Post-Infusion Systemic Reactions/Hypersensitivity per GSK adjudication
  - Serious Acute Post-Infusion Systemic Reactions Excluding Hypersensitivity per GSK adjudication
  - Serious Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Non-Acute Hypersensitivity Reactions per GSK adjudication
- All Infections of Special Interest [see Section 9.5.12, protocol defined AESI]
  - Serious Infections of Special Interest
  - All opportunistic infections per GSK adjudication
    - Serious opportunistic infections per GSK adjudication
  - Opportunistic infections per GSK adjudication excluding Tuberculosis and Herpes Zoster
    - Serious opportunistic infections per GSK adjudication excluding Tuberculosis and Herpes Zoster
  - Active Tuberculosis
    - Non-Serious Active Tuberculosis
    - Serious Active Tuberculosis
    - Non-Opportunistic
      - Serious Non-Opportunistic
    - Opportunistic
      - Serious Opportunistic
  - Herpes Zoster
    - Serious Herpes Zoster
    - Non-Opportunistic
      - Serious Non-Opportunistic
    - Opportunistic
      - Serious Opportunistic
      - Recurrent

- Serious Recurrent
- Disseminated
  - o Serious Disseminated
- Sepsis
  - Serious Sepsis
- Depression/suicide/self-injury
  - Depression (Inc. mood disorders and anxiety)
    - Serious Depression (Inc. mood disorders and anxiety) [see Section 9.5.12, protocol defined AESI]
    - Suicide/self-injury
      - Serious Suicide/self-injury
  - Serious Suicide/Self-injury per GSK Adjudication
    - Suicidal behavior per GSK Adjudication
      - Completed Suicide per GSK Adjudication
    - Suicidal Ideation per GSK Adjudication
    - Self-injurious Behavior Without Suicidal Intent per GSK Adjudication
- Deaths (using start date of fatal SAE to determine whether event occurred during the relevant study period)
- Deaths (using end date of fatal SAE i.e. date of death to determine whether event occurred during the relevant study period)

A listing of all PSAP-defined AESIs will be produced.

#### 11.2.4.1. Post-infusion Systemic Reactions

Summaries of post-infusion systemic reactions will be presented by the first six infusions and PT for the following categories:

- Serious Post-Infusion Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion)
- Serious Acute Post-Infusion Systemic Reactions per GSK adjudication
- Serious Delayed Acute Post-Infusion Systemic Reactions per GSK adjudication
- Serious Delayed Non-Acute Post-Infusion Systemic Reactions per GSK adjudication

## 11.2.5. Columbia-Suicide Severity Rating Scale (C-SSRS)

The definition of treatment-emergent with respect to C-SSRS (suicidal ideation and/or behavior) is given in Section 9.5.15.

Suicidality assessments are completed at every visit. Assessments are done using the C-SSRS. If a "yes" response is given to any suicidal behavior or a "yes" response to suicidal ideation questions with category 3, 4 or 5 on the C-SSRS, the investigator will be

prompted to complete the Possible Suicidality Related Questionnaire (PSRQ). A listing of the PSRQ will be presented.

Listings will be generated for the following:

- Suicidal ideation and behavior data for subjects who have any suicidal ideation or behavior recorded at any point on the study (including screening or baseline).
- Behavior details for subjects who have any suicidal behavior recorded at any point on the study (including screening or baseline)
- The most severe suicidal ideation details for subjects who have any suicidal ideation recorded at any point on the study (including screening or baseline).

#### 11.2.5.1. C-SSRS Suicidal Ideation or Behavior

The number and percentage of subjects with suicidal ideation or behavior at any time during the on-treatment and on-study (to Week 52) periods will be presented. For suicidal ideation, the maximum ideation score (1-5) at any time during the relevant period will be presented. For suicidal behavior, all behaviors (6-10) present at any time during the relevant period will be presented. This will be regardless of whether the subject had pretreatment history (up to and including baseline [see Section 9.5.1 for baseline definition]). The categories of suicidal ideation and behavior are presented in increasing order of severity from 1 to 5, and 6-10 respectively.

#### 11.2.5.2. C-SSRS Suicidal Ideation or Behavior Relative to Pre-Treatment

The number and percentage of subjects with treatment-emergent suicidal ideation or behavior -post-baseline will be presented during the on-treatment and on-study (to Week 52) periods (see Section 9.5.15).

A subject must have at least one pre-treatment C-SSRS assessment (screening and/or baseline) and at least one on-treatment C-SSRS assessment (post-baseline) to be included in this display.

A subject may have treatment emergent suicidal ideation and/or behavior.

The following categories will be presented:

- The number (%) of subjects with any treatment emergent suicidal ideation (1-5)
  - The number (%) of subjects with any treatment emergent more severe suicidal ideation (4-5)
- The number (%) of subjects with any treatment emergent suicidal behavior (6-10)
- The number (%) of subjects with any treatment emergent suicidal ideation (1-5) or suicidal behavior (6-10)

Note: treatment emergent suicidality can only be assessed in subjects with a pre-treatment maximum ideation score of 4 or lower (as subjects with a pre-treatment ideation score of 5 have no potential to worsen on the 1-5 ideation scale)

In addition, a shift table showing the maximum pre-treatment ideation score versus the maximum post-treatment ideation score will be produced for the on-treatment and on-study periods. The maximum pre-treatment behavior score versus the maximum post-treatment behavior score will also be presented in the summary table. These summaries will be provided post Statistical Analysis Complete (SAC).

### 11.2.5.3. C-SSRS Shift Changes in Categories from Pre-Treatment to On-Treatment

A summary of the shift from maximum pre-treatment C-SSRS category to maximum ontreatment and on-study (to Week 52) category will be produced.

The pre-treatment period for ideation is based on the lifetime, current and baseline history. For behavior, it is based on the lifetime and baseline history. A subject must have at least one pre-treatment assessment and at least one on-study assessment to be included in this display.

The table will display the number and percentage of subjects within the specific shift categories: No suicidal ideation or behavior, suicidal ideation, and suicidal behavior.

Each subject will appear in the table only once. For the purposes of this table only, a subject with both suicidal ideation and suicidal behavior in any period (pre-treatment/on-treatment/on-study) will appear in the category of suicidal behavior only.

## 12. EFFICACY ANALYSES

The efficacy analyses will be performed for the ITT population as defined in Section 6 unless otherwise stated. The data will be presented by treatment group.

## 12.1. Major Efficacy Analyses

# 12.1.1. Percent of Subjects with Prednisone Reduction by ≥25% from baseline to ≤7.5 mg/day during Week 40 through Week 52

#### **Primary Analysis**

For this analysis, only steroids used to treat SLE will be included and only subjects with a baseline average daily prednisone dose >7.5mg/day will be included. See Section 9.5.16.1 for derivation of baseline prednisone dose and Section 9.5.16.2 for derivation of average prednisone use between Week 40 to Week 52.

The percent of subjects whose average prednisone dose has been reduced by  $\ge 25\%$  from baseline to  $\le 7.5$  mg/day during Weeks 40 through 52 will be compared between belimumab and placebo using a logistic regression model. Independent variables in the model will include treatment group, baseline prednisone dose, and the following

randomization stratification factors per the eCRF: screening SELENA SLEDAI score ( $\leq 9$  vs.  $\geq 10$ ), and region. A responder is defined as having a prednisone reduction by  $\geq 25\%$  from baseline to  $\leq 7.5$  mg/day during Weeks 40 through 52.

Any subject who withdraws from the study or adds new immunomodulatory agents used to treat SLE (note that this will include switches) prior to the Week 52 visit will be considered having no steroid reduction.

A summary of the number and percentage of subjects who are responders by treatment group, the treatment difference versus placebo, the odds ratio and 95% CI versus placebo, and a p-value for the odds ratio will also be provided.

## Sensitivity Analysis

 To examine the robustness of the results, a sensitivity analysis of the SLErelated steroid reduction will be performed without considering any information related to the use of new immunomodulatory agents (note that this will include switches).

## Additional Summaries of Prednisone

- A summary of the number and percentage of subjects with average SLE-related daily prednisone dose ≤7.5mg/day and >7.5 mg/day at baseline (Day 1) and treatment completion date will be presented for treatment completers.
- The cumulative SLE-related prednisone dose will be derived as described in Section 9.5.16.3. A table of descriptive statistics will be presented including the mean, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum.
- A listing of cumulative SLE-related prednisone dose will be displayed by treatment and subject.

## 12.2. Other Efficacy Analyses

## 12.2.1. Immunomodulatory Agents to Treat SLE

The following summaries will present immunomodulatory agents used to treat SLE only, i.e. those with medication type 'SYSTEMIC LUPUS ERYTHEMATOSUS'.

- A summary of the number and percentage of subjects taking immunomodulatory agents to treat SLE by ATC level 4 term and preferred term will be displayed for the on-study period.
- A summary of the number and percentage of subjects on immunomodulatory agents to treat SLE at baseline (see Section 9.5.17 for derivation of baseline medication) and at the treatment completion date (in treatment completers as defined in Section 9.5.7 with a treatment completion date) will be presented.

A summary of the shift (on versus off immunomodulatory agents to treat SLE) from baseline category to treatment completion date (in subjects who completed IP as

scheduled) and at study agent discontinuation date (subjects who prematurely discontinued IP)

See Section 9.5.17 for detail on defining immunomodulatory medication use at baseline and treatment completion.

All immunomodulatory agents will be indicated in the listing of concomitant medications.

## 12.2.2. Hospitalizations

This information will be derived from the SAEs using the review process outlined in Section 9.3.

The number and percent of subjects hospitalized will be presented along with the number of hospitalizations per subject.

Subjects with hospitalizations and SAEs contributing to hospitalization will be indicated in the listing of SAEs and the number of hospitalization per subject (identified by clinical review, see Section 9.3) will also be listed.

## 12.2.3. SLICC/ACR Damage Index

SLICC/ACR is attached in Appendix 5: SLICC/ACR Damage Index.

A listing of all available SLICC/ACR data will be provided, including the analysis result for each item, the total score and the change from baseline at Week 52.

## 12.2.3.1. SLICC/ACR Damage Index Change from Baseline at Week 52

The change from baseline in SLICC/ACR Damage Index score at Week 52 will be summarized for belimumab and placebo.

The table will display the summary statistics for the SLICC/ACR Damage Index score at baseline and at Week 52. The table will also display the mean change from baseline, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum. Only subjects who complete the full course of study agent through 48 weeks and complete the study to Week 52 will be included in the summary at Week 52.

A separate summary will be produced for subjects who complete the study through 52 weeks, i.e. subjects with off-treatment data will be included. The table will display the summary statistics for the SLICC/ACR Damage Index score at baseline and at Week 52. The table will also display the mean change from baseline, standard deviation, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, minimum and maximum.

#### 12.2.3.2. SLICC/ACR Damage Index Worsening at Week 52

The number and percentage of subjects with worsening in their SLICC/ACR Damage Index score compared with baseline at Week 52 will be presented. Worsening is defined as a change in score (Week 52 visit minus Baseline) >0. The percentage of subjects with

worsening in their SLICC/ACR Damage Index score at Week 52 will be compared between belimumab and placebo using a logistic regression model. The independent variables in the model will include treatment group and randomization strata per the eCRF: steroid dose (≤7.5 mg/day vs >7.5 mg/day prednisone or equivalent used to treat SLE), region, screening SELENA SLEDAI score (≤9 vs. ≥10), and baseline SLICC/ACR Damage Index score.

The table will display the number and percentage of subjects with worsening in their SLICC/ACR Damage Index score by treatment group, the treatment difference versus placebo, the odds ratio and 95% CI versus placebo, and a p-value for the odds ratio.

Only subjects who complete the full course of study agent through 48 weeks and complete the study to Week 52 with a baseline and post-baseline assessment will be included in the analysis. See Section 9.5.19 for further detail.

A separate summary will present the number and percentage of subjects with worsening at Week 52 compared to baseline by organ domain in treatment completers who have a Week 52 SLICC assessment. Only subjects who have potential to worsen in a given domain will be summarized for that domain, i.e. subjects who do not have the maximum damage score for the domain at baseline.

A summary will also be produced for subjects who complete the study through 52 weeks, i.e. subjects with off-treatment data will be included. The table will display the number and percentage of subjects with worsening in their SLICC/ACR Damage Index score by treatment group and the treatment difference versus placebo.

#### Subgroups

The SLICC/ACR worsening at Week 52 will be summarized for treatment completers with a Week 52 assessment for subgroups listed in Section 8.3 using the eCRF data to derive randomization stratification factors.

## 13. PHARMACOGENETIC DATA ANALYSES

Any pharmacogenetic analyses will be described in a separate pharmacogenetic analysis plan and will be reported separately from the main clinical study report.

## 14. REFERENCES

Buyon JP, Petri MA, Kim MY,et al. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: a randomised trial. Ann Internal Med. 2005;142(12 Pt 1):953-62.

Gladman EM, Ginzler E, Goldsmith C et al. SLICC/ACR damage index for SLE. Arthritis Rheum. 1996;39(3):363 9.

Liu GF, Wang J, Liu K, Snavely DB. Confidence intervals for an exposure adjusted incidence rate difference with applications to clinical trials. Stat. Med. 2006;25:1275-86.

Newcombe RG. Interval estimation for the difference between independent proportions: comparison of eleven methods. Stat Med. 1998;17:873-90.

Petri M, Kim MY, Kalunian KC, Grossman J, Hahn BH, Sammaritano LR, et al. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med. 2005;353:2550-8.

Rubin, DB. Multiple imputation for nonresponse in surveys. New York, NY: John Wiley & Sons, 1987.

Stokes ME, Davis CS, Koch GG. Categorical data analysis using SAS, Third Edition. Cary, NC: SAS Institute Inc. 2012: 390-93.

## 15. APPENDICES

# 15.1. Appendix 1: Countries by Region

| Country | Region for Randomization Stratification |
|----------------|-----------------------------------------|
| Canada | US/Canada |
| USA | US/Carlada |
| Argentina | |
| Brazil | |
| Chile | |
| Colombia | Central America/South America/Mexico |
| Mexico | |
| Peru | |
| Puerto Rico | |
| Australia | |
| Bulgaria | |
| Croatia | |
| Czech Republic | |
| Estonia | |
| Hungary | |
| Israel | |
| Italy | |
| Lithuania | |
| New Zealand | |
| Norway | Europe/Australia/Israel |
| Poland | |
| Portugal | |
| Romania | |
| Russia | |
| Serbia | |
| Slovakia | |
| Spain | |
| Switzerland | |
| Turkey | |
| Ukraine | |
| China | |
| Hong Kong | |
| India | |
| Indonesia | |
| Korea | Asia |
| Malaysia | |
| Philippines | |
| Taiwan | |
| Thailand | |

## 15.2. Appendix 2: SELENA SLEDAI Organ System Domains

## **SELENA SLEDAI Organ System Domains**

SELENA SLEDAI assessments consist of 24 individual weighted items in which signs and symptoms, laboratory tests, and physician's assessment for each of 8 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease (marked 'No'), but in practice few subjects have scores >45 [Buyon, 2005; Petri, 2005].

Organ system domain scores are the sum of the weights of items within the organ domain as defined in the table below.

In the eCRF, laboratory items on the SLEDAI may also be ticked 'unknown' to indicate the lab test was not available. The laboratory items are: urinary casts, hematuria, proteinuria, pyuria, low complement, increased DNA binding, thrombocytopenia, and leukopenia.

List of organ systems, items, and weights for the assessments are provided.

| Organ System | Descriptor | Weight | |
|----------------------------------|------------------------|--------|---|
| [1] CNS | Seizure | 8 | |
| | Psychosis | 8 | |
| | Organic Brain Syndrome | 8 | |
| | Visual Disturbance | 8 | |
| | Cranial Nerve Disorder | 8 | |
| | Lupus Headache | 8 | |
| | CVA | 8 | |
| [2] Vascular | Vasculitis | 8 | |
| [3] Musculoskeletal | Arthritis | 4 | |
| | Myositis | 4 | |
| [4] Renal | Urinary Casts | 4 | |
| | Hematuria | 4 | |
| | Proteinuria | 4 | - |
| | Pyuria | 4 | - |
| [5] Mucocutaneous | Rash | 2 | |
| | Alopecia | 2 | |
| | Mucosal Ulcers | 2 | |
| [6] Cardiovascular & Respiratory | Pleurisy | 2 | |
| | Pericarditis | 2 | |
| [7] Immunologic | Low Complement | 2 | |
| | Increased DNA Binding | 2 | |
| [8] Hematologic | Thrombocytopenia | 1 | |
| | Leukopenia | 1 | |
| [9] Constitutional | Fever | 1 | |

# 15.3. Appendix 3: SLE Allowable Medication Categories

| Medication Category | Rule |
|---|---|
| Anti-malarials | Set to "ANTIMALARIALS" if the preferred term |
| | begins with "QUINACRINE", "QUININE", |
| | "HYDROXYCHLOROQUINE", |
| | "MEPACRINE", or "CHLOROQUINE" |
| | AND |
| | the route of administration is not 'TOPICAL', |
| | 'VAGINAL', 'CONJUNCTIVAL', 'INTRANASAL', |
| | 'INHALATION', 'INTRA-OCULAR',<br>'INTRATRACHEAL', 'EPIDURAL', 'INTRA- |
| | ARTICULAR', or 'OTHER'. |
| Steroids | Set to 'STEROIDS' if at least one associated ATC |
| Oteroids | code (ATCCD1 – ATCCD6) begins with 'H02' |
| | AND |
| | Route of administration is |
| | "INTRADERMAL", "INTRAMUSCULAR", |
| | "INTRAVENOUS", "ORAL", "SUBCUTANEOUS", |
| | or "INTRA-ARTICULAR". |
| Immunosuppressants | Set to 'IMMUNOSUPPRESSANTS' if at least one |
| | associated ATC code (ATCCD1 – ATCCD6) begins |
| | with 'L04A' or the preferred term begins with |
| | "CYCLOPHOSPHAMIDE" (oral and parenteral |
| | routes) or "MERCAPTOPURINE" (oral route). |
| NSAIDs | Set to NSAIDs if at least one associated ATC code |
| | (ATCCD1 – ATCCD6) begins with 'M01A'. |
| Aspirin | Set to "ASPIRIN" if CMDECOD contains |
| | "ACETYLSALICYLIC ACID" or |
| | "ACETYLSALICYLATE LYSINE". |
| Prohibited | Set to "PROHIBITED" if any of |
| | the following conditions are met, if CMDECOD |
| | equals "INVESTIGATIONAL DRUG", |
| | "IMMUNOGLOBULIN", |
| | "ADALIMUMAB", "ETANERCEPT", "INFLIXIMAB", "RITUXIMAB", "ABATACEPT", "ANAKINRA", |
| | "GOLIMUMAB", "ABATACEPT", "ANAKINRA", "GOLIMUMAB", "CERTOLIZUMAB" or |
| | "BELIMUMAB". |
| | DELIIVIUIAD . |

## 15.4. Appendix 4: Prednisone Equivalent Conversion

- A concomitant medication is identified as a steroid if at least one associated ATC code (ATCCD1 ATCCD6) begins with 'H02.'
- The following routes are considered to provide systemic exposure: oral, subcutaneous, intramuscular, intradermal, and intravenous. Topical routes of administration are excluded (e.g., topical, conjunctival, intranasal).
- At data base release, all preferred terms identified with an ATC code beginning with 'H02' will be reviewed to ensure a conversion factor exists for all terms with a systemic route of administration.
- Similarly, all routes of administration for preferred terms with an ATC code beginning with 'H02' will be reviewed to ensure all systemic routes have been identified in the list above.
- In order to be converted the frequency and dose of the steroid must be present with the unit dose in milligrams (mg).
- Reported dose for systemic steroid is converted to prednisone equivalent dose using conversion factor for each particular medication (refer to online calculator http://www.globalrph.com/corticocalc.htm).

A two-step process will be used to calculate the prednisone equivalent daily dose:

- 1. DOSE2 (prednisone equivalent dose in mg) = DOSE (collected dose in mg) x Conversion Factor
- 2. DD (daily dose in mg/day) = DOSE2 (prednisone equivalent dose in mg) x Frequency Factor

Where multiple steroids are taken on one day, the sum of these will be the prednisone equivalent daily dose. An intermediate dataset will contain the total daily prednisone equivalent daily dose for each study day. This will be used to derive prednisone endpoints.

| Preferred term | Conversion factor for converting to a prednisone-equivalent dose |
|---|---|
| BETAMETHASONE | 8.333 |
| BETAMETHASONE DIPROPIONATE | 8.333 |
| BETAMETHASONE SODIUM PHOSPHATE | 8.333 |
| BETAMETHASONE VAL | 8.333 |
| BETROSPAM | 8.333 |
| CELESTONA BIFAS | 8.333 |
| CORTISONE | 0.2 |
| CORTISONE ACETATE | 0.2 |
| CRONOLEVEL | 8.333 |
| DEFLAZACORT | 0.8333 |
| DEPO-MEDROL MED LIDOKAIN | 1.25 |
| DEXAMETHASONE | 6.667 |

| Preferred term | Conversion factor for converting to a prednisone-equivalent dose |
|---|---|
| DEXAMETHASONE ACETATE | 6.667 |
| DEXAMETHASONE PHOSPHATE | 6.667 |
| DEXAMETHASONE SODIUM PHOSPHATE | 6.667 |
| FLUOCORTOLONE | 3 |
| HYDROCORTISONE | 0.25 |
| HYDROCORTISONE ACETATE | 0.25 |
| HYDROCORTISONE HYDROGEN SUCCINATE | 0.25 |
| HYDROCORTISONE SODIUM SUCCINATE | 0.25 |
| MEPREDNISONE | 1.25 |
| METHYLPREDNISOLONE | 1.25 |
| METHYLPREDNISOLONE ACEP | 1.25 |
| METHYLPREDNISOLONE ACETATE | 1.25 |
| METHYLPREDNISOLONE HEMISUCCINATE | 1.25 |
| METHYLPREDNISOLONE SODIUM SUCCINATE | 1.25 |
| PARAMETHASONE | 2.5 |
| PREDNISOLONE | 1 |
| PREDNISOLONE SODIUM PHOSPHATE | 1 |
| PREDNISOLONE SODIUM SUCCINATE | 1 |
| PREDNISONE | 1 |
| PREDNISONE ACETATE | 1 |
| TRIAMCINOLONE | 1.25 |
| TRIAMCINOLONE ACETATE | 1.25 |
| TRIAMCINOLONE ACETONIDE | 1.25 |

| Frequency Factors | |
|-------------------|--------|
| Frequency | Factor |
| BID | 2 |
| BIW | 2/7 |
| OAM | 1/30 |
| OD | 1 |
| Once | 1 |
| PRN | Null |
| Q2H | 12 |
| Q2W | 1/14 |
| Q3H | 8 |
| Q3D | 1/3 |
| Q3MO | 1/84 |
| Q3W | 1/21 |
| Q4H | 6 |
| Q4D | 1/4 |
| Q4W | 1/28 |
| Q6H | 4 |
| Q8H | 3 |

| Frequency Factors | |
|-------------------|--------|
| Frequency | Factor |
| Q12H | 2 |
| QAM | 1 |
| QD | 1 |
| QH | 24 |
| QHS | 1 |
| QID | 4 |
| QOD | 1/2 |
| QPM | 1 |
| QW | 1/7 |
| QWK | 1/7 |
| QM | 1/30 |
| TID | 3 |
| TIW | 3/7 |
| UNK | Null |
| 2 TIMES PER WEEK | 2/7 |
| 3 TIMES PER WEEK | 3/7 |
| 4 TIMES PER WEEK | 4/7 |
| EVERY 2 WEEKS | 1/14 |
| EVERY 3 WEEKS | 1/21 |
| EVERY 4 WEEKS | 1/28 |
| EVERY WEEK | 1/7 |

| Unit Conversion Factors | |
|-------------------------|---------|
| Unit | Factor |
| MCG | 0.001 |
| G | 1000 |
| MG/DAY | 1 |
| OZ | 28349.5 |
| UG | 0.001 |
| MG | 1 |

Any additions to the conversion factors or frequency factors noted above, that are identified during final data reconciliation but after RAP approval, will be documented prior to unblinding the study.

# 15.5. Appendix 5: SLICC/ACR Damage Index

| CCI - In | IIS SECTION | contained ( | ofore boye b | come Asses | ssment data | a collection | questionnai | res or indices, | , wnich are p | protected by third |
|---|---|---|---|---|---|---|---|---|---|---|
| party co | pyrigrit iaw | s and there | siore nave t | eri exciuo | ieu. | | | | | |

## CONFIDENTIAL

BEL115467

| Item | Score |
|---|---|
| Musculoskeletal | |
| Muscle atrophy or weakness | 1 |
| Deforming or erosive arthritis (including reducible deformities, excluding avascular necrosis) | 1 |
| Osteoporosis with fracture or vertebral collapse (excluding avascular necrosis) | 1 |
| Avascular necrosis (score 2 if $> 1$ ) | 1(2) |
| Osteomyelitis | 1 |
| Skin | |
| Scarring chronic alopecia | 1 |
| Extensive scarring or panniculum other than scalp and pulp space | 1 |
| Skin ulceration (excluding thrombosis) for > 6 months | 1 |
| Premature gonadal failure | 1 |
| Diabetes (regardless of treatment) | 1 |
| Malignancy (exclude dysplasia) (score 2 if > 1 site) | 1(2) |

(From the Systemic Lupus International Collaborating Clinics (SLICC) and the American College of Rheumatology Diagnostic and Therapeutic Criteria Committee, 1996)

Gladman EM, Ginzler E, Goldsmith C et al. SLICC/ACR damage index for SLE. Arthritis Rheum 1996;39(3):363-9.

## 15.6. Appendix 6: PSAP Sections for AESI Reporting

## **Section 15: Adverse Events of Special Interest**

AESI are defined using preferred terms from the current version of MedDRA. The intent is to update these definitions semi-annually using the newest MedDRA version. Preferred terms used in the current and prior versions of MedDRA can be found in Section 17.

## Section 15.1: Malignant neoplasms

Malignant neoplasms are identified using the sub-SMQs of Malignant or unspecified tumours (20000091), malignancy related conditions (20000092), haematological malignant tumours (20000227), non-haematological malignant tumours (20000228), haematological tumours of unspecified malignancy (20000229) and non-haematological tumours of unspecified malignancy (20000230) under the current version of MedDRA. The sub-SMQ of Malignant or unspecified tumours contains two further subcategories: "Malignant Tumours" and "Tumours of unspecified malignancy." Tumours of unspecified malignancy will be reviewed by GSK and identified as malignant or non-malignant for reporting.

Malignancies other than those in the "Tumours of unspecified malignancy" category will be categorized as hematologic, skin, or solid, based on a CMQ developed by the MAH (Section 17.1). In addition, the following customizations have been made (generally since MedDRA v19.1).

The following terms have been added as hematological tumour types:

Marginal zone lymphoma recurrent

Epstein Barr virus positive mucocutaneous ulcer

Primary gastrointestinal follicular lymphoma

Transformation to acute myeloid leukaemia

FIP1L1/PDGFR alpha fusion kinase positive

Acute bilineal leukaemia

Primary breast lymphoma

The following terms have been added as a solid tumour type:

Malignant meningioma metastatic

Astroblastoma

Langerhans cell sarcoma

Nasopharyngeal cancer metastatic

Phosphaturic mesenchymal tumour

Squamous cell breast carcinoma

Gleason grading score

Oncotype test

Malignant urinary tract obstruction

Sarcomatoid carcinoma

Cystadenocarcinoma pancreas

Paracancerous pneumonia

Chromophobe renal cell carcinoma

Gastrointestinal adenocarcinoma

Pleuropulmonary blastoma

Primary pulmonary melanoma

Dysplastic naevus

ALK gene rearrangement positive

Breast tumour excision

NMP22 test abnormal

The following terms have been added as a skin tumour type:

Naevoid melanoma

Trichoblastic carcinoma

The following terms have been added as a tumour of unspecified malignancy:

Mismatch repair cancer syndrome

Skin neoplasm bleeding

Intestinal metastasis

Maternal cancer in pregnancy

Microsatellite instability cancer

Pulmonary tumour thrombotic microangiopathy

Tumour cavitation

Tumour hyperprogression

Paraneoplastic myelopathy

Carcinogenicity

BRAF V600E mutation positive

Paraneoplastic thrombosis

In addition, the preferred term "Malignant neoplasm progression" was moved from "Non-haematological Malignant Tumour" SMQ in MedDRA Version 20.1 to "Malignancy Related Conditions" SMQ in MedDRA Version 21.0, and was further customized to be a tumour of unspecified malignancy.

The following terms have been removed from the SMQ:

Paraneoplastic glomerulonephritis (as it is a complication of malignancy)

Lymphoma cutis

Mucinous cystadenocarcinoma of pancreas

Serous cystadenocarcinoma of pancreas

Secondary cerebellar degeneration

Bone marrow infiltration

Pseudoachalasia

Malignant exophthalmos

Tumour obstruction

Tumour psuedoprogression

Paraneoplastic arthritis

Tumour pruritus

Oncogenic osteomalacia

Neurogenic tumour

Non-melanoma skin cancer (NMSC) will be categorized using a CMQ developed by the Marketing Authorization Holder (MAH) (Section 17.1).

Note beginning with MedDRA v20.0 in 2017, there will be two new sub-SMQs of Hematological Malignancies. These do not result in any changes to how malignant neoplasms are identified.

Post-study malignancies that are captured in ARGUS prior to CSR approval, but are not captured in the clinical database, will be described within the CSR text but cannot be included in statistical post-text displays. Post-study malignancies are not adjudicated by the SRT.

Additionally, for the BEL115467 "BASE" study, any malignancies that are reported annually (in the Year 2-5 post-treatment follow-up) via malignancy status updates in the CRF and not captured in ARGUS, will not be adjudicated by the SRT.

### Section 15.2: Post-infusion/injection systemic reactions

Post-infusion/injection systemic reactions will be identified using a customization of the Anaphylactic Reaction SMQ (20000021). This SMQ includes a broad list of preferred terms including symptoms of systemic injection/infusion reactions and hypersensitivity reactions and anaphylaxis. For the Anaphylactic Reaction query, 4 categories of preferred terms are considered, including a set of core anaphylactic terms (Category A), upper airway/respiratory terms (Category B), angioedema/urticaria/pruritus/flush terms (Category C), and cardiovascular/hypotension terms (Category D).

The customizations of the SMQ involve terms in Categories A, B and C:

- Category A has been modified to include the following additional terms: "Infusion-related reaction", "Drug hypersensitivity", "Hypersensitivity", and "Urticarial vasculitis".
- Category B has been modified to include the following additional terms: "Oropharyngeal oedema" and "Pharyngeal oedema".
- Category C has been modified to include the following additional terms: "Fixed eruption", "Drug eruption" and "Lipoedema".

GSK has also removed eight terms that are not relevant for an analysis of hypersensitivity reactions to belimumab ("Anaphylactic transfusion reaction", "Dialysis membrane reaction", "Cyanosis", "Nasal obstruction", "Ocular hyperaemia", "Tachypnoea", "Hereditary angioderma with C1 est" and "Acquired C1 inhibitor deficiency").

- Anaphylactic transfusion reaction is an adverse event associated with a blood transfusion, not related to study medication.
- Dialysis membrane reaction is associated with adverse events related to kidney transplants and dialysis, not related to study medication.
- Cyanosis, nasal obstruction, ocular hyperaemia, tachypnoea, hereditary angioderma with C1 est, acquired C1 inhibitor deficiency are adverse events generally not associated with post-infusion/injection systemic reactions.

The terms "Injection site urticaria", "Eye pruritis", and "Procedural shock" are part of the Anaphylactic Reaction SMQ but were inadvertently excluded (identified during PSAP Version 6 update). These terms will be included when the next MedDRA version i.e. MedDRA Version 21.1. is released.

## **Algorithmic Search Criteria**

The post-infusion/injection systemic reactions per Anaphylactic Reaction SMQ algorithmic search are defined as follows:

Subjects must have the following associated with the same infusion/injection:

a. at least 1 AE coding to a Category A preferred term or

- b. 2 AEs, 1 coding to a Category B preferred term and the other coding to a Category C preferred term *or*
- c. 2 AEs, 1 coding to a Category D preferred term and the other coding to either a Category B preferred term or to a Category C preferred term.

For the algorithmic search, if any event at a given infusion/injection meets the definition under criteria a, b or c, then all events in Categories A, B, C and D associated with that injection/infusion will be considered AESI.

GSK SRT will review all serious events identified via the broad search using a 21-day window from the start of an infusion/injection (see PSAP Section 8.3.2 for the definition of the assessment windows), and adjudicate these events as post-infusion/injection systemic reactions or hypersensitivity reactions per the criteria in Section 16.2. Therefore, the window for the narrow, broad and algorithmic searches of AE and SAE data from the clinical database for SRT reporting (PSAP Section 13.3) is 21 days to correspond to the window for adjudication. Adverse events with partial or missing start dates will be included unless there is evidence through comparison of partial dates to suggest otherwise.

Note, for CSR reporting, narrow, broad, and algorithmic searches of AE and SAE data will be run using a 3-day window from the start of an infusion/injection.

#### Sampson Criteria

Sampson et al define anaphylaxis as a severe, potentially fatal, systemic allergic reaction that occurs suddenly after contact with an allergy-causing substance. In addition, one of the following 3 criteria must be met: (1) acute onset of illness with involvement of skin or mucosal tissue, accompanied with either respiratory compromise, reduced blood pressure, or hypotension-related symptoms of end-organ dysfunction (2) reduced blood pressure associated with a known allergen or (3) two or more of the following that occur rapidly after exposure to an allergen: a) involvement of skin-mucosal tissue b) respiratory compromise c) reduced blood pressure d) persistent GI symptoms.

With the exception of GI symptoms, all symptoms required to assess anaphylaxis per Sampson criteria would be identified by Broad Anaphylaxis SMQ or the Anaphylactic Reaction SMQ algorithmic. Therefore, any events falling under the below criteria will be adjudicated by SRT prior to database release to determine if serious anaphylaxis per Sampson criteria is met.

Possible cases of serious anaphylaxis per Sampson criteria will be identified as follows:

- a. Any Infusion/Injection-related Reaction per Anaphylactic Reaction SMQ broad search SAE which occurs during the first 24 hours after the start of an infusion/injection.
- b. Any AE or SAE in the "Gastrointestinal disorders" SOC that coincides with the event that meets the criterion in a) above.
c. Any anaphylaxis and hypersensitivity reactions per Anaphylactic Reaction SMQ algorithmic search SAE which occurs during the first 24 hours after the start of an infusion/injection.

#### **Section 15.3: Infections**

The infections of special interest are described below.

# Section 15.3.1: Opportunistic Infections

Opportunistic infections will be identified using a broad CMQ developed by the MAH (Section 17.1). Any events falling under these preferred terms will be adjudicated by GSK to determine if criteria are met for an opportunistic infection, per the criteria in Section 16.3.

#### Section 15.3.2: Mycobacterium Tuberculosis

Tuberculosis events will be identified using a CMQ developed by the MAH (Section 17.1). Any events falling under these preferred terms will be adjudicated by GSK to determine if criteria are met for an opportunistic infection (Section 16.3).

# Section 15.3.3: Herpes Zoster

Herpes Zoster events will be identified using a CMQ developed by the MAH (Section 17.1). Additional manual adjudication by GSK will identify events that are recurrent or disseminated (Section 16.3).

#### Section 15.3.4: Pneumonia

Pneumonia events will be identified using a CMQ developed by the MAH (Section 17.1). Pneumonia events will not be reported separately, but are being flagged in the event further evaluation is necessary.

# Section 15.3.5: Sepsis

Sepsis events will be identified using a CMQ developed by the MAH (Section 17.1).

# Section 15.4: Depression/suicide/self-injury

# Section 15.4.1: Depression (excluding suicide and self-injury)

Depression events will be identified using a CMQ including the preferred terms from the depression (excluding suicide and self injury) SMQ (20000167) plus additional terms added by the MAH (Section 17.1).

#### Section 15.4.2: Suicide and Self-Injury

Suicide and self-injury events will be identified using the SMQ (20000037) plus additional terms added by the MAH (Section 17.1).

#### **Section 15.5: Fatalities**

All fatalities that are reported while a subject is eligible for SAE reporting will be identified in the clinical database and subsequently adjudicated by the GSK SRT into a general category of death (Section 16.5).

Post-study fatalities that are captured in ARGUS prior to CSR approval, but are not captured in the clinical database, will be described within the CSR text but cannot be included in statistical post-text displays. Post-study fatalities are not adjudicated by the SRT.

Additionally, for the BEL115467 "BASE" study, any fatalities that are reported annually (in the Year 2-5 post-treatment follow-up) via survival status updates in the CRF and not captured in ARGUS, will not be adjudicated by the SRT.

# Section 16: GSK SRT Adjudication of Adverse Events of Special Interest

Adverse events of special interest (AESI) are identified per the preferred terms(Section 17.1) and other criteria described in Section 15. The following AESI are adjudicated instream at the subject level by GSK during regular SRT meetings or during quarterly adjudication, and then prior to database release for CSR reporting purposes, per the criteria described below.

In-stream review/adjudication of AESI is conducted as follows:

#### • Review/Adjudication of AESI in ARGUS

Safety Evaluation and Risk Management (SERM) lists all events in ARGUS each month for SRT to review. AESIs are adjudicated at SRT meetings and entered onto Excel spreadsheets maintained by SERM. These spreadsheets are cumulative and contain events for all belimumab studies (clinical trials, post-marketing studies and spontaneous reports). SERM refer to these as "Cumulative AESI spreadsheets". SERM use these spreadsheets to tabulate the numerators used for PBRER/DSUR rates (see PSAP Section 7.6). The numerators are typically updated shortly after the Data Lock Point, and updated numerators are then used for PBRER/DSUR updates. The numerators are tracked in spreadsheets referred to as "AESI numerator spreadsheets".

# • Review/Adjudication of AESI in the Clinical Database

The SRT central programming team sends spreadsheets of AESIs based upon the CRF (Clinical Database) to SERM for periodic in-stream review. These spreadsheets contain AEs and SAEs and are study specific. SERM enter adjudication based on the SRT adjudication ("Cumulative AESI spreadsheets") and checks for missing serious AESIs between ARGUS and the Clinical Database. SERM send the clinical data derived spreadsheets to the study specific Medical Monitor, who adjudicates the non-serious events. Once updated, the spreadsheets are returned to the SRT central

programming team and are used to create the SRT output for the next periodic instream review.

In addition, as part of individual study close-out procedures, the adjudications should be finalized as follows:

- Just preceding database freeze (DBF), allowing time to send queries or update the eCRF/database as necessary prior to DBF, and are used in the CSR.
- Between DBR and Source Database Lock (as required) to provide final confirmation
  of adjudications and ensure there are no new AESI or relevant data changes to
  adjudicated events since the pre-DBR adjudication. This would be a requirement for
  declaring database freeze (DBF).

Note, at study close-out, the study programming team is responsible for generating spreadsheets of AESIs based upon the clinical data, in consult with the SRT central programming team, and liaising with SERM to finalise the adjudication. Refer to the SRT team site for more information: SRT/Team Documents/SRT documentation/AESI/Belimumab ADAE AEANAL AESI Adjudication Variables Process.doc.

# Section 16.1: Malignancies

All malignancies identified via the terms in Section 17.1 will be reviewed by GSK SRT. The classification of malignancies as solid tumor, hematological, and skin will be reviewed against the verbatim term to confirm an appropriate and accurate preferred term has been assigned, or to recommend follow-up with the investigator for additional specificity on the verbatim term. In addition, malignancies that are flagged more than once, e.g., based on a term for both a diagnostic procedure and a diagnosis, will be adjudicated as one event.

Tumors of unspecified malignancy, as identified per the terms in Section 17.1, will be reviewed clinically by the GSK SRT for reporting. In general, non-serious events in the tumours of unspecified malignancy with insufficient information will be categorized as not malignant. Serious adverse events with insufficient information will be categorized as either not malignant or malignant based on the type of tumor and likelihood the tumor type is malignant (e.g., thyroid nodules are common in SLE patients and are generally not malignant; tumor types with higher likelihood for malignancy would be assumed to be malignant).

#### Section 16.2: Serious hypersensitivity and post-infusion/injection systemic reactions

GSK SRT will review all serious cases identified from the Broad Anaphylaxis SMQ as described in Section 15 and Section 17.1, applying clinical judgment to determine if the preferred terms are indicative of a hypersensitivity or post-infusion/injection reaction. Time to onset after an infusion/injection and details provided in the clinical narratives with respect to the nature and likely cause of the events are taken into consideration. The GSK SRT adjudicates serious hypersensitivity reactions into a category based primarily on time to onset: acute (onset < 24 hours), delayed acute (onset 2-3 days), or delayed, non-acute (onset 4-21 days). In addition to time to onset, description of associated symptoms is taken into account for this categorization. In studies where subjects are

receiving weekly injections, any delayed, non-acute reactions will typically occur in the interval 4-7 days later, but may occur up to 21 days later following a missed injection or after the last injection.

In addition, possible cases of serious anaphylaxis per Sampson criteria will be identified per the criteria in Section 15. Any events falling under these criteria will be adjudicated by GSK prior to database release to determine if serious anaphylaxis per Sampson criteria is met.

# Section 16.3: Potential opportunistic infections

Opportunistic infections (OIs) will be identified using a list of preferred terms (Section 17.1), designed to cast a wide net for events potentially indicative of an opportunistic infection. Any identified events will be adjudicated by the GSK SRT to determine if criteria are met for an opportunistic infection. Targeted follow-up is sought for events with insufficient information. In general, potential OIs that are non-serious with insufficient information to adjudicate will be considered non-opportunistic. Potential OI SAEs with insufficient information to adjudicate will be considered opportunistic. See below for a list of agreed upon pathogens and infections considered to be opportunistic for the purpose of adjudication.

#### **Pathogens and Infections Considered Opportunistic:**

- Acinetobacter infection
- Aspergillosis
- Blastomycosis, extrapulmonary
- Candidiasis of esophagus, bronchi, trachea or lungs
- Capnocytophaga infection
- Coccidioidomycosis, disseminated or extrapulmonary
- Cryptococcosis, extrapulmonary
- Cryptosporidiosis infection, chronic intestinal (greater than 1 month duration)
- CMV disease other than liver, spleen, or nodes
- Herpes simplex bronchitis, pneumonitis, or esophagitis
- Herpes Zoster (adjudication details are below)
- Histoplasmosis disseminated or extrapulmonary
- Human polyomavirus infection
- Isosporiasis, chronic intestinal (greater than one month duration)
- Listeriosis
- Mycobacterium avium complex or M. Kansasii, disseminated or extrapulmonary
- Nocardiosis
- Other non-tuberculous mycobacterium (NTM) infections (other species or unidentified species), disseminated or extrapulmonary\*
- Polyomavirus (JC virus or BK virus) associated nephropathy (including PML)
- Pneumocystis jiroveci infection
- Toxoplasmosis of brain

\* Extra pulmonary NTM infections are generally considered an OI unless the affected extra pulmonary area followed a wound or trauma.

In addition, GSK SRT will review all SAEs, including those coded under preferred terms not listed in Section 17.1, and utilizing the supplemental/narrative information, will adjudicate the SAEs as OI if warranted based on medical judgment.

### Other Infections of Interest but not generally considered opportunistic:

- Mycobacterium tuberculosis (adjudication details are below)
- Salmonella sepsis there may be rare exceptions in which the presentation is atypical, which will be considered on a case-by-case basis by the SRT.
- Hepatitis B
- Hepatitis C

#### Herpes Zoster

Herpes Zoster events will be identified per terms in Section 17.1. Adjudication by GSK SRT will identify events that are recurrent or disseminated. Herpes Zoster is considered disseminated if there is involvement of other organs other than the skin or if skin lesions (1) cross the midline of the body or (2) are in non-adjacent dermatomes or (3) are located in more than three adjacent dermatomes. Herpes zoster is considered an opportunistic infection if it is adjudicated as recurrent or disseminated. However, there may be some uncommon occurrences of a herpes zoster case that is adjudicated as an OI but is neither recurrent or disseminated.

# **Mycobacterium Tuberculosis**

Tuberculosis (TB) cases are reviewed by the GSK SRT to determine if a case is an OI. The following principles are applied: Pulmonary TB in an endemic area is not considered an OI. Pulmonary TB in an non-endemic area would be considered an OI unless the subject had close contact with a person infected with TB. Extra pulmonary TB is generally considered an OI unless the affected extra pulmonary area followed a wound or trauma.

# Section 16.4: Suicide/self-injury

Suicide and self-injury SAEs will be identified using the preferred terms identified in Section 17.1 and subsequently adjudicated into the following categories:

| Adjudicated Category |
|--------------------------------------------------|
| Suicidal Behaviour |
| Completed Suicide |
| Suicidal Ideation |
| Self-Injurious Behaviour without Suicidal Intent |

In addition, GSK SRT will review all SAEs, including those coded under preferred terms not listed in Section 17.1, and utilizing the supplemental/narrative information, will adjudicate the SAEs as suicide/self-injury if warranted based on medical judgment.

#### Section 16.5: Fatalities

All fatalities that are reported while a subject is eligible for SAE reporting will be identified in the clinical database and subsequently adjudicated by the GSK SRT into a general category of death.

All fatalities will be adjudicated into one of the following categories:

| <b>Adjudicated Category of Death</b> |
|--------------------------------------|
| SLE-Related |
| Infectious |
| Vascular |
| Gastrointestinal |
| Respiratory |
| Malignancy |
| Hypersensitivity |
| Suicide |
| Surgical Complication |
| Unknown |
| Hematologic |
| Trauma |

Additional 'categories of death' may be added in the future should a fatality not clearly fit into one of the 'categories' listed above. The 'categories' will not change unless agreed upon by the GSK SRT.

# Section 17: AESI Preferred term definitions under current and prior versions of MedDRA

The AESI definitions under the current version of MedDRA are found via the IMMS pathname in Section 17.1. Prior AESI definitions under legacy versions of MedDRA are found in the subsequent sections.

#### Section 17.1: MedDRA v21

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 21.csv

#### Section 17.2: MedDRA v20.1

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 201.csv

#### Section 17.3: MedDRA v20.0

#### CONFIDENTIAL

BEL115467

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 20.csv

Section 17.4: MedDRA v19.1

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 191.csv

Section 17.5: MedDRA v19.0

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 19.csv

Section 17.6: MedDRA v18.1

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 181.csv

Section 17.7: MedDRA v18.0

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 18.csv

Section 17.8: MedDRA v17.1

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 171.csv

Section 17.9: MedDRA v17.0

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 17.csv

Section 17.10: MedDRA v16.1

The AESI definitions were not updated for MedDRA v16.1.

Section 17.11: MedDRA v16.0

/Study File/GSK1550188/ Project/Meta Analysis/PSAP/AESI 16.csv

# 15.7. Appendix 7: Mortality Missing Data Exploratory Sensitivity Analyses

Whilst extensive efforts have been made to achieve complete ascertainment of vital status (alive, dead) at Week 52 for the As Treated Population, it is acknowledged that it will be unattainable for a low percentage of subjects.

This appendix outlines the methodology for potential exploratory sensitivity analyses of mortality (primary analyses defined in RAP Section 11.1.1). The need to conduct the supplemental estimand sensitivity analysis described in Section 15.7.1.3 will be assessed following study team review of the Statistical Analysis Complete (SAC) package.

The draft ICH E9 addendum has been used as guidance/a framework in determining the strategy for the exploratory sensitivity analyses, including the handling of intercurrent events occurring prior to Week 52. Intercurrent events are defined as "events that occur after treatment initiation and either preclude observation of the variable or affect its interpretation" e.g. premature discontinuation of study agent or study withdrawal.

# 15.7.1. Estimand Framework

#### 15.7.1.1. Main Estimand: While On Treatment

The main estimand aligns to the primary endpoint as defined in the main body of the RAP (Section 11.1.1). It is chosen as the main estimand because the endpoint is being evaluated to address safety objectives.

Therefore, whilst outlined here using an Estimand framework, it does not represent a different analysis to that specified in Section 11.1.1.

#### **Endpoint/Variables**

Mortality status while on treatment (to treatment stop date + 28 days).

#### **Summary Measure**

95% Confidence Interval around the difference in percentage of deaths while on treatment.

# **Population of Interest**

The primary efficacy analyses are based on the As-Treated population, unless otherwise specified.

# Strategy for Intercurrent (Post-Randomization) Events

Premature discontinuation of study agent and/or study withdrawal are not relevant here as we are only using data whilst subjects were on-treatment.

#### **Statistical Analyses / Methods**

# **Statistical Methodology Specification**

#### **Endpoint / Variables**

Mortality status while on treatment

# **Model Specification**

Simple asymptotic Chi-Square (Pearson) method for a 95% CI

#### **Model Results Presentation**

Number of deaths and percentage in each treatment group and the difference in percentage with 2-sided 95% CI.

# 15.7.1.2. Supplemental Estimand: While On Study

This estimand is defined to estimate the treatment difference while subjects were onstudy. This will include observed on- and off- treatment data to Week 52 and aligns to the on-study estimate defined in the main body of the RAP (Section 11.1.1).

Therefore, whilst outlined using an Estimand framework, it does not represent a different analysis to that specified in Section 11.1.1.

# **Endpoint/Variables**

Mortality status at Week 52 (observed data while on study).

# **Summary Measure**

95% Confidence Interval around the difference in percentage of deaths while subjects were on-study.

# **Population of Interest**

The primary efficacy analyses are based on the As-Treated population, unless otherwise specified.

# **Strategy for Intercurrent (Post-Randomization) Events**

Premature discontinuation of study agent and/or study withdrawal are dealt with in the variable given that all data whilst subjects were in the study (i.e. on- and off- treatment data) is included. Data beyond the observed on-study period is not imputed.

### **Statistical Analyses / Methods**

# **Statistical Methodology Specification**

# **Endpoint / Variables**

Mortality status at Week 52 (observed data while on study)

### **Model Specification**

Simple asymptotic Chi-Square (Pearson) method for a 95% CI

#### **Model Results Presentation**

Number of deaths and percentage in each treatment group and the difference in percentage with 2-sided 95% CI will be presented.

# 15.7.1.3. Supplemental Estimand Sensitivity: Treatment Policy

A sensitivity to the Supplemental Estimand targeting the same estimand is defined with a Treatment Policy approach. Subjects with missing vital status at Week 52 have their vital status imputed using observed off-treatment data.

If the imputation of missing vital status is unsuccessful due to insufficient off-treatment data being available, the interaction term will be removed from the Cox Proportional Hazards model. If the imputation is still not possible, this estimand will not be estimated.

# Endpoint/Variables

Mortality status at Week 52 (observed data while on study and imputed data to Week 52).

# **Summary Measure**

95% Confidence Interval around the difference in percentage of deaths at Week 52.

#### **Population of Interest**

The primary efficacy analyses are based on the As-Treated population, unless otherwise specified.

# **Strategy for Intercurrent (Post-Randomization) Events**

A Treatment Policy strategy will be used for all intercurrent events. If data are available after the intercurrent event, e.g. where subjects continue in the study post premature study agent discontinuation, these data will be included in the summary. For subjects with missing vital status at Week 52, time to death will be imputed using observed off-treatment data and from this vital status at Week 52 will be derived to allow us to calculate incidence at Week 52.

### **Statistical Analyses / Methods**

#### Statistical Methodology Specification

#### **Endpoint / Variables**

Mortality status at Week 52 (observed data while on study and imputed data to Week 52)

# **Model Specification**

Simple asymptotic Chi-Square (Pearson) method for a 95% CI

#### **Model Results Presentation**

Number of deaths and percentage in each treatment group and the difference in percentage with 2-sided 95% CI will be presented.

#### Methodology

The multiple imputation of vital status at Week 52 will be performed using time to event modelling to predict the time to death for subjects with missing vital status, with the treatment difference being estimated for each imputed dataset and then combined as described below:

- Step 1: The data will be structured so each subject has up to two records; one record for the on-treatment data and one record for the off-treatment data (where off-treatment data is present). Bootstrap from these data and fit a Cox Proportional hazard model  $h(t) = h_0(t) \exp\{\beta x + \delta z + \gamma xz\}$ , where x represents treatment groups (x=0 for placebo subjects and x=1 for belimumab subjects) and z is an indicator variable for either the "on" or "off" treatment component of the subjects' data (z=0 for on-treatment and z=1 for off-treatment), to estimate the hazard with censoring at random assumption.
- **Step 2:** Obtain the data from the subjects to be imputed. Use the above estimated baseline hazard to estimate hazard for subjects with missing vital status at Week 52.
- **Step 3:** Obtain the value of  $\beta x + \delta z + \gamma xz$  for those subjects and modify the baseline hazard accordingly.
- **Step 4:** Impute the time to death for subjects who were censored prior to Week 52 based on their assigned hazard.
- **Step 5:** Aggregate the subjects' on and off-treatment records to obtain the subjects' time to death. For subjects whose time to death is  $\leq$  Study Day 372 assign as death and for subjects whose time to death is  $\geq$  Study Day 372, censor at Study Day 372.
- **Step 6:** Repeat the above step for 'm' number of times to obtain 'm' imputed values in 'm' datasets.
- **Step 7:** For each imputed dataset, compute the proportions of deaths in each treatment arm and the associated standard errors. Then calculate the difference in proportions between the treatment arms and associated standard error.
- **Step 8:** Lastly use Rubin's rule [Rubin, 1987] to combine the results to estimate the treatment difference and 95% CI combined across 'm' datasets.

# 16. ATTACHMENTS

# 16.1. Table of Contents for Data Display Specifications

See separate TFL document.

# 16.2. Data Display Specifications

See separate TFL document.

# 16.3. Headline Results

The following TFLs will be included as headline results:

| Display<br>Type | Display<br>Number | Display Title |
|---|---|---|
| Table | 1.02 | Summary of Study Populations |
| Table | 1.06 | Summary of Subject Status and Reason for Study<br>Withdrawal |
| Table | 1.07 | Summary of Subject Status and Reason for Discontinuation of Study Agent |
| Table | 1.12 | Summary of Demographic and Baseline Characteristics |
| Table | 1.20 | Summary of Baseline Disease Activity |
| Table | 2.01 | Summary of Mortality (On-Treatment Period) |
| Table | 2.03 | Summary of Mortality (On-Study Period) |
| Table | 2.05 | Summary of Protocol-Defined Adverse Events of<br>Special Interest (On-Treatment Period) |
| Table | 2.06 | Summary of Protocol Defined Adverse Events of<br>Special Interest (On-Study Period) |
| Table | 3.001 | Adverse Events of Special Interest and Serious Adverse<br>Events Summary (On-Treatment Period) |
| Table | 3.003 | Adverse Events of Special Interest and Serious Adverse Events by SOC (On-Treatment Period) |
| Table | 3.004 | Adverse Events of Special Interest and Serious Adverse Events by SOC and PT (On-Treatment Period) |
| Table | 3.009 | Serious Adverse Events by SOC (On-Treatment Period) |

| Display<br>Type | Display<br>Number | Display Title |
|---|---|---|
| Table | 3.010 | Serious Adverse Events by SOC and PT (On-Treatment Period) |
| Table | 3.015 | Study Agent Related Adverse Events of Special Interest<br>and Serious Adverse Events by SOC (On-Treatment<br>Period) |
| Table | 3.019 | Adverse Events of Special Interest and Serious Adverse<br>Events leading to Study Agent Discontinuation by SOC<br>and PT (On-Treatment Period) |
| Table | 3.037 | Adverse Events of Special Interest (PSAP-Defined) by<br>Category (On-Treatment Period) |
| Table | 3.048 | Deaths by Category and PT (On-Treatment Period) |
| Figure | 2.03 | Time to Mortality (On-Treatment Period) |
| Figure | 2.04 | Time to Mortality (On-Study Period) |

Additional TFLs may be added depending on the results of the study if agreed upon by the Study team.

# 16.4. Disclosure Outputs

The following outputs are required for disclosure:

| Display<br>Type | Display<br>Number | Display Title | Required by |
|---|---|---|---|
| Table | 1.01 | Randomization by Site | EudraCT |
| Table | 1.06 | Summary of Subject Status and Reason for Study Withdrawal | FDAAA, EudraCT |
| Table | 1.12 | Summary of Demographic and Baseline<br>Characteristics | FDAAA, EudraCT |
| Table | 1.13 | Summary of Age Ranges | EudraCT |
| Table | 1.14 | Summary of Race and Racial<br>Combination Details | FDAAA, EudraCT |
| Table | 3.010 | Summary of Serious Adverse Events by | FDAAA, EudraCT |

# CONFIDENTIAL

# BEL115467

| Display<br>Type | Display<br>Number | Display Title | Required by |
|---|---|---|---|
| | | SOC and PT (On-Treatment Period) | |
| Table | 3.024 | Common (>=1%) Non-Serious Adverse<br>Events of Special Interest by PT (On-<br>Treatment Period) | FDAAA, EudraCT |